## **COMprehensive Post-Acute Stroke Services (COMPASS) Study**

#### Principal-Investigator:

• Pamela Duncan, PhD, PT

#### Co-Investigators:

#### Wake Forest

- Cheryl Bushnell, MD, MHS (Co-PI)
- Walter Ambrosius, PhD
- Ralph D'Agostino, PhD
- Sabina Gesell, PhD
- Allison Brashear, MD, MBA
- Brian Wells, MD, PhD

#### UNC Chapel Hill

- Wayne Rosamond, PhD (Co-PI)
- Janet Freburger, PhD, MS
- Jacqueline Halladay, MD, MPH
- Anna Kucharska-Newton, PhD, MPH, MS

#### **UNC Wilmington**

• Barbara Lutz, PhD, RN

#### East Carolina University

• Doyle "Skip" Cummings, PharmD

#### **Duke University**

- Janet Prvu Bettger, ScD
- Amy Pastva, PhD, PT

### Sponsor:

Patient-Centered Outcomes Research Institute (PCORI)

## Contents

| COMprehensive Post-Acute Stroke Services (COMPASS) Study | 1 |
|---|---|
| Background | 5 |
| Objectives & Specific Aims | 6 |
| Primary Study Question: | 6 |
| Primary Aim: | 6 |
| Secondary Aims: | 6 |
| Exploratory Aims: | 6 |
| Methods and Measures | 8 |
| Study Design | 8 |
| Study Setting | 8 |
| Study Population | 8 |
| Randomization | 8 |
| Subjects Selection Criteria | 9 |
| Inclusion Criteria: | 9 |
| Exclusion Criteria: | 9 |
| Sample Size: | 9 |
| Intervention and Interactions | 10 |
| Phase 1: Patients in Control Hospitals | 10 |
| Phase 1: Patients in COMPASS-Intervention Hospitals | 11 |
| Phase 2: COMPASS-Intervention & COMPASS-Sustain Hospitals | 13 |
| Phase 1 Only: Caregivers Outcomes Survey | 15 |
| Phase 1 & Phase 2: Community-Engagement | 15 |
| Outcome Measures | 17 |
| Patient Participant Study Outcomes (Phase 1 and 2): | 17 |
| Caregiver Participant Study Outcomes (Phase 1 only): | 20 |
| Study outcomes collected and linked to insurance claims data (Phase 1 & Phase 2): | 21 |
| Clinical Data collection: | 22 |
| Analytical Plan | 24 |
| Human Subjects Protection | 26 |
| Informed Consent | 28 |
| Confidentiality and Privacy | 30 |
| Overview | 30 |
| COMPASS Analytic Database at EMSPIC | 30 |
| Electronic Care (eCare) Plan Informatics Database | 30 |
| Carolina Survey Research Lab Database and Security | 31 |
| Sheps Center Data Security | 32 |
| Description of the Secure Data Transfers | 33 |

## March 19, 2021 Application - IRB00035998 REDCap (Research Electronic Data Capture) 34 Data and Safety Monitoring......35 Responsibilities 35 References 37 Appendix 16 - Two-Day Post-Discharge Follow-up .......94 Appendix 18 - Caregiver Assessment 108

| Application - IRB00035998 | |
|---|---|
| Appendix 30 - Caregiver Thank You Note | 175 |
| Appendix 31 - IRB Approval Letter for PCORI Stakeholder Interviews | 176 |
| Appendix 32 - DSMB Template Sections | 177 |
| Appendix 33 – CTSI Supplemental Proposal (Implementation of COMPASS) | 178 |
| Appendix 34 – 2Day Disposition Form | 181 |
| Appendix 35 – Clinic Disposition Form | 182 |
| Appendix 36 – Phase 2 Patient Brochure for Sustaining COMPASS Hospitals | 186 |
| Appendix 37 – Phase 2 Patient Brochure for Intervention Sites (formerly Usual Care) | 187 |
| Appendix 38 – Phase 2Enrollent Form | 188 |
| Appendix 39 – Consent Matrix | 193 |

## **Background**

Stroke is the fifth-leading cause of death in the United States (US) and a major cause of long-term disability. North Carolina (NC) is in the Stroke Belt, a region of the US with a very high stroke incidence. Eastern NC is the "buckle" of the Stroke Belt, where stroke mortality is 40% higher than the US average and hospital admission rates are the highest in NC. African Americans, over 20% of the population in NC, are more likely than their white counterparts to die of stroke at relatively young ages. There is also evidence that African-Americans are more likely to be readmitted after stroke.

Stroke exemplifies a complex co-morbidity condition, with 85% of Medicare beneficiaries with stroke having four or more other chronic health conditions,<sup>4</sup> and their health care is costly. Stroke patients with congestive heart failure have per capita costs that are about five times higher than the average spending for Medicare fee-for-service beneficiaries.<sup>4</sup> In addition, stroke patients are frequently readmitted to the hospital.<sup>5,6</sup> A PCORI-funded study shows that 25% of stroke patients discharged home without post-acute care are readmitted within 90 days<sup>7</sup>. These data align with what stroke survivors and caregiver advocates from across NC have said that stroke patients need. One of our patient partners who started a support group for other stroke survivors stated:

"You can't just place an individual back in their home with a bottle of pills and a follow-up visit...There is a real need for assistance when patients get home...What is in place for the patient? Nothing... No visiting nurse, no one to answer questions, or help them get what they need. That is why people end up back in the hospital."

Roughly half of stroke patients in NC are discharged directly home, often with new disability. Around 44% cannot walk independently at discharge. Complications from immobility account for up to 51% of deaths in the first 30 days after ischemic stroke. Other complications are common early after stroke and include falls and fractures, aspiration pneumonia, deep vein thrombosis, infections, depression, and adverse events associated with warfarin therapy. 11–16 Even those with mild post-stroke disability can have physical and cognitive deficits which often go undetected during acute hospitalization. These mild disabilities interfere with function, and management of risk factors and medication. 17,18

Fewer than 50% of individuals with stroke have their risk factors assessed, treated, or controlled. Of those overweight at initial evaluation, 90% remain overweight. Nearly half of hypertensive individuals do not have blood pressure controlled. Smokers do not quit and few participate in exercise programs. At three months post-discharge, only 75% of stroke patients are still taking their preventive medications. About 40% remain dependent on others. Stroke also affects caregivers. Caregivers have poorer mental health, less social contact and activity, and are at increased risk for depression.

Comprehensive post-acute services for stroke require bridging hospital-based acute care with expanded care teams for rehabilitation, primary care management, access to community resources, and caregiver support. Evidence-based reviews have concluded that stroke morbidity and mortality could be reduced through effective transitional care, <sup>22–24</sup> secondary prevention, <sup>25</sup> and rehabilitation early post-stroke. <sup>26</sup> Involvement with a stroke liaison worker or case manager is associated with more knowledge about stroke and satisfaction with services. <sup>27,28</sup> Caregiver-oriented, individualized discharge planning for stroke patients going home improves caregiver preparedness. <sup>29</sup>

Given the significant impact of stroke on public health, the high risk and complexity of these patients early after discharge, and the strain on caregivers, an effective post-acute care model is needed. A pragmatic trial is the ideal method to test a care model that can be readily disseminated and implemented.

## **Objectives & Specific Aims**

The COMprehensive Post-Acute Stroke Services (COMPASS) Study will determine the effectiveness of a post-acute comprehensive intervention.

#### **Primary Study Question:**

Does implementation of the COMPASS for stroke patients discharged directly home, improve functional outcomes (measured by the Stroke Impact Scale-16) at 90 days post-stroke? Intention-to-treat principles will be used to determine all primary and secondary outcomes.

#### **Primary Aim:**

Comparative effectiveness of COMPASS verses usual care (Control) on stroke survivor functional status (measured by the Stroke Impact Scale) at 90 days post-stroke.

#### **Secondary Aims:**

- 1) Using responses from the 90 day caregiver survey, determine if the COMPASS intervention reduces caregiver strain (measured by the Modified Caregiver Strain Index) at 90 days post-stroke.
- 2) Using responses from the 90 day survey, we will measure self-rated general health; medication adherence (MMAS-4); self-monitoring of blood pressure; global disability; physical activity; depression (PHQ2); cognition (Mini MOCA); falls; fatigue; and satisfaction of care.
- 3) Using claims data from multiple payer sources up to 12 months after stroke hospitalization, we will measure effectiveness of COMPASS vs usual care for all-cause readmissions at 30 and 90 days and 1-year post-discharge.
- 4) Comparative effectiveness of the COMPASS vs usual care on: mortality; health care utilization; (emergency department visits, admissions to skilled nursing facilities/inpatient rehabilitation facilities); and use of transitional care management billing codes. We will use claims data from multiple payer sources up to 12 months after stroke hospitalization.
- 5) For all outcomes we will adjust analyses to account for race, sex, age, stroke severity, and insurance status.

#### **Exploratory Aims:**

- 1) Phase 2: The implementation sustainability objectives for Phase 2 of the COMPASS Study are to characterize whether rates of transitional care management (TCM) delivery and eCare plan delivery are sustained, worsen, or improve during the sustainability period of the COMPASS study for hospitals randomized to the intervention during Phase 1.
- 2) Phase 2: The effectiveness sustainability objective for Phase 2 of the COMPASS Study is to characterize whether patient outcomes are sustained, worsen, or improve during the sustainability period of the COMPASS study for hospitals randomized to the intervention during Phase 1.
- 3) Phase 2: The primary comparative effectiveness objective for Phase 2 of the COMPASS Study is to evaluate whether Stroke Impact Scale 16 (SIS-16) scores are improved during Phase 2 (i.e., the intervention phase) for hospitals randomized to usual care in Phase 1.
- 4) Phase 2: Using Claims, the Pre-Post analyses compared outcomes in hospitals randomized to provide UC in Phase 1 with outcomes among those that crossed over and delivered the INV in Phase 2 for mortality; health care utilization; (emergency department visits, admissions to skilled nursing facilities/inpatient rehabilitation facilities); and use of transitional care management billing codes. We will use claims data from multiple payer sources up to 12 months after stroke hospitalization.
- 5). Phase 2: Using Claims, the Sustainability analyses compared outcomes in hospitals randomized to deliver the INV in Phase 1 with outcomes among those that sustained the intervention (SUS) in Phase 2 for mortality; health care utilization; (emergency department visits, admissions to skilled nursing facilities/inpatient rehabilitation

Application - IRB00035998

facilities); and use of transitional care management billing codes. We will use claims data from multiple payer sources up to 12 months after stroke hospitalization.

### **Data Collected for Ancillary Studies:**

- 1) Analysis of individual, organizational, and community factors affecting implementation of COMPASS through supplemental funding (CTSI Award lead by Co-I Dr. Gesell). This pilot project will contribute to a process evaluation of our Phase1, intervention-randomized health systems adopting COMPASS.
- 2) An exploratory analysis that compares patient clinic return rate and use of services to physical locations of patients and services (i.e. distance and drive times to/from clinics and community resources).
- 3) At the 90 day survey, we will also use the PROMIS Global-10 instrument that assesses general domains of health and functioning including overall physical health, mental health, social health, pain, fatigue, and perceived quality of life. These are similar in nature to our primary outcome, the SIS-16.

#### Hospital Performance Metrics (to support participating sites in delivery of the intervention):

1) Evaluate compliance with the new model of post-acute stroke care by exploring quality indicators among intervention hospitals, (e.g., proportion of patients called within 2 days after hospital discharge; proportion of patients seen by an advanced practice provider [MD/NP/PA] within 7 to 14 days from hospital discharge; and proportion of eligible patients receiving home or outpatient rehabilitation therapy).

#### **Methods and Measures**

#### **Study Design**

The COMPASS Study is a pragmatic, cluster-randomized trial of 41 hospitals in North Carolina designed to determine the effectiveness of a model of post-acute stroke care (i.e. the COMPASS Intervention) compared with usual care (Control).

#### **Study Setting**

The COMPASS intervention will be implemented in hospitals and communities in 2 phases over a 5-year period. We will recruit 41 hospitals that represent diverse geographic locations (i.e. rural vs urban), primary stroke center certification status, and stroke patient volumes. Included in this IRB Application (Appendix 1) is an attachment (Titled: COMPASS Hospital Characteristics) which provides a side-by-side comparison of hospitals expected to participate in the COMPASS trial with All North Carolina Hospitals. A list of our COMPASS Hospitals is also included. The data used to make the comparison is from CMS Hospital Compare<sup>30</sup>. COMPASS will ask participating hospitals to fill out a Hospital Survey (Appendix 2) at the start of the study to better understand the current state of transitional care at each hospital.

#### **Study Population**

In 2013, data from hospitals in the North Carolina Stroke Care Collaborative (NCSCC) indicated that 46% of patients were discharged directly home from the hospital after a stroke (our proposed study population). Using this data we anticipate an estimated sample of approximately 6,000 potentially eligible participants. In that population, the mean age was 65.0 years (SD 14.4), 25% were African American, and 48% were women. Stroke severity, measured by the NIH Stroke Severity score and ranging from 0 (no deficit) to 42 (maximum deficits), was on average 3.2 for those discharged home.

#### **Randomization**

Since individual stroke patients cannot easily be randomized to receive the COMPASS intervention, we determined that the optimal statistical design for this pragmatic trial utilizes a cluster randomized approach. Thus, 41 individual hospitals will be randomized to either receive the COMPASS intervention at the beginning of the study (Phase 1) or in Phase 2 (see Figure 1). Two of the participating 41 hospitals were randomized together, therefor we have 40 randomized units. Hospitals randomized to receive the intervention in Phase 2 will be referred to as the control group. Randomization per hospital will be stratified by volume of stroke patients and primary stroke center status. In this intention-to-treat design, all stroke patients who are discharged directly home from randomized acute care hospitals will be included in



Figure 1: Hospital Randomization to the COMPASS Intervention in Phase 1 and Phase 2

analyses. The analyses will be performed at the individual level with adjustment for lack of independence between hospitals. The primary analysis of patient-centered outcomes will occur at the end of Phase 1.

## **Subjects Selection Criteria**

#### **Inclusion Criteria:**

 Patients aged 18 years or older, discharged home from a participating COMPASS Study hospital with a diagnosis of ischemic or hemorrhagic stroke or transient ischemic attack (TIA).

#### **Exclusion Criteria:**

- Patients transferred to another short-term acute care hospital, skilled nursing facility, inpatient rehabilitation facility, or hospice.
- Patients with a diagnosis of subdural or aneurysmal subarachnoid hemorrhage.
- Patients who speak neither English nor Spanish.

#### **Sample Size:**

- Approximately 6,000 potentially eligible participants during Phase 1
- Approximately 6,000 potentially eligible participants during Phase 2

#### **Intervention and Interactions**

As described in the Methods section above, the trial has two Phases (see Figure 1).

- Phase 1: Patient enrollment for Phase 1 of the trial will run from June 2016 to March 2018. Phase 1 includes a control arm (Control Hospital) and an intervention arm (COMPASS-Intervention Hospitals). Details of these arms and interactions are described below. Figure 2 depicts the patient flow of activities for Phase 1 when there is a control arm and COMPASS intervention arm.
- Phase 2: Patient enrollment for Phase 2 of the trial will run from November 2017 January 2019. Phase 2 includes an intervention arm (COMPASS-Intervention hospital) and the other arm is COMPASS Hospitals who will sustain the COMPASS intervention using their own hospital resources (COMPASS-Sustain hospital). Detail of these arms and interactions are described below.
- Note, that there is some overlap between Phases 1 and 2. The overlap is due to differences in the timing of hospital recruitment and enrollment (i.e. larger hospitals enrolled patients faster).

COMPASS will support hospitals in implementing structured post-acute stroke services consistent with CMS transitional care codes and management. Hospitals which participate are implementing COMPASS as the new standard of care. The goal of COMPASS is to structure and organize the processes of post-acute care to optimize patient recovery function, reduce caregiver stress, improve risk factor management, and facilitate self-management of risk factors.

#### **Phase 1: Patients in Control Hospitals**

Prior to hospital discharge, the Post-Acute Coordinator (PAC) will identify stroke and TIA patients for eligibility using the Eligibility Screening Form (Appendix 3). Determining eligibly will involve daily review of stroke admissions to the hospital by screening the electronic medical records. This will be done under Limited HIPAA Waiver.

If eligible, the patient will be enrolled, a COMPASS ID is assigned and the PAC will fill out the Enrollment Form (Appendix 4). For those not eligible, no further information is collected and a COMPASS Identification number is not assigned. Enrollment will be done under a Full HIPAA Waiver.

The PAC will visit eligible patients in the hospital, notify the patient that the hospital is participating in the COMPASS Study, and give the patient a handout with information on the COMPASS Study (Appendix 5). The information informs the patient that their hospital is participating in a statewide study to evaluate best models of post-stroke care. The patient will be informed if their hospital is in the usual care group or in the COMPASS intervention group. The handout that patients receive in the control arm is

Control COMPASS Prior to Eliaibility Hospital Eliaibility Discharge Prior to Enrollment, Enrollment Hospital COMPASS Handout COMPASS Handout Discharge NCSCC Registry Retween NCSCC Registry 0-30 Days Stroke Card Stroke Card Follow-up 2 Day 2 Days Phone Call 7-14 Day 7-14 Days APP Visit 30 Day Reminder 30 Day Reminder 30 Days Letter Letter Follow-up 30 Day 30 Days Phone Call 60 Day Reminder 60 Day Reminder 60 Days Letter Letter Follow-up 60 Day 60 Days Phone Call 80 Day Reminder 80 Day Reminder Letter, and Copy of 80 Days Letter, and Copy of the Survey the Survey 90 Day Phone 90 Day Phone 90 Days Survey Survey 1 Year Link to Claims Data Link to Claims Data

Figure 2: Flow of Intervention Activities for Phase 1, Control and COMPASS Participants

tailored to the hospital. Each control arm hospital brochure will include the PAC name, the PAC contact information and a tailored description of the post-acute "standard care" that the patient will receive at that hospital. This information will equip patients with information to fully inform them of the COMPASS Study and how this will impact them and what to expect from the hospital. The PAC will also explain that the patient will get a phone call in about three months asking

Application - IRB00035998

them to participate in a telephone survey and that they will get three reminder letters in the mail to remind them about the survey (Appendix 6-8). The PAC will record patient and caregiver contact information on the COMPASS enrollment form. In the COMPASS analytical database, the PAC will record the date, time and method (i.e. in person or over the phone) of informing the patient of the COMPASS Study, and confirm that the patient was given the brochure. As a pragmatic study, we anticipate that PACs may miss a patient (for example a patient may be missed on the weekends) and the patient will need to be enrolled retrospectively and notified of the study and mailed the brochure. The PAC will attempt to reach the patient over the phone to follow-up on the mailed brochure. The brochure also has contact information for the patient to call the study if they would like additional information.

As part of case ascertainment and consistent with the North Carolina Stroke Care Collaborative (NCSCC) methodologies to characterize all stroke admissions and processes of acute stroke care the PAC will complete the NCSCC Stroke Care Card (Appendix 9).

Patients will receive three letters in the mail to remind them about the 90 day survey and to provide educational information and resources from the American Stroke Association (Appendix 6-8). Although the 90 day phone survey will be relying on a Full HIPAA Authorization Waiver, the letter mailed to the patient at 80 days includes a statement on HIPAA to inform the patient on how they have been identified for the study and that agreeing to participate in the phone survey will be authorizing the use of identifiable health information and how that information will be used in the study. The 80 day letter will also include \$10 cash as a thank you gift for considering participation in the phone survey.

At 90 Days, stroke survivors will receive a phone call from the Carolina Survey Research Lab (CSRL). CSRL will follow a telephone script which includes consent (Appendix 10) and conduct blinded assessments (Appendix 23 and 24). If the patient prefers s/he can request that a proxy answer questions and provide verbal consent and HIPAA Authorization on her/his behalf. In the event contact is never made with the patient by phone or connection is lost (e.g. the number is not in service, no one answers the phone calls, call is answered but is disconnected prior to the researcher sharing the reason for calling, or there is loss of connection during the call) we will mail an abbreviated version of the survey with a letter explaining the survey purpose (Attachment 25). We will also include a self-addressed envelope with prepaid postage to the patient to gather responses via paper survey. This abbreviated survey contains the SIS-16, global health rating scale and blood pressure questions.

Approximately one year later the study will acquire claims data from Medicare, Medicaid, State Insurance Plan, and Blue Cross Blue Shield. We plan to use a HIPAA Waiver to acquire the data sets and along with this application we are asking for a waiver of signed consent to link all enrolled patients to the claims data sets.

#### **Phase 1: Patients in COMPASS-Intervention Hospitals**

In addition to the activities outlined in the Control Hospitals section above, patients who enter the study through a COMPASS Intervention hospital will receive: (1) a follow-up phone call 2 days after being discharged from the hospital, (2) a 7-14 day Advanced Practice Provider visit, (3) a follow-up 30 day phone call, and (4) a follow-up 60 day phone call. The structure and processes of this COMPASS intervention are consistent with the Center for Medicare and Medicaid (CMS) Transitional Care Management Codes. In essence the COMPASS study is an evaluation of the implementation of CMS recommendations for post hospital care coordination.

The process for determining Eligibility for COMPASS patients is identical to that of Control patients.

If the patient is eligible, they will be enrolled in a similar manner to that of the Control patients: The PAC will visit each patient in the hospital and give the patient a tailored handout about the COMPASS Study (Appendix 12). The information informs the patient that their hospital is participating in a state-wide study to evaluate best models of post stroke care. The patient will be informed if their hospital is in the usual care group or in the COMPASS intervention group. This brochure is tailored to the hospital. The PAC name and the PAC contact information will be provided on an appointment card. This information will equip patients with information to fully inform them of the COMPASS Study and how this will impact them and what to expect from the hospital. The PAC will also give an additional handout about COMPASS

Application - IRB00035998

intervention activities (Appendix 13), a Blood Pressure Log (Appendix 14) and Blood Pressure Handout (Appendix 15). The PAC will work with the patient to schedule follow-up visits with the patients Primary Care Physician (PCP) and the Advanced Practice Provider (APP) for the 7-14 day follow-up visit. The PAC will let the patient know they will be calling them in a couple of days for the 2-day follow-up phone call. The PAC will record patient and caregiver contact information on the COMPASS enrollment form. In the COMPASS analytical database, the PAC will record the date, time and method (i.e. in person or over the phone) of informing the patient of the COMPASS Study, and confirm that the patient was given the brochure. As a pragmatic study, we anticipate that PACs may miss a patient (for example a patient may be missed on the weekends) and the patient will need to be enrolled retrospectively and notified of the study and mailed the brochure. The PAC will attempt to reach the patient over the phone to follow-up on the mailed brochure. The brochure also has contact information for the patient to call the study if they would like additional information.

As part of case ascertainment and consistent with the North Carolina Stroke Care Collaborative methodologies to characterize all stroke admissions and processes of acute stroke care the PAC will complete the NC Stroke Care Card (Appendix 9). (Note: this is identical to the Control group).

At 2 days post- hospital discharge, the PAC will call the patient and discuss medication use, symptoms, and confirm (or schedule) follow-up appointments with the patients Primary Care Physician and the Advanced Practice Provider. The PAC will provide patient education to ensure they know about signs of a subsequent stroke. The script for the 2 day follow-up call is in Appendix 16.

Following the 2day call, the PAC will complete a disposition form (Appendix 34) to record if the call took place (yes/no) and if the call did not take place a categorical reason why the call did not take place. These questions are similar to what is acquired in claims data research. Use of data from this form will be done under a request for Full HIPAA Waiver for all patients who are enrolled in an intervention hospital.

Between 7 and 14 days, the patient will attend a follow-up visit with the advanced practice provider (APP). The PAC will also attend this visit. The goal of this visit is to create an individualized patient Care Plan and, if needed, make additional referrals for the patient. At this visit, the PAC will clinically assess the patient using the Post-stroke Functional Assessment (Appendix 17). Based on responses from this assessment, the PAC may also conduct the Caregiver Assessment (Appendix 18) with the patient's caregiver if the caregiver is present. The provider will assess the patient using the Post-stroke Advanced Practice Assessment (Appendix 19). Responses to these assessments will be used by the provider to develop an individualized patient Care Plan. These three assessments have been programmed into an electronic platform (eCare Application) to ease administration, assessments, data capture and development of the individualized patient Care Plan (eCare Plan) which will be conducted on an iPad. The tool will summarize the three assessments and make suggestions for the provider in creation of the individualized patient Care Plan (Appendix 20 is an example; the provider customizes these recommendations). As the decision-making authority in patient care, the final individualized patient Care Plan and any referrals are given by the provider. The PAC will review the Care Plan with the patient, establish preferences for care and coordinate referrals for services. A copy of the Care Plan will go forward to the patient's primary care provider and rehabilitation providers. The APP will send a summary of the visit and the Care Plan to the patient's primary care provider and rehabilitation providers. During this visit the patient will be asked for consent and HIPAA Authorization to use clinical data for future analyses (Appendix 21).

Following this clinic visit, the PAC will complete a clinic visit disposition form (Appendix 35) which records if the clinic visit was conducted (yes/no) and date of visit. This form also records which clinic forms were completed during the visit to determine to what extent the COMPASS intervention was implemented for quality improvement on processes and delivery of care. This form also summarizes care and community service recommendations, which were made for patient care and to record for quality improvement initiatives. This form includes yes/no and categorical responses similar to what is acquired in claims data. Use of data from this form will be done under a request for Full HIPAA Waiver for all patients who are enrolled in an intervention hospital.

Application - IRB00035998

At 30 and 60 days, patients will be called by the PAC to follow-up on their Care Plan. The PAC will ask the patient if they are having any challenges with implementing the care and treatment plans that their health providers have given them (Appendix 22).

Patients will also receive three letters in the mail to remind them about the 90 day survey and to provide educational information and resources from the American Stroke Association (Appendix 6-8). Although the 90 day phone survey will be relying on a Full HIPAA Authorization Waiver, the letter mailed to the patient at 80 days includes a statement on HIPAA to inform the patient on how they have been identified for the study and that agreeing to participate in the phone survey will be authorizing the use of identifiable health information and how that information will be used in the study. The 80 day letter will also include \$10 cash as a thank you gift for considering participation in the phone survey. (Note: this is identical to the Control group).

At 90 Days, stroke survivors will receive a phone call from the Carolina Survey Research Lab (CSRL). CSRL will follow a telephone script which includes consent (Appendix 10) and conduct blinded assessments (Appendix 23 and 24). If the patient prefers s/he can request that a proxy answer questions and provide verbal consent and HIPAA Authorization on her/his behalf. In the event contact is never made with the patient by phone or connection is lost (e.g. the number is not in service, no one answers the phone calls, call is answered but is disconnected prior to the researcher sharing the reason for calling, or there is loss of connection during the call) we will mail an abbreviated version of the survey with a letter explaining the survey purpose (Attachment 25). We will also include a self-addressed envelope with prepaid postage to the patient to gather responses via paper survey. This abbreviated survey contains the SIS-16, global health rating scale and blood pressure questions. (Note: this is identical to the Control group)

Approximately one year later the study will acquire claims data from Medicare, Medicaid, State Insurance Plan, and Blue Cross Blue Shield. We plan to use a HIPAA Waiver to acquire the data sets and along with this application we are asking for a waiver of signed consent to link all enrolled patients to the claims data sets. (Note: this is identical to the Control group).

## Phase 2: COMPASS-Intervention & COMPASS-Sustain Hospitals

Hospitals which were randomized to the control-arm in Phase 1 of the study will be encouraged to cross over to provide the COMPASS Intervention during Phase 2 of the study. Hospitals that were randomized to the COMPASS Intervention-arm during Phase 1 of the study will be encouraged to continue providing all of the COMPASS Intervention to eligible patients (Sustain Sites). Both the Intervention and the Sustain Sites will provide the same intervention as described in this section. This intervention is nearly identical to the Phase 1 Intervention. Minor changes were made in order to streamline some of the intervention activities based on lessons-learned from Phase 1. The structure, however, remains unchanged: Patients who enter the study through a participating hospital will receive: (1) a follow-up phone call 2 days after being discharged from the hospital, (2) a 7-14 day Advanced Practice Provider visit, (3) a follow-up 30 day phone call, and (4) a follow-up 60 day phone call.

The process for determining Eligibility for patients is identical to Phase 1 of the study: Prior to hospital discharge, the Post-Acute Coordinator (PAC) will identify stroke and TIA patients for eligibility using the Eligibility Screening Form to assist in determining eligibility (Appendix 3). Determining eligibly will involve daily review of stroke admissions to the hospital by screening the electronic medical records. This will be done under Limited HIPAA Waiver.

If eligible, the patient will be enrolled, a COMPASS ID is assigned and the PAC will fill out the Enrollment Form which has been streamlined for Phase 2 of the study (Appendix 38). For those not eligible, no further information is collected and a COMPASS Identification number is not assigned. Enrollment will be done under a Full HIPAA Waiver.

Once the patient is enrolled, the patient will be notified of the study. The PAC will visit each patient in the hospital and give the patient a tailored, Phase 2 handout about the COMPASS Study (Appendix 36 & Appendix 37). Like Phase 1 of the study, the information informs the patient that their hospital is participating in a state-wide study to evaluate best

Application - IRB00035998

models of post stroke care. The patient will be informed their hospital is providing the COMPASS intervention. The PAC name and the PAC contact information will be provided on an appointment card. This information will equip patients with information to fully inform them of the COMPASS Study and how this will impact them and what to expect from the hospital. The PAC will also give an additional handout about COMPASS intervention activities (Appendix 13), a Blood Pressure Handout and Log (Appendix 14). The PAC will work with the patient to schedule follow-up visits with the patients Primary Care Physician (PCP) and the Advanced Practice Provider (APP) for the 7-14 day follow-up visit. The PAC will let the patient know they will be calling them in a couple of days for the 2-day follow-up phone call. In the COMPASS data application, the PAC will record the date, time and method (i.e. in person or over the phone) of informing the patient of the COMPASS Study, and confirm that the patient was given the brochure. As a pragmatic study, we anticipate that PACs may miss a patient (for example a patient may be missed on the weekends) and the patient will need to be enrolled retrospectively and notified of the study and mailed the brochure. PACs are encouraged to notify patients over the phone as follow-up on the mailed brochure. The brochure also has a toll-free study phone number for patients to call the study if they would like additional information or to opt-out of the study.

In Phase 2, hospitals will not be <u>required</u> to complete the North Carolina Stroke Care card (Appendix 9), however, this card will be made available to hospitals if they find it beneficial.

**At 2 days post- hospital discharge, the PAC will call the patient** and discuss medication use, symptoms, and confirm (or schedule) follow-up appointments with the patients Primary Care Physician and the Advanced Practice Provider. The PAC will provide patient education to ensure they know about signs of a subsequent stroke. The script for the 2 day follow-up call is in Appendix 16. **(Note this is identical to Phase 1 Intervention)** 

Following the 2day call, the PAC will complete a disposition form (Appendix 34) to record if the call took place (yes/no) and if the call did not take place a categorical reason why the call did not take place. These questions are similar to what is acquired in claims data research. Use of data from this form will be done under a request for Full HIPAA Waiver for all patients who are enrolled in an intervention hospital. (Note this is identical to Phase 1 Intervention)

Between 7 and 14 days, the patient will attend a follow-up visit with the advanced practice provider (APP). The PAC will also attend this visit. The goal of this visit is to create an individualized patient Care Plan and, if needed, make additional referrals for the patient. At this visit, the PAC will clinically assess the patient using the Post-stroke Functional Assessment (Appendix 17). Based on responses from this assessment, the PAC may also conduct the Caregiver Assessment (Appendix 18) with the patient's caregiver if the caregiver is present. The provider will assess the patient using the Post-stroke Advanced Practice Assessment (Appendix 19). Responses to these assessments will be used by the provider to develop an individualized patient Care Plan. These three assessments have been programmed into an electronic platform (eCare Application) to ease administration, assessments, data capture and development of the individualized patient Care Plan (eCare Plan) which will be conducted on an iPad. The tool will summarize the three assessments and make suggestions for the provider in creation of the individualized patient Care Plan (Appendix 20 is an example: the provider customizes these recommendations). As the decision-making authority in patient care, the final individualized patient Care Plan and any referrals are given by the provider. The PAC will review the Care Plan with the patient, establish preferences for care and coordinate referrals for services. A copy of the Care Plan will go forward to the patient's primary care provider and rehabilitation providers. The APP will send a summary of the visit and the Care Plan to the patient's primary care provider and rehabilitation providers. During this visit the patient will be asked for consent and HIPAA Authorization to use clinical data for future analyses (Appendix 21). (Note this is identical to Phase 1 **Intervention**)

Following this clinic visit, the PAC will complete a clinic visit disposition form (Appendix 35) which records if the clinic visit was conducted (yes/no) and date of visit. This form also records which clinic forms were completed during the visit to determine to what extent the COMPASS intervention was implemented for quality improvement on processes and delivery of care. This form also summarizes care and community service recommendations, which were made for patient care and to record for quality improvement initiatives. This form includes yes/no and categorical responses similar to what is acquired in claims data. Use of data from this form will be done under a request for Full HIPAA Waiver for all patients who are enrolled in an intervention hospital. (Note this is identical to Phase 1 Intervention)

At 30 and 60 days, patients will be called by the PAC to follow-up on their Care Plan. The PAC will ask the patient if they are having any challenges with implementing the care and treatment plans that their health providers have given them (Appendix 22). (Note this is identical to Phase 1 Intervention)

Patients will also receive three letters in the mail to remind them about the 90 day survey and to provide educational information and resources from the American Stroke Association (Appendix 6-8). Although the 90 day phone survey will be relying on a Full HIPAA Authorization Waiver, the letter mailed to the patient at 80 days includes a statement on HIPAA to inform the patient on how they have been identified for the study and that agreeing to participate in the phone survey will be authorizing the use of identifiable health information and how that information will be used in the study. The 80 day letter will also include \$10 cash as a thank you gift for considering participation in the phone survey. (Note this is identical to Phase 1)

At 90 Days, stroke survivors will receive a phone call from the Carolina Survey Research Lab (CSRL). CSRL will follow a telephone script which includes consent (Appendix 10) and conduct blinded assessments (Appendix 23 and 24). If the patient prefers s/he can request that a proxy answer questions and provide verbal consent and HIPAA Authorization on her/his behalf. In the event contact is never made with the patient by phone or connection is lost (e.g. the number is not in service, no one answers the phone calls, call is answered but is disconnected prior to the researcher sharing the reason for calling, or there is loss of connection during the call) we will mail an abbreviated version of the survey with a letter explaining the survey purpose (Attachment 25). We will also include a self-addressed envelope with prepaid postage to the patient to gather responses via paper survey. This abbreviated survey contains the SIS-16, global health rating scale and blood pressure questions. (Note this is identical to Phase 1)

Approximately 6-months later the study will acquire claims data from Medicare, Medicaid, State Insurance Plan, and Blue Cross Blue Shield. We plan to use a HIPAA Waiver to acquire the data sets and along with this application we are asking for a waiver of signed consent to link all enrolled patients to the claims data sets. (Note, this is identical to Phase 1 with the exception we are doing 6 months of claims data follow-up in Phase 2. As a reminder, in Phase 1, the study is doing 12 months of follow-up.)

#### **Phase 1 Only: Caregivers Outcomes Survey**

COMPASS Study team will mail the patient's caregiver a letter (Appendix 26), and the Caregiver Survey (Appendix 27). Non-respondents will be mailed a second letter (Appendix 29) with the survey (Appendix 27). If the caregiver still does not respond they will receive a reminder telephone call from UNC Carolina Survey Research Lab. (Note, Phase 2 will not include a Caregiver Outcomes Survey)

#### Phase 1 & Phase 2: Community-Engagement

This is a community-engaged study. Patients, family caregivers, and others stakeholders will be involved in all phases of the research process. These community members will be engaged in non-research activities (e.g., revising study materials for clarity) as well as research activities (e.g., participating in focus groups). By design, community-engaged research requires decision making by many stakeholders and frequent IRB amendments. For clarity and oversight purposes we have submitted a separate IRB (PCORI Stakeholder Interviews: IRB00028495; Appendix 31) for research activities involving stakeholders.

#### **Phase 1 Only: Implementation Analysis**

We will be asking participating staff at implementing sites (approximately 20 PACs and COMPASS team members) to agree to have their responses on the Bi-weekly Implementation Calls and surveys recorded and transcribed and analyzed to better understand the process of implementing the COMPASS Care Model. We will be asking participating staff at implementing sites (approximately 40 therapy care providers and COMPASS team members) to agree to have their responses on the Bi-weekly Home Health and Outpatient Calls and surveys recorded and transcribed and analyzed to

Application - IRB00035998

better understand the process of implementing the COMPASS Care Model. We will also be asking study staff COMPASS Director of Implementation and members of the Implementation Committee for individual semi-structured interviews. Additional detail to this study activity is provided in Appendix 33.

## **Data Collection and Outcome Measures**

## Patient Participant Study Outcomes (Phase 1 and 2):

| | Measure | Assessment(s) | When Collected | Appendix |
|---|---|---|---|---|
| Primary<br>Outcome | Physical Function | Stroke Impact Scale (SIS-16) | @90 days,<br>consenting patients<br>asked by CSRL | 23 |
| Secondary<br>Outcome | Self-rated General Health | A question rating<br>health on a 5-point<br>scale & a question on<br>perception of health<br>improvement | @90 days,<br>consenting patients<br>asked by CSRL | 24 |
| Secondary<br>Outcome | Disability and<br>Dependence | Modified Rankin Scale | @90 days,<br>consenting patients<br>asked by CSRL | 24 |
| Secondary<br>Outcome | Physical Activity | Three questions which ask about time spent walking | @90 days,<br>consenting patients<br>asked by CSRL | 24 |
| Secondary<br>Outcome | Depression | Patient Health Questionnaire (PHQ-2) Note: these items do not ask about suicidal thoughts or actions | @90 days,<br>consenting patients<br>asked by CSRL | 24 |
| Secondary<br>Outcome | Cognition | MOntreal Cognitive<br>Assessment (MOCA)<br>Mini | @90 days,<br>consenting patients<br>asked by CSRL | 24 |
| Secondary<br>Outcome | Medication Adherence | 4-item Morisky<br>Green-Levine Scale | @90 days,<br>consenting patients<br>asked by CSRL | 24 |
| Secondary<br>Outcome | Secondary Prevention<br>Self-Monitoring of BP | By asking: "Do you check your blood pressure at home?" | @90 days,<br>consenting patients<br>asked by CSRL | 24 |
| Secondary<br>Outcome | Blood Pressure<br>Management<br>Effectiveness | For those who check<br>BP at home, we ask:<br>"Is your blood pressure<br>less than 140/90 most<br>of the time?" | @90 days,<br>consenting patients<br>asked by CSRL | 24 |
| Secondary<br>Outcome | Falls and Hospitalization* | Questions to capture: Number of falls, injuries, and hospitalizations *Note: Note: Outcome is binary variable of Fall either Yes or No. Hospitalizations, injuries and number of falls were collected but were not used in the analyses | @90 days,<br>consenting patients<br>asked by CSRL | 24 |

| Secondary<br>Outcome | Fatigue | PROMIS Fatigue<br>Instrument – Adult<br>Short Form 4A | @90 days,<br>consenting patients<br>asked by CSRL | 24 |
|---|---|---|---|---|
| Secondary<br>Outcome | Satisfaction with care | Questions on how the patient felt about care and treatment from health care providers. | @90 days,<br>consenting patients<br>asked by CSRL | 24 |
| Exploratory Aim | Use of Community<br>Resources | By asking: "Since<br>discharge from the<br>hospital, have you used<br>services such as Senior<br>Services, Meals on<br>Wheels, in-home aides,<br>or stroke survivor or<br>caregiver support<br>groups?" | @90 days,<br>consenting patients<br>asked by CSRL | 24 |
| Data collected to support the operations of the trial. | Initial Presentation Data | Hospital arrival and Mode of arrival, Ambulatory status prior to admission, Diagnosis at admission, NIHSS, Imaging performed, etc. | Entered into the COMPASS Database by the hospital | 9 |
| Data collected to support the operations of the trial. | Demographic Data | DOB, Race, Gender,<br>Insurance, Medical<br>History, Medication,<br>etc. | Entered into the COMPASS Database by the hospital | 9 |
| Data collected to support the operations of the trial. | t-PA Data | Time t-PA was initiated, BP and Glucose levels, bleeding complications, etc. | Entered into the COMPASS Database by the hospital | 9 |
| Data collected to support the operations of the trial. | In-hospital Data | Admission data, secondary prevention counseling, treatment, lipid profile, medications, treatments, etc. | Entered into the COMPASS Database by the hospital | 9 |
| Data collected to support the operations of the trial. | Discharge Data | Resources and stroke education materials, assess for rehabilitation, ambulatory status, Rankin Score, final diagnosis, discharge disposition, ICD-10 data, etc. | Entered into the COMPASS Database by the hospital | 9 |

# March 19, 2021 Application - IRB00035998 Patient Participant Study Outcomes (Phase 2):

| Ancillary Study General Heath and PROMIS Global-10 @90 days, consenting 23 Function patients asked by CSRL | | Measure | Assessment(s) | When Collected | Appendix |
|---|---|---|---|---|---|
| | Ancillary Study | | PROMIS Global-10 | patients asked by | 23 |

# March 19, 2021 Application - IRB00035998 Caregiver Participant Study Outcomes (Phase 1 only):

| | Measure | Assessment(s) | When Collected | Appendix |
|---|---|---|---|---|
| Secondary<br>Outcome | Caregiver Burden | Modified Caregiver<br>Strain Index | @95 days, mailed to the caregiver | 27 |
| Data collected to support the operations of the trial. | Relation to stroke patient | Relation to stroke patient | @95 days, mailed to<br>the caregiver | 27 |
| Data collected to support the operations of the trial. | Demographics | Age, Gender, Race | @95 days, mailed to the caregiver | 27 |
| Data collected to support the operations of the trial. | Primary Caregiver | Are you the primary caregiver | @95 days, mailed to<br>the caregiver | 27 |
| Data collected to support the operations of the trial. | Length of Caregiving service | How long have you<br>been providing care?<br>How many hours per<br>day do you spend<br>providing care?<br>Do others help provide<br>care? | @95 days, mailed to the caregiver | 27 |
| Data collected to support the operations of the trial. | Type of caregiving activities | Type of caregiving activities | @95 days, mailed to the caregiver | 27 |
| Data collected to support the operations of the trial. | Awareness and use of<br>Community Resources | Awareness and use of<br>Community Resources | @95 days, mailed to the caregiver | 27 |
| Data collected to<br>support the<br>operations of the<br>trial. | Self-rated General<br>Health | Compared to others your age, how would you rate your health using a scale of 1 to 5, with 1 being "Poor" and 5 being "Excellent?" | @95 days, mailed to the caregiver | 27 |
| Data collected to support the operations of the trial. | Accessed the COMPASS Website | Have you explored the information on the COMPASS website | @95 days, mailed to the caregiver | 27 |

## Study outcomes collected and linked to insurance claims data (Phase 1 & Phase 2):

| | Measure | Assessment(s) | When Collected | Appendix |
|---|---|---|---|---|
| Secondary<br>Outcome | Readmissions | 30-day, 90-day and 1-<br>year all-cause<br>readmission | Approximately 1 year post-stroke in Phase 1 | This will be collected<br>via Administrative<br>Claims Data sets from<br>Medicare, Medicaid,<br>and Blue Cross Blue<br>Shield |
| Secondary<br>Outcome | Mortality Mortal | ity | Approximately 1 year post-stroke in Phase 1 | This will be collected<br>via Administrative<br>Claims Data sets from<br>Medicare, Medicaid,<br>and Blue Cross Blue<br>Shield |
| Secondary<br>Outcome | Emergency<br>Department (ED)<br>Visits | Number of patient<br>emergency department<br>visits | Approximately 1 year post-stroke in Phase 1 | This will be collected via Administrative Claims Data sets from Medicare, Medicaid, and Blue Cross Blue Shield |
| Secondary<br>Outcome | Admissions to skilled<br>nursing facilities and<br>inpatient rehabilitation<br>facilities | Number of patient<br>admissions and<br>number of days in to<br>skilled nursing<br>facilities, and number<br>of patient admissions<br>to inpatient<br>rehabilitation facilities | Approximately 1 year post-stroke in Phase 1 | This will be collected<br>via Administrative<br>Claims Data sets from<br>Medicare, Medicaid,<br>and Blue Cross Blue<br>Shield |
| Secondary<br>Outcome | Use of transitional billing codes | Use of Transitional Care Management (TCM) billing codes and Chronic Care Management (CCM) billing codes | Approximately 1 year post-stroke in Phase 1 | This will be collected via Administrative Claims Data sets from Medicare, Medicaid, and Blue Cross Blue Shield |

## **Clinical Data collection:**

• We will collect clinical data to inform the patient's individualized care plan that will be routine for implementing transitional care, and would like to keep this data for future analyses:

| - Caribrioliai ( | Measure | Assessment(s) | When Collected | Appendix |
|---|---|---|---|---|
| Data collected to<br>support the<br>operations of the<br>trial. | Neurological Status and<br>Deficits | Post Stroke Advanced<br>Practice Assessment | 7-14 Day Visit | 19 |
| Data collected to support the operations of the trial. | Stroke Complications | Post Stroke Advanced<br>Practice Assessment | 7-14 Day Visit | 19 |
| Data collected to<br>support the<br>operations of the<br>trial. | Stroke Risk Factor<br>Management | Post Stroke Advanced<br>Practice Assessment | 7-14 Day Visit | 19 |
| Data collected to support the operations of the trial. | Lifestyle Coaching | Post Stroke Advanced<br>Practice Assessment | 7-14 Day Visit | 19 |
| Data collected to<br>support the<br>operations of the<br>trial. | Medication Access and Use | Post Stroke Functional<br>Assessment | 7-14 Day Visit | 17 |
| Data collected to support the operations of the trial. | Knowledge of Stroke<br>Risk Factors | Post Stroke Functional<br>Assessment | 7-14 Day Visit | 17 |
| Data collected to support the operations of the trial. | Self-rated General<br>Health | Post Stroke Functional<br>Assessment | 7-14 Day Visit | 17 |
| Data collected to support the operations of the trial. | Mobility | Post Stroke Functional<br>Assessment | 7-14 Day Visit | 17 |
| Data collected to<br>support the<br>operations of the<br>trial. | Falls and<br>Hospitalizations | Post Stroke Functional<br>Assessment | 7-14 Day Visit | 17 |
| Data collected to<br>support the<br>operations of the<br>trial. | Social and Caregiver<br>Support | Post Stroke Functional<br>Assessment | 7-14 Day Visit | 17 |
| Data collected to<br>support the<br>operations of the<br>trial. | Activities of Daily<br>Living | Post Stroke Functional<br>Assessment | 7-14 Day Visit | 17 |
| Data collected to support the operations of the trial. | Home Health,<br>Outpatient services | Post Stroke Functional<br>Assessment | 7-14 Day Visit | 17 |

| Application - IRB000 | 035998 | | | |
|---|---|---|---|---|
| Data collected to support the operations of the trial. | Durable Medical<br>Equipment | Post Stroke Functional<br>Assessment | 7-14 Day Visit | 17 |
| Data collected to support the operations of the trial. | Living Will | Post Stroke Functional<br>Assessment | 7-14 Day Visit | 17 |
| Data collected to support the operations of the trial. | Relation | Caregiver Assessment | 7-14 Day Visit | 18 |
| Data collected to support the operations of the trial. | Demographics | Caregiver Assessment | 7-14 Day Visit | 18 |
| Data collected to support the operations of the trial. | Caregiving activities | Caregiver Assessment | 7-14 Day Visit | 18 |
| Data collected to support the operations of the trial. | Self-rated General<br>Health | Caregiver Assessment | 7-14 Day Visit | 18 |
| Data collected to support the operations of the trial. | Stress | Caregiver Assessment | 7-14 Day Visit | 18 |
| Data collected to support the operations of the trial. | Signs of a stroke | Caregiver Assessment | 7-14 Day Visit | 18 |

## **Analytical Plan**

As described above, this pragmatic trial utilizes a cluster randomized design with 41 hospitals being randomized to receive the COMPASS intervention (N=20) or control (N=20) in Phase 1. In Phase 2, the control group hospitals will be rolled into the intervention (Figure 1). All stroke patients who are discharged directly home from one of the randomized hospitals will be included in the intention-to-treat analyses. Analyses will be performed at the individual (patient) level, with adjustments for hospital and/or patient level characteristics to control for possible correlations of patients within hospitals.

We used two stratification factors in randomization: annual stroke patient volume per hospital (3 levels: <100, 100-299, 300+ patients) and whether the hospital is a primary stroke center (Yes/No). Thus, there will be a total of 6 strata. We will use a random permuted block design with block size of two; within each stratum we will randomize an even number of hospitals. This will allow us to maintain balance between the treatment groups while also protecting the validity of the randomization process. Study team involved with site selection will not have access to the randomization schedule which will be held by Dr. Walter Ambrosius. Likewise, Dr. Ambrosius will not be involved in site selection. Although patients in the intervention cannot be blinded to their group assignment, interviewers gathering outcome data will be blinded. Our estimated sample size will permit pre-specified subgroup analyses by race, gender, age, stroke severity and insurance status.

For the primary aim, the primary endpoint is the Stroke Impact Scale (SIS-16) measured 90 days post-stroke. The secondary aims include the Modified Caregiver Strain Index at 90 days; 30- and 90-day all-cause readmissions; and mortality, health care utilization, continuity of care, utilization of transitional care, and medication adherence, all measured 1 year after index discharge. In addition, analyses by race, gender, age, stroke severity and insurance status will determine if there is evidence of heterogeneity of the intervention effect across any subgroups. Finally, for the two exploratory aims, we will (1) examine hospital-level measures of stroke care quality indicators in the COMPASS hospitals, and (2) compare administrative claims outcomes and post-acute stroke performance outcomes between COMPASS patients in Phase 1 (intervention phase) and Phase 2 (sustainability phase).

Since the primary endpoint (SIS-16) is measured on a continuous scale, we will use a mixed model to compare the COMPASS and control groups. Although the stratified randomization of hospitals should balance most important hospital-level characteristics between groups, since imbalances may exist between groups on patient-level characteristics, we propose to include both fixed and random effects in this mixed model. The first model will include two fixed effects: stratum (1 to 6) and the intervention effect (COMPASS vs. control) and one random effect: hospital. This additive model can be written as:  $Y_{ijk} = \mu + \gamma_k + \alpha_j + \beta_{k(j)} + \epsilon_{i(jk)}$ , where  $Y_{ijk}$  is the outcome (i.e. SIS at 90 days) measured on the  $i^{th}$  patient, under the  $j^{th}$  intervention (j=1 (COMPASS), 2(Control) in the  $k^{th}$  hospital;  $\mu$  is the grand mean;  $\gamma_k$  is the stratum (1 to 6) for hospital k;  $\alpha_j$  is the fixed treatment effect for group j (COMPASS/CNT);  $\beta_{k(j)}$  is the random effect of the  $k^{th}$  hospital nested within the exposure group; and  $\epsilon_{i(jk)}$  is the error term for the  $i^{th}$  patient nested within the treatment group and hospital. Other fixed effects can be added at the patient level (e.g. age, gender, race, stroke severity, or SES) for sensitivity analyses. The random hospital effect allows the possibility of correlated observations (patients) within hospitals. Of primary interest is the treatment effect ( $\alpha_i$ ), which indicates difference in the dependent variable (SIS-16) between groups.

After we fit our primary model, we will consider other models that may include more patient-level and hospital-level characteristics. For instance, since some patients may be transferred to a different hospital before being discharged home, we can include a yes/no variable on that point. Although hospitals will be stratified pre-randomization based on stroke volume, we can include a hospital-level covariate for the total number of stroke patients discharged home for each hospital. With 40 clusters (of the 41 hospitals, 2 were randomized together) included, we will be able to add other cluster-level covariates to the model if needed.

For secondary aims and outcomes measured on a continuous scale, we will use a similar approach as above (i.e. for the Modified CSI). For binary outcomes such as whether a patient is readmitted within 30 or 90 days (Secondary Aim 2), we will use mixed logit models to fit the relationship between the intervention and outcome measures. The mixed logit model is similar to the mixed model presented above but uses a logit link in a generalized linear mixed model. Software is

Application - IRB00035998

readily available (e.g., SAS PROC GLIMMIX) that can fit these models. The mixed logit model approach will also allow a mixture of fixed and random effects to be included as in the mixed model above. Other Secondary Aim 2 variables will be analyzed using a mixed model or alternatively generalized linear mixed models (e.g., Poisson regression [with overdispersion] for the number of inpatient days).

We will examine 1-year mortality rates as a binary outcome and use the methods described above to compare groups, but we will also consider mortality as a time-to-event outcome and compare groups using Cox proportional hazards models. In these survival analysis models, the treatment indicator will be included as the primary independent variable and the stratum included as stratification factor.

## **Human Subjects Protection**

COMPASS is implementation of CMS recommendations for post hospital care coordination. COMPASS is using a pragmatic, randomized controlled trial approach because it facilitates consistent delivery in post-acute stroke care management. Hospitals are being asked to implement the COMPASS Intervention as a new standard of care for all stroke patients. Because specific informed consent would not typically be sought in a clinical setting, stroke patients at the participating hospitals will not have the option to consent to (or opt out of) the site intervention. It is unlikely that our study can seamlessly implement the new models of transitional care in routine clinical care delivery if the traditional informed-consent process for research participation is required. COMPASS will incorporate an Integrated Consent Model for Pragmatic Trials.<sup>31</sup> In this model, the "consent" will inform the patient that they are seeking care in a hospital that has been randomized to provide their usual standard of post hospital care or a hospital that is going to incorporate the COMPASS model of post hospital care. This integrated consent model simply incorporates information about the hospital randomization process and whether their hospital is randomized to usual standard of care or the COMPASS intervention.

A stroke coordinator (PAC), who is a hospital employee, will visit patients in the control sites and in the intervention sites prior to hospital discharge and provide patients with a tailored study brochure. The PAC will review the content of the informational brochure (Appendix 5 and Appendix 12) and inform patients that the hospital is participating in a statewide study to evaluate the best way to provide post-acute services after hospitalization for a stroke. The PAC will also inform the patient that there are many ways to care for patients after they leave the hospital and we are not sure which model is best.

The PAC can answer any questions that the patient has regarding this conversation and provide their contact information, the COMPASS toll-free phone number and website as a reference for additional information. For additional assurance, the study will ask PACs to document into the COMPASS Study data portal the date and time the patient was informed. The goal of this study is to capture all patients discharged directly home. In the event that a patient is discharged on a weekend or before the PAC is able to visit the patient, the PAC will make a call attempt to the patient to inform them of the hospital study and then the PAC will mail the brochure to the patient's preferred mailing address. The PAC will also document in the COMPASS Study data portal that the patient was called and the brochure was mailed to the patient.

Our protocol and process for consent reflects this integrated model. All enrolled stroke patients will be told that the hospital is enrolled in a state-wide initiative to evaluate and improve post-acute stroke care:

- Phase 1 & 2 Consent for the Clinical Data (COMPASS Intervention Patients only at 7-14 Day APP Visit): A signed consent and HIPAA Authorization (collected on the iPad eCare Application or, if the PAC prefers, this can be conducted on paper) to use data collected from patient during clinical care for research purposes (i.e., to better understand recovery and factors that might influence response to the COMPASS intervention).
- Phase 1 & 2 Consent for the 90 day phone survey for patients: A verbal consent over the phone, performed by the UNC Carolina Survey Research Laboratory. COMPASS will rely on the Full HIPAA Waiver for this phone survey, however we have included in the 80 day reminder letter, information on HIPAA for the patient to make an informed decision on if they would like to participating in the phone survey.
- <u>Phase 1 only Consent for the 95 day paper survey mailed to caregivers: A returned, completed survey constitutes consent.</u>
- Phase 1 & 2 Consent for the Claims Data Analysis: A waiver of consent is requested as this activity (1) is low risk, (2) does not affect the right and welfare of patients, and (3) cannot be practically carried out without this waiver.

Minimal/No Risk Intervention: Participation in the COMPASS study does not expose patients to any additional risks and therefor it is a minimal-risk or no-risk intervention. The COMPASS model and intervention activities are not experimental. COMPASS is evidence-based, and considered best practice for management of post-acute care. CMS supports the delivery of these types of post-acute services and has implemented billing codes (TCM and CCM) to actualize implementation of these services. Hospitals which participate in the COMPASS Study will be asked to implement at the hospital-level these evidence-based services into the systematic delivery of post-acute care to all stroke patients. The COMPASS Study will determine effectiveness of this model on self-reported functional outcomes.

In order to minimize potential differences in loss to follow-up between the control and intervention groups we will send reminder letters (as described in the intervention section) to both control and intervention groups. These letters will include resources from the American Stroke Association (ASA). We will include a refrigerator magnet to remind them that we will call stroke survivors and survey caregivers at 90 days to assess outcomes.

#### **Informed Consent**

As a pragmatic trial, our eligibility and outcomes assessment will include all patients discharged home from participating hospitals who are adopting the non-experimental, evidence-based intervention as the new model of care. Our approach has been to minimize patient risk and maximize participation by providing an informational brochure to patients and their families during the hospital stay (or informing by mail), and allow them to opt out of the follow-up phone call at 90 days.

Patients will not be asked for consent to participate at the hospital. It is unlikely that our study can seamlessly implement the new models of transitional care in routine clinical care delivery if the traditional informed-consent process for research participation is required. COMPASS will incorporate an Integrated Consent Model for Pragmatic Trials.<sup>31</sup> In addition, during focus groups, patient stakeholders informed us that this would not be the optimal time for informed consent. Patients are often overwhelmed during the hospital stay as they are introduced to a large amount of new information in addition to processing the recent health event (stroke). This was described during the focus group as an emotional and difficult time. Patient stakeholders reported that they are asked to sign a lot of paperwork during the stay and at discharge. According to our stakeholders, the process can be confusing. The COMPASS Study team did not want to add additional burden on the patients and study staff to gain informed consent at the hospital for this low/no risk study.

Figure 3 depicts the flow of Control (left and during Phase 1 only) and COMPASS Intervention (right during Phase 1 and 2) activities and how research activities are covered at each step (center).

A HIPAA Waiver which is included as a part of this application is used to confirm eligibility, enrollment, and collect NCSCC Registry Stroke Card data, contact the participants with letters and surveys.

Consent for the Clinical Data (COMPASS Intervention Arm only): At the 7-14 day APP visit, COMPASS participants will be asked for written informed consent and HIPAA Authorization for the study to keep clinical data (2 day phone call, 7-14 day visit, 30 day phone call and 60 day phone call) for future analyses (e.g. follow-up with recommendations for care, demographic and clinical factors that predict follow up and outcomes in the intervention arm). The post-acute coordinator will ask for informed consent and will use the eCare Application on the iPad to capture signature. The abbreviated consent and HIPAA Authorization contains the following elements of informed consent: the purpose of the study; the types of clinical data that will be captured and analyzed; explaining how information the patient provides will be used; data



Figure 3: HIPAA Waiver and Consent of COMPASS

will be kept confidential and secure and will abide to HIPAA regulations; a reminder that providing consent is voluntary; identification of funding agency, study PI, and institution; contact information should the patient want to withdraw

Application - IRB00035998

(Appendix 21). Patient will use his/her finger to sign and date on the iPad for capture of written signature. (A paper version of the consent form is also available.) The PAC who will be conducting the consent process will also sign and date. A hard copy of consent script will be printed out for the patient to take with them. If the patient declines consent, this will also be noted. In order to not disrupt the clinical work-flow, consent will be collected during the visit either inbetween assessments or at the end of the visit.

Consent for the 90 Day Phone Survey for Patients (All Patients): All stroke patients (or representing proxies) will consent to (or decline) participation in the survey of outcomes. COMPASS will rely on the Full HIPAA Waiver for this phone survey, however we have included in the 80 day reminder letter, information on HIPAA for the patient to make an informed decision on if they would like to participating in the phone survey. Verbal consent at the introduction of the telephone survey should adequately protect the individuals' rights of patient participants. Study-eligible patients are discharged home, and thus proxy support is unlikely to be needed. If the patient prefers a proxy to complete the survey, the patient can ask the proxy to support them in responding. We will record whether the data are provided by the proxy or the patient.

Consent for the 95 Day Paper Survey Mailed to Caregivers (<u>All Caregivers</u>): Caregivers will be asked to respond to a paper survey questionnaire. This questionnaire does not have any questions about the patient, therefore we are not asking for permission from patients to send this survey to caregivers. Response to the questionnaire will be considered consent and HIPAA Authorization to participate in the study.

Consent for the Claims Data Analysis (<u>All Patients</u>): We will acquire claims data sets using a HIPAA waiver. We will link patient data collected at study enrollment (this data collected is under a HIPAA Waiver) to the claims data. A waiver of consent is requested and included in this application as this activity (1) is low risk, (2) does not affect the right and welfare of patients, and (3) cannot be practically carried out without this waiver.

**Consent for Engagement Activities:** Consent for research-related engagement activities (i.e. focus groups) will be covered under separate IRBs (PCORI Stakeholder Interviews: IRB00028495; Appendix 31).

Consent for Implementation Analysis (Phase 1 only): Additional detail to this study activity is provided in Appendix 33

We will be asking participating staff at implementing sites (approximately 20 PACs, 40 therapy providers and COMPASS team members) to agree to have their responses on the Bi-weekly Implementation Calls and surveys recorded and transcribed and analyzed to better understand the process of implementing the COMPASS Care Model:

- Some of these calls and surveys have been previously recorded because our sites started launching in June 2016 and the funding for the CTSI Implementation Analysis will not start until April 2017. Retrospective recordings of the calls will be covered under a Waiver of Consent granted by the IRB as this is low-risk to the call participants, this data is needed to run this research analysis and because gaining consent would be difficult considering that there has been some staff turnover at some of our participating sites.
- For any future calls and surveys we will gain consent of participants by informing them that the (1) the call/survey is being recorded and (2) responses may be used for research to analyze implementation of COMPASS program, and (3) responses will be aggregated to maintain confidentiality (meaning any identifying information will be removed prior to publicly using any responses/data). This will require Waiver of Signature since by participating they are providing implicit consent.

We will also be asking study staff COMPASS Director of Implementation and members of the Implementation Committee for individual semi-structured interviews for which we will gain verbal approval. We estimate that we will interview her for 3 hours. For her time, we will offer compensation of \$200 for her participation in this research.

## **Confidentiality and Privacy**

#### **Overview**

The Principal Investigators and Co-Investigators will ensure the privacy and confidentiality of all study data. All COMPASS Study Investigators and team members are required to complete a yearly HIPAA training and will have research training from CITI (or its equivalent research training).

High-levels of security have been put in place to ensure confidential and secure collection, storage and transfer of data. Patient-level data will be stored on secure servers in four different locations, three of which are at UNC-CH and one at Wake Forest Baptist Health:

- 1. COMPASS Analytic Database housed by (UNC-CH) EMS Performance and Improvement Center (EMSPIC)
- 2. COMPASS eCare Plan Informatics Database housed by Wake Forest Baptist Medical Center (WFBMC)
- 3. Carolina Survey Research Lab (UNC-CH) will temporarily store data that is needed to conduct the phone surveys and send reminder letters.
- 4. Sheps Center (UNC-CH) will support COMPASS and house claims data.

The sections below describe the information technology protections put in place to ensure security of all patient-level data at all times in each database.

#### **COMPASS Analytic Database at EMSPIC**

All COMPASS participants will be assigned a unique participant ID that will be used to link participant records and identify participants within the database. Only key study investigators, team members and clinicians will have access to the identity of participants.

A comprehensive Data Use Agreement governs the use of the data collected and stored by the UNC EMS Performance and Improvement Center (EMSPIC) for research purposes.

Data security is achieved through storage in a secure data center (Peak10), data inspection and monitoring (StillSecure), and complex application security. Access to COMPASS data will require three levels of security: a badge and security code to enter EMSPIC, a badge and fingerprint scan to access the data center, and a security code for each data rack. All outside access to servers and databases must be accomplished through a Virtual Private Network (VPN). All EMSPIC applications use a strong and sophisticated security module, which restricts access based on entity assignments, and security rights monitored by EMSPIC staff. All applications are only accessible via Hypertext Transfer Protocol Secure (HTTPS). HTTPS is a layering of the standard internet protocol (HTTP) onto an SSL (Secure Sockets Layer) protocol. This results in bidirectional encryption of communications between the client and server and serves as reasonable security against eavesdropping on or tampering with the contents of that communication. The HTTPS protocol will be used for all application through SSL hardware encryption and signed by an accepted root certificate authority.

EMSPIC does not allow the use of portable storage devices and unencrypted data will never be stored on flash drives, external hard disks, or laptops. All applications developed at the EMSPIC prevent SQL Injection attacks from occurring by isolating all form data by escaping incoming string data.

#### Electronic Care (eCare) Plan Informatics Database

The COMPASS eCare Plan Application is a secure web-based application created by a HIPAA-trained programming team at Wake Forest Baptist Medical Center to capture intervention-related data. As described in the intervention section, the eCare Plan Application supports health care providers in efficiently and systematically evaluating patients and identifying next steps for referrals. Data collected into this application will be used to support providers in creation of an individualized care plan (eCare Plan) for patients and generate referral note(s) to other providers (if needed).

Application - IRB00035998

The eCare Plan Application is a secure application utilizing TLS level security (a more secure version of SSL). Communication and data transfer between the user's device (iPad, Desktop, Laptop) and eCare Plan Application are encrypted at all times. To access the eCare Plan Application, health care providers must user-authenticate into the COMPASS portal. The eCare Plan Application will employ role-based security which will limit users access to only information they were authorized to access. Users will be asked to change their password regularly. Data will not be stored locally on any devices to minimize the risk associated with any lost or stolen devices.

The eCare Plan Informatics Database is part of a SQL Server relational data warehouse which is housed in the Wake Forest Health Sciences A1a data center on 3rd Street in Winston-Salem, NC. The webserver hosting the eCare Plan Application is also hosted in the A1a data center. The webserver is a virtual server so in the event of disaster or unexpected significant and lengthy interruption, we can migrate the server into a second data center on Miller St in Winston-Salem, NC. The servers are contained within a secure data center with environmental controls which detect abnormal conditions such as power outages, high heat or humidity, and loud sound. The A1a data center has several secure access points that are accessible only by a badge reader. Only authorized staff will have access to these areas. The building is surrounded by a 10-foot fence with a gate access through badge control. The outside building door is accessed through badge control. The data center room is housed in a locked computer room that is accessed through badge control. Each of these access controls is in place 24 hours a day and seven days a week. All servers have uninterruptible power supplies (UPS). The building has a backup generator that will automatically initiate in the event of a power failure. The computer room is equipped with fire suppression equipment. This equipment is tested on a scheduled timetable by the institution. The entire Data Center is fire- protected by a clean agent system which is backed up by a dry-pipe pre-action sprinkler system. The Data Center room is located on the second floor of the building in an area with no windows and has a raised floor to protect against flooding.

#### Carolina Survey Research Lab Database and Security

Staff at the CSRL must complete training on Human Subjects Protection, Conflict of Interest, and sign a Confidentiality Agreement. The team is provided a wide variety of computing resources for data collection, statistical computing, and office automation. Staff members and research assistants are provided with a Pentium class microcomputer running Windows 7 and Microsoft Office Professional, as well as SAS 9.3 and SUDAAN 10.0 for statistical analysis, virus detection software, and a wide variety of other standard microcomputer software.

CSRL computers communicate securely through the UNC- ITS systems for Internet communications and for access to secure files which have automatic back-up. All sensitive information is hosted on a server that meets the University Information Security policy (<a href="http://its.unc.edu/files/2014/08/Information-Security-Policy.pdf">http://its.unc.edu/files/2014/08/Information-Security-Policy.pdf</a>). This policy includes, but is not limited to, the following configurations: host based and network based firewalls, least functionality, least privileged, weekly vulnerability scans, secure backup (located in a separate location on campus), secured physical access, password enforcement policy, warning banner, incident management plan, monitored malware protection, and patch management.

CSRL manages information in a variety of forms including paper, diskettes, and electronic databases. The CSRL maintains a secure file room in an interior room within a suite for the storage of original paper forms and sensitive data on diskettes. This room is locked at all times and only select staff have access to it. For electronic databases, the CSRL employs two servers: (1) data collection machines, which may collect personal identifiers, are protected on a server behind a physical firewall that is cut-off from the Internet; and (2) data analysis machines have access to a server that stores de-identified data; that is, data collected through the calling room machines that have been stripped of any potential identifiers.

To facilitate surveys, patient and caregiver names, phone numbers and addresses, date of hospital discharge, preferred day and time of contact, as well as PAC information will be exported as a CSV file from the Analytic Database. This file will be stored on a secure server (\cecil.schsr.unc.edu) and accessed by staff at CSRL for pre-loading into their phone system once per week. All access to this secure server will only be granted through UNC secure VPN.

Application - IRB00035998

Trained and approved staff at CSRL will have access to COMPASS Analytic Database to record responses and avoid storing patient level-data in a database outside of the primary COMPASS database.

#### **Sheps Center Data Security**

The Sheps Center will be housing administrative claims data and the server to which EMSPIC and CSRL will post their shared files. Claims data files at the Sheps Center are placed on a secure dataset server configured specifically to handle large-scale health utilization data. Each data file has access restricted to those users authorized by the relevant DUA. The primary dataset directories on the dataset server provide one inventory of our current claims data files. Disk-to-disk backups of claims data files on our dedicated dataset server are made nightly to two separate backup servers at two different Data Center locations on the UNC campus.

Claims data files are housed on a dedicated secure dataset server configured specifically for sensitive health utilization data. The server is physically located in a Tier II data center at 440 W Franklin St, Chapel Hill as part of the UNC campus. These facilities have 24x7 surveillance, multiple power sources and backup power sources, climate control, etc. Our systems administrators get access via electronic pass cards. Each card entry gets recorded with time/date stamps in facility access logs. The dataset server is behind a firewall, accessible only to Sheps Center IP addresses and UNC Secure VPN addresses. There is no printer attached to the dataset server. Only aggregated (anonymized) data and SAS output are taken off the server and onto local computers.

The server is a Linux (RedHat enterprise) server with all unneeded services disabled. Access to the claims data on the Sheps Dataset Server will be restricted to users authorized by the PI. The server is routinely patched with system updates and receives twice-weekly vulnerability scans using Qualys. Identified vulnerabilities are addressed according to UNC Security Policy. Access to the server is via SSH. Off campus access is restricted to UNC VPN connections requiring a user to authenticate with VPN before server login. VPN also provides an encrypted tunnel. SAS and Stata are typical data programs used.

The Sheps Center makes two daily disk-to-disk backups of the secure dataset server. One backup goes to a dedicated backup server within the same Tier II data center at 440 W Franklin. The second goes to a second dedicated backup server at a second Tier II data center located across town at 211 Manning Drive, Chapel Hill. The backup data travel via an SSH tunnel over the same VLAN within the UNC campus firewalls. Both backup servers are behind a firewall denying the ability of other computers or servers to initiate a connection to the backup servers. Instead, the backup servers reach out to the secure dataset server and "pull" the backup data over.

The hard drives and CDs on which data have been delivered will be stored in a locked cabinet at the Sheps Center. Only authorized staff will have keys to the cabinet. The office will be locked when not occupied. In addition, the Sheps Center is locked 24 hours a day.

User level access to claims data files is restricted based on authorized roles. Unix groups are leveraged to provide layered controls. Users may access the data in the following ways:

- Using a computer that is on the UNC Active Directory domain and is managed by UNC ITS security tools that
  perform required scans for viruses and malware and force updated software and operating system patches. Users
  with this type of computer (desktop or laptop) can access the server directly from campus or via a remote VPN
  using SSH.
- 2. Using a computer not managed by UNC ITS security tools via a specifically designated secured UNC Virtual Computer (virtual computing lab), which connects to the server. This virtual desktop is setup, maintained, and managed by Sheps Center sys admins. At the end of a working session, the virtual computer is destroyed along with any data that may have been used locally in the virtual computer instance.

Logical access is safeguarded at multiple levels:

1. The claims data files will be housed on a dedicated secure dataset server configured specifically for sensitive health utilization data. The server is physically located in a Tier II data center at 440 W Franklin St, Chapel Hill,

#### Application - IRB00035998

an extension of the UNC campus. These facilities are governed by the UNC ITS Data Center Operations policies and procedures. They have 24x7 surveillance, required visitor sign-in with escorts, multiple power sources and backup power sources, climate control, etc. Our systems administrators get access via electronic pass cards. Each card entry gets recorded with time/date stamps in facility access logs. While other sys admins of ITS have access to the same physical space where our server racks are housed, these are trusted people governed by central campus ITS policies and procedures. Also, the Data Center space has logged entry of individuals and is under constant surveillance where any unauthorized physical access would be monitored and recorded. Significant sanctions are known and apply, up to and including job termination and possible criminal prosecution.

- 2. The designated server is firewalled allowing only SSH port 22 to be open. All unnecessary ports are closed and all unnecessary services are disabled. User level access to files is restricted based on authorized roles. SSH connections are limited to UNC subnets and UNC VPN addresses. Access to the designated secure dataset server is restricted to computers within the UNC network domain. Connections originating outside the UNC network are restricted to UNC VPN authentication first and then system-level user/pw authentication. Users may only connect using SSH and Kerberos authentication leveraging the UNC Single Sign-on policies and procedures.
- 3. Nightly secure backups are performed to two dedicated backup servers one backup within the same data center within the firewalled subnet and the second backup in another data center across town via the same VLAN. The original CMS data is not backed up to tape but instead the delivery media is kept for backup, if needed. In case of (a) data center disaster, or (b) backup failure, a second backup computer is housed in a second campus data center. Two system administrator computers are allowed to connect to backup servers to control them. Firewall prevents all other computers from reaching backup servers. Backup computers initiate the network connections to the server. It is not possible for any user to initiate a connection to a backup server from the main server or from any other computer except for those owned by two system administrators. All network connections are encrypted.
- 4. The designated server is kept up-to-date with recommended operating system patches and patches for applications. The server is scanned twice weekly for vulnerabilities using the UNC licensed QualysGuard SaaS software. System administrators monitor event logs, security logs, and system logs. UNC uses Snort for intrusion detection and Tipping Point for intrusion prevention. These systems/appliances are monitored and handled centrally by the UNC ITS Security Office. Suspicious activity is reported to the Sheps Center's Security Liaison for investigation and handling with assistance from the central ITS Security Office. If these data will be delivered via CD or hard drive, the media will be kept in a locked storage location provided by the project, with key access only to research team members.
- 5. Project staff at the Sheps Center will access the secure dataset server via SSH using computers physically in the Sheps Center Building. The Sheps Center Building's exterior doors are locked 24x7. Individual offices inside the Sheps Center are also locked. Staff enter using an authorized key. Visitors must be buzzed in using a video intercom system and then must report to the receptionist and sign in. There are no servers physically located in the Sheps Center Building.

#### **Description of the Secure Data Transfers**

Secure Data Transfer between the COMPASS DB and eCare Plan Informatics (eCPI) DB

Data transfer between the COMPASS Database and the eCPI Database will be via RESTful web services designed specifically for the limited datasets being exchanged. Secure data transfer protocols will be in place to provide fully encrypted transmissions. The eCare Application may retrieve and update patient data from the COMPASS Database (the database of record for patient data) for use during a patient visit in order to foster the use of that data in creating an eCare Plan. Patient data is requested based on key identifiers and the resulting match reflected in the eCare application. The web service will allow for the transmission of data stored in the eCPI database to the COMPASS Database for use in analysis as well as patient status updates and notifications to appropriate study personnel. The eCare database remains the database of record for those intervention data while making the COMPASS DB and associated application aware of the analytical data needed for the study. The eCare application will contain the logic necessary during the flow of its data collection to validate data with the patient as well as prevent implausible and/or out-of-range responses.

Application - IRB00035998

#### Secure Data Transfer between COMPASS DB and CSRL

As described above, to facilitate surveys, patient and caregiver names, phone numbers and addresses, date of hospital discharge, preferred day and time of contact, as well as PAC information will be exported as a CSV file from the Analytic Database. This file will be stored on a secure server (\ceil.schsr.unc.edu) and accessed by staff at CSRL for pre-loading into their phone system once per week.

#### **Data Access for Analysis**

We have in place secure operations for sharing SAS datasets between investigators to ensure safety and confidentiality of patients. Datasets will be stored on a secure server that is accessed through a virtual network. Study investigators will be granted access to this server for running data reports and analyses of the study data. These internal datasets will contain the COMPASS Unique participant IDs to link data in different files together. PHI (including date of birth, medical record number, names, addresses, phone numbers, and email addresses) will be removed from datasets prior to export of these SAS datasets from the COMPASS Database. Data sharing with investigators outside of UNC will occur through data transfers using secure File Transfer Protocols.

#### REDCap (Research Electronic Data Capture)

COMPASS Study will use REDCap at Wake Forest Baptist Medical Center to store responses from hospital stakeholders and track stakeholder engagement activities.

Vanderbilt University, with collaboration from a consortium of institutional partners, has developed a software toolset and workflow methodology for electronic collection and management of research and clinical trial data. REDCap (Research Electronic Data Capture) is hosted at Wake Forest Baptist Medical Center through the Biomedical Informatics program of the Translational Science Institute. REDCap servers are located within the Wake Forest Baptist Health firewall and all web-based information transmission is SSL (Secure Socket Layer) encrypted; the databases are backed up nightly through the institution's enterprise backup system. Users are granted access to the system using their unique medical center username and password with specific access rights setup for each study. REDCap was developed specifically around HIPAA-Security guidelines and is used by 1,000+ academic/non-profit consortium partners on six continents with over 195,000 research end-users (www.project-redcap.org).

Application - IRB00035998

#### **Data and Safety Monitoring**

The COMPASS Data and Safety Monitoring Board (DSMB) will serve to support as an independent review board of the study and study activities to protect patients. Adverse events among this patient population are likely; however because COMPASS is a minimal/no risk study, COMPASS will not be tracking adverse events. Therefore the COMPASS DSMB will provide thrice-annual review of study activities providing external review and assurance on the performance of the study. This thrice-annual review will include case ascertainment and enrollment; expected versus observed outcomes; review of percentage of participants in the intervention receiving the 2-day call, the 7-14 day visit, the eCare Plan; and review of protocol deviations.

To avoid any appearance of conflict of interest, it is critical that DSMB members not be involved in the study, have no vested interest in its outcome, have no ties to the study investigators (e.g., not from the same institution and no history of extensive collaboration), and have no financial ties to any commercial concerns likely to be affected by the study's outcome. If at any time a DSMB member perceives that he/she or another member of the Board has a potential conflict of interest, he/she is obligated to bring the issue to the attention of the full DSMB for open discussion and resolution.

#### **Responsibilities**

- 1. COMPASS DSMB members will be responsible for assuring study participants are not exposed to unnecessary, unreasonable or unexpected risk, and is charged with ensuring that the study is conducted according to the highest scientific and ethical standards.
- 2. Specifically, oversight will include the following areas:
  - Review of the COMPASS Manual of Operations and Procedures (MOP), the analysis plan, and implementation of the study procedures at the first DSMB meeting.
  - Review of study protocol including our informed consent processes.
  - The DSMB may recommend modifications or request clarifications of the protocol.
  - Review of the study outcomes and their clear definition, study procedures, informed consent documents, data security, and investigator responsibilities.
  - In subsequent meetings, the DSMB will focus on case ascertainment and enrollment; expected versus observed outcomes; review of percentage of participants in the intervention receiving the 2-day call, the 7-14 day visit, the eCare Plan; and review of protocol deviations.
  - Any other areas the DSMB considers oversight to be necessary.

#### Frequency of Meetings and Communication between DSMB and COMPASS

COMPASS DSMB members will meet annually. The first meeting will take place in person, in early 2016. Subsequent meetings will take place remotely over webinar. Meetings will be closed to the public. Only DSMB members and members of the COMPASS Executive Leadership Committee will attend. ELC members will prepare in advance a DSMB report for review (Appendix 32). Each meeting will start with discussion between COMPASS Executive Leadership Team and DSMB and then the DSMB will meet privately without study personnel.

At the end of each annual meeting, the DSMB will provide a verbal report to the Executive Leadership Team noting any areas of concern in study performance and/or operations. Care will be exercised to ensure no information will be conveyed that could compromise the study or its outcomes. Within two weeks, the DSMB Chair will provide a written report to PCORI and the Executive Leadership Team, which includes the DSMB recommendation for continuing, discontinuing, amending, or suspending the study. This written report will cover data reviewed, recommendations, and date of the next scheduled review. This report will be forwarded by the PIs to the Central IRB at Wake Forest Medical Center and the Data Coordination IRB at the University of North Carolina and PCORI.

#### Membership

The process for identifying the DSMB included feedback from PCORI, recommendations from the Steering Committee and vetting by the Executive Leadership Committee (ELC). The ELC reviewed each recommendation and consulted with PCORI for additional guidance and input on the final selection of DSMB members. Once DSBM members were

Application - IRB00035998

approved by the ELC, the Project Manager sent out a formal letter to the proposed DSMB members inviting them to serve. COMPASS DSMB members include:

#### **DSMB Chair:**

1. Jason Conner, PhD – Director and Senior Statistical Scientist for Berry Consultants. Dr. Connor has expertise in Bayesian statistics and designing adaptive clinical trials. He serves on the Clinical Trials Advisory Panel (CTAP) for PCORI. Dr. Connor has accepted to serve as a DSMB member.

#### **DSMB Members:**

- 2. Judy Lichtman, PhD, MPH Chair, Chronic Disease Epidemiology, Yale University. Dr. Lichtman focuses on stroke research and is experienced in outcomes research, quality improvement and CMS data linkage. Dr. Lichtman has accepted to serve as a DSMB member.
- 3. Brett Kissela, MD Chair of Department of Neurology and Rehabilitation Medicine at the University of Cincinnati (UC) College of Medicine and UC Health. Dr. Kissela is a stroke neurologist and stroke researcher. Dr. Kissela has accepted to serve as a DSMB member.
- 4. Theresa Damush, PhD Associate Research Professor of Medicine, Indiana University School of Medicine. Dr. Damush is a research health psychologist focusing on implementing evidence-based practices for stroke survivors and caregivers. She specializes in the design and evaluation of patient centered programs. Dr. Damush has accepted to serve as a DSMB member.

## **Reporting of Unanticipated Problems or Deviations**

Any unanticipated problems, deviations or protocol changes will be promptly (within 10 days) reported by the principal investigator or designated member of the research team to the IRB and sponsor or appropriate government agency if appropriate.

This study is not collecting or reporting adverse events.

#### **System-Level Protocol Deviations include:**

- Loss of participating site (i.e. a hospital drops out of the study).
- Change of personnel or study staff at the hospital without notifying the COMPASS Team of change of study personnel.

#### **Patient-level Protocol Deviations include:**

- Not notifying enrolled patients that the hospital is participating in the COMPASS Study by either (1) providing the COMPASS brochure packet to the patient prior to discharge or (2) mailing the patient brochure (if the patient is discharged before study staff can inform the patient).
- For Intervention-randomized sites conducting the consent: Consent needs to be conducted by research trained study staff or clinicians.

#### **Study-Level Deviations include:**

• Including any patient participants in analysis (for research purposes) if they have not provided consent and authorization according to our outlined protocols and our "consent matrix" (Appendix 39).
#### References

- 1. American Heart Assosiation. Heart Disease and Stroke Statistics—2015 Update. Circulation. 2015;131:e29–e322.
- 2. Bertoni AG, Ensley D, Goff DC. 30,000 fewer heart attacks and strokes in North Carolina: a challenge to prioritize prevention. *N. C. Med. J.* 2012;73:449–456.
- 3. Kennedy BS. Does race predict stroke readmission? An analysis using the truncated negative binomial model. *J. Natl. Med. Assoc.* 2005;97:699–713.
- 4. Centers for Medicare and Medicaid Services. Chronic Conditions among Medicare Beneficiaries. Baltimore, MD: 2012.
- 5. Olson DM, Cox M, Pan W, Sacco RL, Fonarow GC, Zorowitz R, LaBresh KA, Schwamm LH, Williams L, Goldstein LB, Bushnell CD, Peterson ED. Death and Rehospitalization after Transient Ischemic Attack or Acute Ischemic Stroke: One-year Outcomes from the Adherence Evaluation of Acute Ischemic Stroke–Longitudinal Registry. *J. Stroke Cerebrovasc. Dis.* 2013;22:e181–e188.
- 6. Fonarow G, Smith E, Reeves M, Pan W, Olson D, Hernandez A, Peterson E, Schwamm L. Hospital-level variation in mortality and rehospitalization for Medicare beneficiaries with acute ischemic stroke. *Stroke*. 2011;42:159–166.
- 7. Rosamond W, Johnson A, Bennett P, O'Brien E, Mettam L, Jones S, Coleman S. Monitoring and improving acute stroke care: The North Carolina Stroke Care Collaborative. *N. C. Med. J.* 2012;73:494–498.
- 8. Bernhardt J, Dewey H, Thrift A, Donnan G. Inactive and Alone Physical Activity Within the First 14 Days of Acute Stroke Unit Care. *Stroke*. 2004;35:1005–1009.
- 9. Bamford J, Dennis M, Sandercock P, Burn J, Warlow C. The frequency, causes and timing of death within 30 days of a first stroke: the Oxfordshire Community Stroke Project. *J. Neurol. Neurosurg. Psychiatry.* 1990;53:824–829.
- 10. Johnston KC, Li JY, Lyden PD, Hanson SK, Feasby TE, Adams RJ, Faught RE, Haley EC. Medical and Neurological Complications of Ischemic Stroke Experience From the RANTTAS Trial. *Stroke*. 1998;29:447–453.
- 11. Whitson HE, Pieper CF, Sanders L, Horner RD, Duncan PW, Lyles KW. Adding injury to insult: fracture risk after stroke in veterans. *J. Am. Geriatr. Soc.* 2006;54:1082–1088.
- 12. Davenport RJ, Dennis MS, Wellwood I, Warlow CP. Complications after acute stroke. *Stroke J. Cereb. Circ.* 1996;27:415–420.
- 13. White JH, Attia J, Sturm J, Carter G, Magin P. Predictors of depression and anxiety in community dwelling stroke survivors: a cohort study. *Disabil. Rehabil.* 2014;:1–8.
- Husseini NE, Goldstein LB, Peterson ED, Zhao X, Pan W, Olson DM, Zimmer LO, Williams JW, Bushnell C, Laskowitz DT. Depression and Antidepressant Use After Stroke and Transient Ischemic Attack. *Stroke*. 2012;43:1609–1616.
- 15. Kelly J, Rudd A, Lewis RR, Coshall C, Moody A, Hunt BJ. Venous Thromboembolism After Acute Ischemic Stroke A Prospective Study Using Magnetic Resonance Direct Thrombus Imaging. *Stroke*. 2004;35:2320–2325.
- 16. Lai S-M, Studenski S, Duncan PW, Perera S. Persisting Consequences of Stroke Measured by the Stroke Impact Scale. *Stroke*. 2002;33:1840–1844.
- 17. Bushnell CD, Zimmer LO, Pan W, et al. Persistence with stroke prevention medications 3 months after hospitalization. *Arch. Neurol.* 2010;67:1456–1463.
- 18. Kopunek SP, Michael KM, Shaughnessy M, Resnick B, Nahm E-S, Whitall J, Goldberg A, Macko RF. Cardiovascular Risk in Survivors of Stroke. *Am. J. Prev. Med.* 2007;32:408–412.
- 19. Rigby H, Gubitz G, Eskes G, Reidy Y, Christian C, Grover V, Phillips S. Caring for stroke survivors: baseline and 1-year determinants of caregiver burden. *Int. J. Stroke Off. J. Int. Stroke Soc.* 2009;4:152–158.
- 20. Rigby H, Gubitz G, Phillips S. A systematic review of caregiver burden following stroke. *Int. J. Stroke*. 2009;4:285–292.
- 21. Prvu Bettger J, Alexander KP, Dolor RJ, Olson DM, Kendrick AS, Wing L, Coeytaux RR, Graffagnino C, Duncan PW. Transitional Care After Hospitalization for Acute Stroke or Myocardial Infarction Systematic Review. *Ann. Intern. Med.* 2012;157:407–416.
- 22. Fearon P, Langhorne P, Early Supported Discharge Trialists. Services for reducing duration of hospital care for acute stroke patients. *Cochrane Database Syst. Rev.* 2012;9:CD000443.

#### Application - IRB00035998

- 23. Langhorne P, Taylor G, Murray G, Dennis M, Anderson C, Bautz-Holter E, Dey P, Indredavik B, Mayo N, Power M, Rodgers H, Morten Ronning O, Rudd A, Suwanwela N, Widen-Holmqvist L, Wolfe C. Early supported discharge services for stroke patients: a meta-analysis of individual patients' data. *Lancet*. 2005;365:501–506.
- 24. Kernan WN, Ovbiagele B, Black HR, Bravata DM, Chimowitz MI, Ezekowitz MD, Fang MC, Fisher M, Furie KL, Heck DV, Johnston SC (Clay), Kasner SE, Kittner SJ, Mitchell PH, Rich MW, Richardson D, Schwamm LH, Wilson JA. Guidelines for the Prevention of Stroke in Patients With Stroke and Transient Ischemic Attack A Guideline for Healthcare Professionals From the American Heart Association/American Stroke Association. *Stroke*. 2014::STR.000000000000024.
- 25. Teasell R. Evidence-Based Review of Stroke Rehabilitation [Internet]. [cited 2014 Jun 14]; Available from: <a href="http://www.ebrsr.com/">http://www.ebrsr.com/</a>
- 26. Legg LA, Quinn TJ, Mahmood F, Weir CJ, Tierney J, Stott DJ, Smith LN, Langhorne P. Non-pharmacological interventions for caregivers of stroke survivors. *Cochrane Database Syst. Rev.* 2011;:CD008179.
- 27. Forster A, Brown L, Smith J, House A, Knapp P, Wright JJ, Young J. Information provision for stroke patients and their caregivers. *Cochrane Database Syst. Rev.* 2012;11:CD001919.
- 28. Salter K, Allen L, Richardson M, Teasell R. Community Reintegration [Internet]. EBRSR.COM; 2013. Available from: <a href="http://www.ebrsr.com/sites/default/files/Chapter19">http://www.ebrsr.com/sites/default/files/Chapter19</a> Community-reintegration FINAL 16ed.pdf
- 29. Tu J, Willison D, Silver F, Fang J, Richards J, Laupacis A, Kapral M. Impracticability of informed consent in the Registry of the Canadian Stroke Network. *New Engl J Med.* 2004;350:1414–1421.
- 30. Centers for Medicare & Medicaid Services. Hospital Compare Datasets. [https://data.medicare.gov/data/hospital-compare]
- 31. Kim, SYH and Miller FG. Informed Consent for Pragmatic Trials The Integrated Consent Model. N Engl J Med 2014; 370:769-772

March 19, 2021 Application - IRB00035998 **Appendices** 

### **Appendix 1 - COMPASS Hospital Characteristics**

In order to provide additional details on hospitals that the COMPASS Study is recruiting to participate, we have prepared a side-by-side comparison of the COMPASS Hospitals we expect to randomize with All North Carolina Hospitals (Table 1). We gathered the comparison data from the publicly reported CMS Hospital Compare Information (CMS. Hospital Compare Datasets: https://data.medicare.gov/data/hospital-compare).

For each of the hospitals that we expect to randomize, we have generated Table 2 which provides additional details on the percentage of hospitals that are a Primary Stroke Center (PSC) or a Certified Stroke Center (CSC) and annual stroke volume. This data comes from our North Carolina Stroke Care Collaborative (NCSCC) Data.

Table 3, is the list of hospitals participating in the study. This list was updated in December 2016.

\*\*Table 1. Comparison of Anticipated Participating Hospitals with All NC Hospitals \*\*

| Table 1. Comparison of Anticipated 1 articipating Hospitals with | COMPASS | All NC Hospitals |
|---|---|---|
| | (N=47*) | (N=85) |
| 30-day Mortality Rate for Stroke Patients | 15.6 (14.2 - 16.7) | 15.4 (14.1 - 16.6) |
| 30-day Unplanned Readmission Rate for Stroke Patients | 12.6 (11.8 - 13.4) | 12.8 (12.1 - 13.6) |
| CMS HCAHPS 5-Star Quality Rating, median score | | |
| Overall summary score | 3 (3 - 4) | 3 (3 - 4) |
| Care transition score | 3 (3 - 4) | 3 (2 - 4) |
| Stroke quality measures, % of patients that received measure | | |
| Venous Thromboembolism (VTE) Prophylaxis | 98 (96 - 100) | 99 (96 - 100) |
| Discharged on Antithrombotic Therapy | 100 ( 99 - 100) | 100 ( 99 - 100) |
| Anticoagulation Therapy for Atrial Fibrillation/Flutter | 100 (96 - 100) | 100 (96 - 100) |
| Thrombolytic Therapy | 95 (91 - 100) | 93 (84 - 99) |
| Antithrombotic Therapy by End of Hospital Day 2 | 100 (98 - 100) | 100 (98 - 100) |
| Discharged on Statin Medication | 98 (96 - 100) | 99 (96 - 100) |
| Stroke Education | 97 (92 - 100) | 97 (90 - 100) |
| Assessed for Rehabilitation | 100 (99 - 100) | 100 (98 - 100) |

<sup>\*</sup>Data from Murphy Medical Center are not available from Hospital Compare.

Notes: Values are presented as median (25th, 75th percentile). HCAHPS represents Hospital Consumer Assessment of Healthcare Providers and Systems.

<sup>\*\*</sup>This Table was last Updated in Jan 2016

\*\*Table 2. Characteristics of Anticipated Hospitals (N=48)

| | N | Percent |
|------------------------------------------------------|----|---------|
| Teaching hospital | 2 | 4% |
| Joint Commission stroke certified sites (PSC or CSC) | 22 | 46% |
| Geographic region | | |
| Piedmont | 26 | 54% |
| Western | 11 | 23% |
| Eastern | 11 | 23% |
| Annual stroke volume | | |
| <100 discharges | 12 | 25% |
| 100-299 discharges | 23 | 48% |
| 300+ discharges | 13 | 27% |

<sup>\*\*</sup>This Table was last Updated in Jan 2016

Application - IRB00035998
Table 3. List of Participating Hospitals (Table Updated December 2016)

| Table 3. List of Participating Hospitals (Table Updated December 2016) # Hospital Wave Arm Stroke 2013 Stroke | | | | | |
|---|---|---|---|---|---|
| # | Hospital | wave | Arm | Stroke<br>Center | 2013 Stroke<br>Discharges |
| 1 | Cana Foor Valley Medical Center | 1 | Usual Care | PSC | 300+ |
| 2 | Cape Fear Valley Medical Center | 1 | Intervention | PSC | 300+ |
| 3 | FirstHealth Moore Regional | | | | |
| | Onslow Memorial Hospital | 1 | Usual Care | PSC | 100-299 |
| 4 | Carteret County General Hospital | 1 | Intervention | PSC | 100-299 |
| 5 | WFBH Lexington Medical Center | 1 | Usual Care | PSC | 100-299 |
| 6 | Hugh Chatham Memorial Hospital | 1 | Intervention | PSC | 100-299 |
| 7 | Pardee Health | 1 | Usual Care | No | 100-299 |
| 8 | Lenoir Memorial Hospital | 1 | Intervention | No | 100-299 |
| 9 | CHS NorthEast | 2 | Intervention | PSC | 300+ |
| 10 | Novant Health Presbyterian Medical Center | 2 | Usual Care | PSC | 300+ |
| 11 | New Hanover Regional MC | 2 | Usual Care | PSC | 300+ |
| 12 | Mission Hospital | 2 | Intervention | PSC | 300+ |
| 13 | Novant Health Huntersville Medical Center | 2 | Intervention | PSC | 100-299 |
| 14 | Novant Health Matthews Medical Center | 2 | Usual Care | PSC | 100-299 |
| 15 | CHS University | 2 | Intervention | No | 100-299 |
| 16 | CHS Blue Ridge | 2 | Usual Care | No | 100-299 |
| 17 | CHS Union | 2 | Intervention | PSC | 100-299 |
| 18 | CHS Cleveland | 2 | Usual Care | PSC | 100-299 |
| 19 | CHS Kings Mountain | 2 | Usual Care | No | <100 |
| 20 | Wilkes Regional Medical Center | 2 | Intervention | No | 100-299 |
| 21 | Northern Hospital of Surry County | 2 | Usual Care | PSC | <100 |
| 22 | Frye Regional Medical Center | 2 | Intervention | PSC | 300+ |
| 23<br>a | Carolinas Medical Center | 3 | Intervention | PSC | 300+ |
| 23<br>b | CHS Mercy (randomized with CMC as a single unit) | 3 | Intervention | PSC | <100 |
| 24 | WakeMed Health & Hospitals | 3 | Usual Care | PSC | 300+ |
| 25 | Duke Raleigh Hospital | 3 | Usual Care | PSC | 100-299 |
| 26 | CHS Stanly | 3 | Intervention | PSC | 100-299 |
| 27 | Ashe Memorial Hospital | 3 | Intervention | No | <100 |
| 28 | Alleghany | 3 | Usual Care | No | <100 |
| 29 | Betsy Johnson Hospital | 3 | Usual Care | No | 100-299 |
| 30 | Morehead Memorial Hospital | 3 | Intervention | No | <100 |
| 31 | UNC Hospital | 3 | Usual Care | CSC | 300+ |
| 32 | Rex Healthcare | 3 | Intervention | PSC | 300+ |
| 33 | CHS Lincoln | 3 | Usual Care | No | <100 |
| 34 | Caldwell Memorial Hospital | 3 | Intervention | No | 100-299 |
| 35 | Vidant Duplin Hospital | 3 | Intervention | PSC | <100 |
| 36 | Blue Ridge Regional | 3 | Usual Care | No | <100 |
| 37 | Vidant Edgecombe Hospital | 3 | Usual Care | No | 100-299 |
| 38 | Angel Medical Center | 3 | Intervention | No | <100 |
| 39 | Washington County Hospital | 3 | Intervention | No | <100 |
| 40 | SouthEastern Regional Medical Center | 3 | TBD | No | 300+ |

# March 19, 2021 Application - IRB00035998 Appendix 2 - COMPASS Hospital Survey

| COMPASS Study Hospital Surve | ey . | |
|---|---|---|
| The goal of this survey is to understand your hospital's current<br>through post-discharge management. We also wish to capture<br>cases and whether you would be willing to consider participation<br>COMPASS) trial. | information about how your hospital is | dentifies stroke |
| We appreciate your time and attention to the survey. If you ha<br>(sara.jones@unc.edu). | ve any questions, please contact Sara | Jones |
| Thank you! | | |
| The COMPASS Team | | |
| RESPONDENT INFORMATION | | |
| Title | 7-01-100-4-01-01-01-01-01-0 | |
| Full Name: | | |
| Email address: | | |
| Hospital Name: | | |
| Hospital City: | | |
| Hospital Zip Code: | | |
| Please check the description that best defines your position: Director of care coordination and/or case management Director of translational care clinic Quality improvement director Stroke care coordinator Other | | |
| If other, please specify | | |
| 01/21/2016 5:27pm | www.projectredcap.org | ₽EDCap |

| | |
|---|---|
| ACUTE STROKE CARE | |
| How many patients with ischemic or hemorrhagic str<br>your hospital in 2015 or the last calendar year for wh | roke or TIA meeting the ICD-9/10 criteria below were treated at hich you have data? Click below to view the ICD table. |
| [Attachment: "ICD table.PNG"] | |
| Enter the most recent calendar year for which you have data | |
| In the last calendar year, how many stroke and TIA<br>patients were discharged directly home from your<br>hospital? | |
| How frequently are patients with presumptive stroke | P/TIA diagnosis (stroke-like symptoms) identified in your hospital |
| Daily Two or more times per week One time per week One time every 2 weeks One time per month | |
| | troke/TIA diagnosis during the weekend entered into a daily |
| ○Yes ○No | |
| What information is used to develop a roster of patie that apply) | ents admitted with a presumptive stroke/TIA diagnosis? (check al |
| □ Diagnosis (ICD-10 codes) □ Census for selected units (ICU or dedicated neuro □ Hospital problem list - principle problems □ Hospital problem list - other problems □ Census for the entire hospital □ Review of daily admissions/arrivals for admitting □ □ Use of stroke admission order sets □ Code stroke logs □ Neurology consult orders □ Stroke rounds by attending and/or residents □ Shared *stroke patient* lists □ Other | |
| Please specify what other information is used | |
| Who in your hospital is responsible for developing a | list of patients admitted with a presumptive stroke/TIA diagnosis |
| Stroke care coordinator Direct care nurse Stroke care provider (MD, NP, PA) Nursing operations supervisors Nursing unit managers Nursing unit team leaders Other | |
| Please specify other responsible party | |
| 01/21/2016 5:27pm | www.projectredcap.org |

| Conf | idential |
|---|---|
| 7 | Who in your hospital abstracts stroke patient information into the NCSCC Stroke Care Card or Get-With-The-Guidelines-Stroke PMT? |
| | <ul> <li>Stroke care coordinator</li> <li>Data abstractor other than stroke coordinator</li> <li>NA, data captured electronically with no manual abstraction</li> <li>NA, do not participate in NCSCC or GWTG-Stroke</li> <li>Other</li> </ul> |
| | Please specify other hospital abstractor |
| 8 | Who in your hospital is responsible for compliance with CMS Medicare and Medicaid Performance Metrics for acute stroke care? |
| | <ul> <li>Stroke care coordinator</li> <li>Quality performance manager</li> <li>Other</li> </ul> |
| | Please specify other responsible party |
| 9 | Can patients who are admitted to your hospital with a presumptive stroke/TIA be identified concurrent with practice? Yes No |
| 9a | If no, what are the barriers to concurrent identification of stroke/TIA patients? (check all that apply) |
| | Please specify other barrier to identification |
| 10 | For questions 10a-10i Indicate the frequency with which each provider type (includes MDs, NP/PA) admits patients with a presumptive stroke/TIA |
| 10a | Hospitalists |
| | <ul> <li>△ All of the time</li> <li>✓ Mostly</li> <li>Occasionally</li> <li>Rarely</li> <li>Never</li> </ul> |
| 10b | Intensivists |
| | All of the time Mostly Occasionally Rarely Never |
| | 01/21/2016 5:27pm www.projectredcap.org REDCap |

| | TEOUSES AND THE STATE OF THE ST | |
|---|---|---|
| Cont | idential | |
| 10c | Neurologists | |
| | All of the time Mostly Occasionally Rarely Never | |
| 10d | Neurosurgeons | |
| | All of the time Mostly Occasionally Rarely Never | |
| 10e | Nephrologists | |
| | All of the time Mostly Occasionally Rarely Never | |
| 10f | Oncologists | |
| | <ul> <li>△ All of the time</li> <li>✓ Mostly</li> <li>✓ Occasionally</li> <li>✓ Rarely</li> <li>✓ Never</li> </ul> | |
| 10g | Cardiologists | |
| | All of the time Mostly Occasionally Rarely Never | |
| 10h | Internal medicine (non-hospitalists) | |
| | <ul> <li>△ All of the time</li> <li>△ Mostly</li> <li>○ Occasionally</li> <li>○ Rarely</li> <li>○ Never</li> </ul> | |
| 10i | Other | |
| | All of the time Mostly Occasionally Rarely Never | |
| | Please specify type of other | |
| 11 | Is information on patients discharged following stroke/TIA (e.g. name, address, telephone) available at | t your hospital? |
| | ○ Yes ○ No | |
| | | _ |
| | 01/21/2016 5:27pm www.projectredcap.org | <b>₹EDCap</b> |

| Cont | fidentia | | |
|---|---|---|---|
| 12 | Is inform | mation on the patient's post-acute caregiver (e.g. name, address, telephone) available at your | hospital? |
| | ○ Yes | | |
| | 20 M | | |
| 13 | | our hospital have a dedicated stroke team? | |
| | ○ Yes | ○ No | +X 15 |
| 13a | | he actively involved (i.e. participating in at least 75% of meetings each year) members of the<br>le. (check all that apply) | stroke team by |
| | ☐ Neur | | |
| | ☐ Nurs | e practitioner | |
| | | charge nurse<br>manager (e.g. RN) | |
| | Phar | macist | |
| | | ical Therapist<br>Ipational Therapist | |
| | ☐ Spee | ech therapist | |
| | ☐ Nutr<br>☐ Beha | itionist<br>ivioral or mental health specialist | |
| | | al worker (e.g. MSW) | |
| | Please | describe the other role | |
| 14 | Does yo | our hospital have a stroke unit or dedicated beds in a specific unit for stroke patients? | |
| | Yes | ○ No | |
| 15 | | our hospital use telestroke for acute care (i.e. access to acute stroke experts via two-way live ation and image sharing technology)? | video and audio |
| | Yes - | - as a hub hospital<br>- as a spoke hospital (supported by telestroke service) | |
| 15a | Please | provide name of the hub hospital | |
| 16 | with coo<br>for exar<br>provide<br>O Yes | our hospital have a patient navigator for your stroke patients? [The patient navigator is some ordination of healthcare services and offers assistance in reducing barriers to receiving care a mple, arranging for financial support, arranging transportation services, coordination of visits are.] - supporting acute care only - supporting post-acute care only | ind treatment; |
| | O Yes | supporting both acute and post-acute care | |
| | ○ No | | |
| 17 | Does yo | our hospital have an inpatient peer/mentor support program for your stroke patients? | |
| | Yes | ○ No | |
| | 01/21/20 | 16 5:27pm www.projectredcap.org | <b> ♠</b> EDCap |

| |
|---|
| DISCHARGE PLANNING FOR PATIENTS GOING HOME |
| Do you have a multidisciplinary discharge planning team for stroke patients? [By multidisciplinary discharge planning team, we mean a team of physicians, nurses, and key ancillary service specialists involved in managing a patient's discharge] |
| ○ Yes ○ No ○ Do not know |
| Please identify members of your discharge planning team. (check all that apply) |
| Neurologist Hospitalist Nurse practitioner Unit charge nurse Case manager (e.g., RN, BSN, or MSN) Pharmacist Physical therapist Occupational therapist Speech therapist Nutritionist Behavioral or mental health specialist Social worker (e.g. MSW) Other Specify type of other member |
| Does your hospital conduct an assessment of stroke patient's and family's transitions needs prior to discharge? |
| ○ Yes ○ No ○ Do not known |
| What areas are assessed and documented in the patient's medical record? (Check all that apply) |
| <ul> <li>□ Caregiver availability after discharge for supervision and assistance</li> <li>□ Activities of Daily Living</li> <li>□ Physical Mobility (Balance, Strength, Endurance, and Walking)</li> <li>□ History of Falls</li> <li>□ Assessment of cognitive function using standardized assessments (e.g. Mini Mental Status Exam, Montreal Cognitive Assessment -MOCA)</li> <li>□ Home environment assessment for safety and mobility</li> </ul> |
| ☐ Need for assistive equipment ☐ Availability of transportation for follow-up appointments |
| ☐ Confirmation of primary care provider ☐ Appointment made for follow-up with primary care provider ☐ Depression and need for follow-up care |
| <ul> <li>Advanced directives and end of life planning</li> <li>Need and referral for other follow-up: home visit by RN, NP/PA or MD, home health, outpatient rehabilitation, other outpatient specialty care</li> <li>Knowledge and need for community services, e.g., meals on wheels, support groups, etc.</li> <li>Other</li> </ul> |
| Describe other areas |
| Does your hospital assess the stroke patient/family's understanding of their discharge instructions and transition home (e.g. teach-back)? |
| ○ Yes ○ No ○ Do not know |
| 01/21/2016 5:27pm www.projectredcap.org <b>REDCap</b> |

| Con | |
|---|---|
| 200 | DAMACOLA POLICIO |
| 3a | What areas are assessed for patient/family understanding? (check all that apply) Risk factors for stroke Management of risk factors following discharge Medications and plan for medication management Follow up appointments, procedures and services Stroke signs and symptoms Expected level of recovery within 90 days Other |
| | List other areas that are assessed |
| 4 | Does your hospital include a transition of care plan in the discharge summary for the stroke patient/family? |
| | Yes No Do not know |
| 5 | Is an appointment made with a primary care provider prior to discharge? |
| | ○ Yes ○ No |
| 5a | What are the challenges with getting a primary care appointment within 14 days of discharge? (check all that apply) |
| | None Insurance type Patient does not have insurance Patient does not have a primary care provider Unable to reach the primary care provider's office to make the appointment Availability of primary care appointments within 7 to 14 days post-stroke Patient refusal Other |
| | Specify other challenge |
| 5b | For what proportion (percentage) of your stroke patients are you able to make a follow-up appointment with a primary care provider within 14 days? |
| 50 | Is a hospital discharge summary sent to the patients' primary care provider when an appointment is made? |
| - | O Yes O No O Do not know |
| 6 | Is a patient specific transitional care plan sent to the primary care provider and/or rehab providers? |
| | ○ Yes ○ No ○ Do not know |
| | ### ## |
| 1 | 01/21/2016 5:27pm www.projectredcap.org REDCap |

| fidential |
|---|
| POST-DISCHARGE PATIENT MANAGEMENT AND FOLLOW-UP |
| (For stroke/TIA patients discharged home) |
| Does the hospital perform follow-up telephone calls for stroke patients after discharge? |
| No - there is no patient follow-up by telephone Yes - within 48-72 hours of discharge Yes - within 7 days Yes - within 14 days Yes - other time point (enter time below) |
| Enter the number of days after discharge |
| Specify other provider |
| Who usually makes this follow-up call? |
| <ul> <li>Stroke care coordinator</li> <li>Stroke care nurse</li> <li>Designated transitional care coordinator</li> <li>Other</li> </ul> |
| Specify other |
| How would you best describe the setting in which stroke patient's follow-up care is delivered? |
| Neurology Clinic Hospitalist Clinic Paramedicine Program Stroke Follow-up Clinic General Follow-up Clinic (not stroke-specific) Primary Care Practitioner's Clinic Chronic disease Transitional Care Clinic Other |
| Specify other setting |
| Does your hospital/health system provide in-person specialty follow-up with neurology to all stroke patients? |
| No clinic or outpatient follow-up with neurology Yes - clinic or outpatient visit within 14 days of hospital discharge Yes - clinic or outpatient visit within 30 days of hospital discharge Yes - clinic or outpatient visit within 60 days of hospital discharge Other in-person follow-up arrangement In-person home visit (please indicate days after hospital discharge below) |
| Describe other follow-up arrangement |
| Enter the number of days after discharge |
| 01/21/2016 5:27pm www.projectredcap.org REDCap |

| Con | fidential |
|---|---|
| , | 3.4 €4 (PP-343500) |
| 4 | If there is follow-up that occurs within 14 days of hospital discharge (either with a general primary care provider or neurology specialist), who is the health care professional primarily responsible for the in-person follow-up? |
| | ○ No in-person follow-up is performed within 14 days ○ Nurse Practitioner only |
| | Physician Assistant only Physician only |
| | Either Nurse Practitioner or Physician Assistant Nurse Practitioner or Physician Assistant and a Physician Other |
| | Specify other type of health professional |
| 4a | Please indicate what are the objectives of the in-person follow-up appointment/visit or neurology specialty follow up. Select all that apply. |
| | Conduct a thorough neurological examination Review medication use, access, and adherence, and reconcile as needed |
| | Assess risk factor levels Coordinate access to primary care |
| | Coordinate use of home health services, outpatient physical therapy, occupational therapy, or speech therapy (as needed) |
| | Provide referral to community services Other |
| | Specify other objectives of the in-person follow-up |
| 5 | Does your hospital have an electronic patient care plan for post-acute management accessible to the patient and all of his or her providers (e.g. primary care, rehabilitation teams, home health) caring for stroke patients after hospital discharge? |
| | Yes - available to the patient and all post-acute providers Yes - available to all post-acute providers (no direct patient access) Yes - available to select post-acute providers only No |
| | Please describe the select providers |
| 6 | Does your hospital share electronic medical record information with any of the following non-hospital services for stroke patients following discharge home? Select all that apply. |
| | ☐ No, information is not shared with non-hospital services ☐ Primary care practices ☐ Home health agencies |
| | ☐ Outpatient therapy practices<br>☐ Mental health providers |
| | ☐ Outpatient neurology care ☐ Outpatient specialty care |
| | ☐ Telehealth sites and care providers after hospital discharge ☐ EMS after hospital discharge |
| | <ul> <li>☐ Hospital or health system sponsored stroke support group</li> <li>☐ Community resources for stroke (e.g., external stroke support groups, caregiver support groups, AAA, community exercise programs, senior centers)</li> <li>☐ Other</li> </ul> |
| | Specify other |
| | 01/21/2016 5:27pm www.projectredcap.org <b>REDCap</b> |

| Conf | fidential | 1 | | | | | | 27 000000000000000000000000000000000000 |
|---|---|---|---|---|---|---|---|---|
| 7 | | | tal have integrate<br>y of the following. | | | d coordination | and communicati | on for stroke |
| | Prima | ☐ No, integrated care plans with non-hospital providers are not in place ☐ Primary care practices ☐ Home health agencies ☐ Outpatient therapy practices | | | | | | |
| | | tal healti | | | | | | |
| | | | eurology care | | | | | |
| | | | ecialty care<br>ter hospital discha | irge | | | | |
| | | | spital discharge<br>ealth system spon | sored stroke sunr | port group | | | |
| | ☐ Com | munity r | esources for strok | e (e.g., external s | | roups, caregive | r support groups, | AAA, |
| | Othe | | xercise programs, | senior centers) | | | | |
| | Specify | other pla | ans | | | | | |
| 8 | patients | s? (The 1 | | codes 99495 an | | | CM) billing codes to<br>ion with patient a | |
| | Yes | ○ No | O Not Sure | | | | | |
| 9 | stroke p | oatients? | | | | | ement (CCM) billi<br>provided to patient | |
| | ○ Yes | ○ No | O Not Sure | | | | | |
| 10 | | | al measure patient<br>tion and disability | | ephone for strok | e patients afte | r discharge (e.g., ı | medication |
| | O Yes, | calls ma | assessment by tel<br>de 30 days after d | ischarge | | | | |
| | | | de 60 days after d<br>de 90 days after d | | | | | |
| | OYes, | | de 180 days after | discharge | | | | |
| | 200000000000000000000000000000000000000 | | iming of calls | | | | | |
| | Describ | e other t | ining or cans | | | | | |
| 10a | Please i | indicate | what outcomes are | acsassed Salar | rt all that annly | | | |
| 100 | | | | assessed. Selec | c an enac apply. | | | |
| | | nitive fun | tion/disability<br>iction | | | | | |
| | | | n or depression<br>dherence | | | | | |
| | Risk | factor kr | nowledge | | | | | |
| | ☐ Care | giver str | ain | | | | | |
| | Specify | other ou | tcomes | | | | | |
| 11 | Does yo | ou hospit | al use metrics to a | ssess the quality | of care transitio | ns? | | |
| | ○ Yes | ○ No | O Do not know | | | | | |
| 11a | List met | trics used | 4 | | | | | |
| | 01/21/201 | 16 5:27pm | | | | Ware | .projectredcap.org | <b> REDCap</b> |
| | 100000000000000000000000000000000000000 | | | | | 17,556 | | cela |

| | | 1000033996 | | |
|---|---|---|---|---|
| Cont | idential | | | |
| 12 | Does your hospi<br>readmissions for | tal have any other programs or strategies not already des<br>r stroke patients? | scribed that specifically focu | s on reducing |
| | ○Yes ○No | O Do not know | | |
| 12a | Describe progra | ms or strategies | | |
| 13 | Does your hospi<br>reduce readmiss | tal have any other transitional care management progran<br>sions for diagnoses other than stroke? | ns or efforts to improve care | transitions and |
| | ○Yes ○No | O Do not know | | |
| 13a | Describe these p | programs and patient population targeted. | | |
| 14 | Please add anyt | hing else you would like to share about the transitional ca | are services available at you | r hospital. |
| | 01/21/2016 5:27pm | | www.projectredcap.org | <b>₹EDCap</b> |

| identi al | | |
|---|---|---|
| DESCRIPTIVE DATA | | |
| What was the 30-day all-cause readmission rate for stroke patie 99] | ents last calendar year (enter a %)? [If t | inknown, enter |
| What was the 90-day all-cause readmission rate for stroke patie | ents last calendar year (enter a %)? [If t | ınknown, enter |
| | | <b> ♠ EDCap</b> |

# March 19, 2021 Application - IRB00035998 Appendix 3 - Eligibility Screening Form

| 1 | COMPREHENSIVE POST-ACUTE STROKE SERVICES Participant Eligibility Screening Form |
|---|---|
| ID Nur | mber: Form Code: E L G Date: 100CT2016 Version 1.2 |
| ADMINI | STRATIVE INFORMATION (0a-0d and 0f are auto-populated) |
| 0a. Comp | oletion Date: Month / Day / Year Ob. Staff ID: |
| 0c. NCS | |
| 0e. Medio | cal Record #: Of. Form Status: |
| ELIGIBI | LITY CRITERIA |
| 1. Patier | nt date of birth Day / Year |
| 2. What | is the patient's primary language? □ English □ Spanish □ Other |
| 3. Was t | he patient admitted for the sole purpose of elective carotid endarterectomy? ☐ Yes ☐ No |
| 4. What | is the final hospital diagnosis (see clinical algorithm for assistance)? |
| [ | □ Ischemic stroke Stroke symptoms persisting > 1 hour with at least 1 of the following: 1) MRI confirmation of infarct/ischemia; 2) receipt of tPA; or 3) high suspicion of cerebrovascular cause OR transient stroke symptoms with MRI confirmation of infarct/ischemia. Exclude suspected stroke mimics. ICD-10 code examples: 163.0, 163.1, 163.2, 163.3, 163.4, 163.50, 163.6, 163.8, 163.9, 166.19, 166.29, 166.9, 167.89, H34.1 [retinal vascular occlusion], H34.23 [retinal artery branch occlusion] |
| [ | Non-traumatic intraparenchymal hemorrhage Stroke symptoms with CT and/or MRI confirmation of IPH. ICD-10 code example: I61.0-I61.4, I61.8-I61.9 |
| | Other non-aneurysmal intraventricular hemorrhage Intraventricular blood suspected to have originated from brain (e.g. thalamus) and with no evidence of aneurysm. |
| Г | □ Ischemic stroke with hemorrhage<br>Hemorrhagic conversion noted within an ischemic stroke (would be coded similar to IS above) |
| [ | ☐ Stroke not otherwise specified Stroke symptoms without MRI confirmation (e.g. patients who cannot receive MRI due to pacemaker) and stroke cannot be seen on CT scan. |
| [ | ☐ Transient ischemic attack (TIA) → Go to Question 4a Transient episode of neurological dysfunction without infarction. Exclude diagnosis of TIA vs. complicated migraine, syncope, infection, reactivation of old stroke symptoms, medication reaction, delirium ICD-10 code examples: all G45 except G45.3 [amaurosis fugax] |
| | □ Aneurysmal subarachnoid hemorrhage<br>Headache or stroke symptoms with CT and/or MRI confirmation of SAH and aneurysm. ICD-10 code<br>example: 160.0-161-9 |

| 4a. Was a brain MRI performed? ☐ Yes → Go to Question 4b ☐ No | |
|---|---|
| 4b. Did MRI show evidence of an acute infarct? ☐ Yes ☐ No | |
| 5. What is the patient's discharge disposition? | |
| <ul> <li>Home with self-care</li> <li>Home with home health</li> <li>Hospice – home</li> <li>Hospice – health care facility</li> <li>Acute care facility</li> <li>Other health care facility → Go to Question 5a</li> <li>Expired</li> <li>Left against medical advice</li> <li>Jail, prison, or other detention facility</li> <li>Not documented or unable to determine</li> </ul> | |
| 5a. If 'OTHER HEALTH CARE FACILITY, specify the type: | |
| ☐ Skilled nursing facility ☐ Inpatient rehabilitation ☐ Long-term care ☐ Intermediate care facility ☐ Other | |
| END OF PARTICIPANT ELIGIBILITY SCREENING FORM | |
| Eligibility Screening Form | Page 2 of 2 |

| COMPREHENSIVE POST | ASS ST-ACUTE STROKE SERVICES Participant Enrollment Form |
|---|---|
| ID Number: | Form Code: E N R Date: 06JUN2016 Version 1.0 |
| ADMINISTRATIVE INFO | ORMATION (auto-populated) |
| 0a. Completion Date: | Month / Day / Year Ob. Staff ID: |
| 0c. NCSCC ID: | 0d. Hospital ID: 0f. Form Status: |
| A. PATIENT CONTACT | |
| 1. Patient full name | |
| | First Middle Last |
| 2. Telephone number(s) | |
| a. Primary number: ( | ( |
| Best time to call: | □ Home □ Mobile □ Work □ Other <u></u> □ Weekday daytime □ Weekday evening □ Weekend □ Anytime |
| b. Alternate 1: ( | ( |
| | □ Home □ Mobile □ Work □ Other |
| Best time to call: L | □ Weekday daytime □ Weekday evening □ Weekend □ Anytime |
| c. Alternate 2: ( | |
| | □ Home □ Mobile □ Work □ Other<br>□ Weekday daytime □ Weekday evening □ Weekend □ Anytime |
| 3. Email address | |
| 4. Home address | Address line 1 |
| | Address line 2 |

| for example, in p | | nember or friend who will help ther<br>g or taking medications, schedulin | |
|---|---|---|---|
| 5. Caregiver full nar | ne | | |
| | First | Middle | Last |
| 6. Caregiver gende | r: □ Male □ Female | | |
| 7. Telephone numb | er(s) | | |
| a. Primary numb | er: ( | - | |
| Ту | oe: □ Home □ Mobile □ Wor | rk □ Other | |
| b. Alternate 1: | ( | - | |
| Ту | oe: □ Home □ Mobile □ Wor | rk □ Other | |
| 8. Email address | | | |
| | Address line 1 | | |
| | Address line 2 | | |
| | City | State | Zip |
| 10. What is the care | giver's primary language? | | |
| | ☐ English☐ Spanish☐ Other | | <u></u> |
| 11. Caregiver relation | onship to the patient? | | |
| | <ul> <li>□ Spouse (husband or wife</li> <li>□ Sibling</li> <li>□ Son or daughter</li> <li>□ Friend or neighbor</li> <li>□ Parent or legal guardian</li> </ul> | ·) | |

| ☐ Patient unable or | unwilling to provide an additional contact / not documented → Go | to Question 16 |
|---|---|---|
| 12. Full name | - | |
| | First Middle | Last |
| 13. Telephone numbe | ers | |
| a. Primary number | : ( | |
| Туре | e: 🗆 Home 🗆 Mobile 🗆 Work 🗆 Other | _ |
| b. Alternate 1: | ( | |
| Туре | e: 🗆 Home 🗆 Mobile 🗆 Work 🗆 Other | |
| 14. Email address: | | |
| 15. Relationship to pa | atient? | |
| | <ul><li>□ Son or daughter</li><li>□ Friend or neighbor</li></ul> | |
| D DEMOGRAPHIC | ☐ Parent or legal guardian ☐ Other, specify: AND IN-HOSPITAL DATA | |
| 16. Patient gender: | ☐ Other, specify: | |
| D. DEMOGRAPHIC 16. Patient gender: 17. Patient race (check) | □ Other, specify: | |

| 20. Does the patient have document | ed past medical | history of the fol | lowing (check all that ap | oply): |
|---|---|---|---|---|
| <ul><li>☐ Stroke</li><li>☐ Transient ischemic attack</li></ul> | <ul><li>☐ Hypertension</li><li>☐ Dyslipidem</li></ul> | | <ul><li>☐ Chronic renal insuff</li><li>☐ Heart Valve</li></ul> | iciency |
| ☐ Atrial Fibrillation or Flutter | ☐ Smoking | | ☐ Current pregnancy | or within 6 |
| ☐ Myocardial infarction or CAD | ☐ Depression | f | weeks post-partum ☐ Hormone replacem | ent therapy |
| <ul><li>☐ Congestive heart failure</li><li>☐ Carotid stenosis</li></ul> | <ul><li>□ Drug/alcoh</li><li>□ Family history</li></ul> | | ☐ Sickle cell☐ Sleep apnea | |
| ☐ Peripheral arterial disease | ☐ Migraines | | ☐ Diabetes mellitus | |
| 21. Please enter the body mass inde | ex (BMI) | kg/m² | ☐ Not documented | |
| 22. What was the patient's ambulato | ry status <u>prior to</u> | admission? | | |
| ☐ Able to am | bulate independ | ently (with or wit | hout a device) | |
| ☐ With assist☐ Unable to a | tance (from pers | on) | | |
| ☐ Not docum | | | | |
| 23. NIH Stroke Scale Score (00-42) | | □ N | lot documented | |
| | | - | | |
| 24. Has this patient been admitted w | ithin the past 90 | days for a TIA o | r stroke? | |
| □ Yes → F | ill in date and l | CD code below | | |
| Date of Ad | _ | Month Day | / Year | |
| Discharge | ICD code: | | | |
| □ No<br>□ Not docum | ented | | _ | |
| 25. Did the initial exam show aphasia | a? □Yes | □ No / not doc | umented | |
| 26. Hospital admission date for this e | event: | | / 🗌 📗 | |
| ☐ No admission date; patient wa | s not admitted a | s an inpatient (s | elect reason below) | |
| | | | inpatient admission | |
| ☐ Other reaso | | | | |
| | | s after discharge | e? □ Yes → Go to 27a | □ No → Go to 27b |
| ☐ Other reaso | | s after discharge | e? □ Yes → Go to 27a | □ No → Go to 27b |
| ☐ Other reason. 27. Was the patient referred for reha | bilitation service:<br>/<br>erapy | □ Outpatient Ph | nysical Therapy<br>ccupational Therapy | □ No <b>→</b> Go to 27b |

| 28. What was the | patient's ambulatory status <u>at discharge</u> ? | |
|---|---|---|
| | <ul> <li>□ Able to ambulate independently (with or without a device)</li> <li>□ With assistance (from person)</li> <li>□ Unable to ambulate</li> <li>□ Not documented</li> </ul> | |
| 29. Modified Rank | in Score at discharge (0-6) | ed |
| 30. Hospital disch | arge date: | |
| 31. Was a follow-<br>care clinic, ne | ip clinic visit with a nurse, nurse practitioner, or physician assistant (i.e. primary care, trans<br>irologist, or other doctor visit) scheduled prior to discharge? | ition |
| | ☐ Yes → Fill in date below ☐ No | |
| If YES, enter | visit date: Month / Day / Year | |
| 32. Name of patie | nt's primary care provider: Not known | |
| 33. Phone number | er of patient's primary care provider: | |
| | ( | ļ |
| 34. Did the PAC r | otify the patient of the COMPASS study and distribute the brochure? | |
| | <ul> <li>☐ Yes, discussed in person and distributed brochure</li> <li>☐ Yes, discussed over the phone and mailed brochure to patient</li> <li>→ Fill in date bel</li> <li>☐ No</li> </ul> | |
| If YES, enter<br>notification of | | |
| | END OF PARTICIPANT ENROLLMENT FORM | |

### Appendix 5 - Control-Arm Patient Handout - COMPASS Study

## Your recent hospital visit means that you are eligible for the COMPASS Study. Will you help us?

Your hospital is participating in a statewide study called the Comprehensive Post-Acute Stroke Services (COMPASS) Study. This study includes people who have had a stroke or transient ischemic attack (TIA), sometimes referred to as a mini-stroke. The purpose of the COMPASS Study is to determine the best ways to care for patients after they go home – to help survivors find their way forward to recovery.

In the COMPASS Study, North Carolina hospitals have been randomly assigned into two groups (similar to flipping a coin). One group of hospitals is providing patients with their usual standard of care after the patient goes home. The other group of hospitals is providing their usual care with the addition of an evaluation by a nurse practitioner, physician assistant or doctor within two weeks of hospital discharge, during which patients will receive a plan of care that will be shared with their other doctors, therapists and nurses.

#### Our hospital is providing the usual standard of post-acute care which includes:

- A hospital discharge summary that will go to the doctor that cares for you
- · A discharge plan of care provided to you
- [insert other post-acute stroke transitional care services provided by the hospital]

We are committed to finding the best way to improve health and recovery after experiencing this health episode. The COMPASS study will not interfere with the usual standard of care at our hospital or your usual and planned follow up visits with your primary care doctors.

**After you have left the hospital,** the **COMPASS** team would like to learn about your overall experience. They will:

- Call you in 3 months to ask questions about your recovery and satisfaction with your care.
- Mail you 3 reminder letters before you are called. The last letter will include a small gift to thank
  you for your time, so be sure to open it.
- Mail a survey to the family member, friend, or neighbor whom you identify as helping you in your recovery (care helper).

Whether or not you choose to participate in the survey, our hospital is committed to providing you with high-quality care for you during your recovery. All information you and your *care helper* provide will be kept strictly confidential and secure.

If you have any questions about the COMPASS Study, or prefer not to participate, feel free to ask the stroke coordinator, or you can call the COMPASS Study team using the toll-free number below.

Hospital Stroke Coordinator: [insert stroke coordinators name and phone number]

COMPASS toll-free number: 1-844-501-7668
COMPASS Study website: <a href="https://www.nccompass-study.org">www.nccompass-study.org</a>



## Appendix 6 - Letter to the Patient at 30 Days and Magnet

Dear < NAME>, < DATE>

Greetings from the COMPASS Study! We are contacting you on behalf of <HOSPITAL>, which is participating in our study. You may remember your nurse gave you a brochure about our study purpose while in the hospital. As a reminder, our goal is to improve healthcare and the lives of North Carolinians who had a transient ischemic attack (TIA), mini-stroke, stroke, or related episode.

#### What to expect:

In a couple months you will receive a call from a team member at the Carolina Survey Research Lab to ask you to take part in a phone survey. During this call, we would like to talk with you about how you have been doing since your hospital visit. The survey is brief, and is completely voluntary and confidential. Your participation will be very valuable in helping other patients and their families find their way forward to recovery.

#### How you can participate:

- [-] Your call is tentatively scheduled for the week of **DATE** >
- [-] We will call you at <PHONE #>
- [-] We have enclosed a COMPASS Study refrigerator magnet and will send a gift to you in a future letter so be sure to open it!

If the phone number above is incorrect or if you would like to opt-out of this call and future letters, please contact us as soon as you can at the toll-free number: 1-844-501-7668.

#### Find out more about the COMPASS Study:

[-] To learn more about the COMPASS Study please visit our website: <a href="https://www.nccompass-study.org">www.nccompass-study.org</a>

[-] If you would like to speak with a team member about the study, call us at: 1-844-501-7668

Thank you very much for your time and we look forward to speaking with you soon! Best regards,

The COMPASS Study Team

P.S Don't forget to mark your calendar. Your response matters!



Finding Your Way Forward After a Stroke or TIA

#### Appendix 7 - Letter to the Patient at 60 Days

Dear <NAME>,

Greetings from the COMPASS Study team! This is another reminder that you will be receiving a call from a team member at the UNC Carolina Survey Research Lab. They will ask you to take part in a phone survey. The survey is brief, completely voluntary and confidential. Your participation will be very valuable in helping other North Carolinians and their families.

#### How you can participate:

- [-] Your call is tentatively scheduled for the week of <DATE>
- [-] We will call you at <PHONE #>
- [-] We will send you one more reminder letter a week before the call. That letter will include a copy of the survey questions and our thank you gift so be sure to open it!

Please contact us at the toll-free number 1-844-501-7668 if any of the information above is incorrect or you would like to opt out of the phone call and future letters.

We encourage you to explore resources provided by the American Heart/ American Stroke Associations. The free *Stroke Family Warmline* connects you to other individuals and their families who have had experiences similar to yours (1-888-4-STROKE). The *Stroke Connection Magazine* is also an excellent resource. You can read a digital copy and subscribe by visiting: http://strokeconnection.strokeassociaton.org

#### Find out more about the COMPASS Study:

- [-] To learn more about the COMPASS Study and to find other useful information about care after stroke or mini-stroke, please visit our website: <a href="https://www.nccompass-study.org">www.nccompass-study.org</a>
- [-] If you would like to speak with a team member about the study, call us at: 1-844-501-7668

Best regards,

The COMPASS Study Team

### **Appendix 8 - Letter to the Patient at 80 Days**

Dear <NAME>, <DATE>

Greetings from the COMPASS Study team! As you know, we are working to determine the best ways to care for individuals after they go home from the hospital. <HOSPITAL NAME> and your doctor have identified you as a participant in this study.

A team member at the UNC Carolina Survey Research Lab is planning to call. We want to hear how you've been doing since your hospital visit a few months ago. Attached is a copy of the survey questions if you would like to review them before the call. We appreciate your help in improving healthcare in North Carolina!

#### How you can participate:

- [-] We have enclosed \$10 to say THANK YOU in advance!
- [-] Your call is scheduled for the week of <DATE >
- [-] We will call you at <PHONE #>
- [-] Our records show your preferred call window is: <BEST TIME TO CALL>

Please contact us as soon as you can at the toll-free number 1-844-501-7668 if any of the information above has changed.

At the beginning of the call, you will be asked if you wish to participate. Participation is completely voluntary and confidential and any information you provide will be held securely. We hope that you will provide your input.

#### Find out more about the COMPASS Study:

[-] To learn more about the COMPASS Study please visit our website:

#### www.nccompass-study.org

[-] If you would like to speak with a team member about the study, call us at:

1-844-501-7668

We look forward to speaking with you soon!

Best regards,

The COMPASS Study Team

#### [pg 2]

**HIPAA Authorization Note:** The COMPASS Study team has worked with your hospital and doctor to identify you as a potential participant for this research study. The Carolina Survey Research Lab (CSRL) will ask for your consent to participate when they call you next week. We do hope that you will agree to participate in the survey but this is voluntary and optional. Any responses you provide will be held confidential and securely.

By agreeing to participate in the phone survey, you will be giving permission to CSRL to use or disclose your identifiable health information for the COMPASS research study. The health information that we may use or disclose for this research includes information from your recent hospital visit, visits to your doctor, medications, and other information about your insurance claims. The health information listed above may be used by and/or disclosed to the study investigators at this site and others, study management centers, the study sponsor, and other groups, including federal agencies, which have a responsibility to assist in the oversight and management of the research study.

Please note that <HOSPITAL NAME> may not refuse to treat you if you do not provide consent for this Authorization and phone survey. Once you have agreed, you may change your mind and take back the Authorization at any time. Even if you take back this Authorization, the organization may still use information that was previously collected about you. To take back the Authorization, you must call 1-844-501-7668 or email thecompassstudy@gmail.com. Authorization does not have an expiration date.

# March 19, 2021 Application - IRB00035998 Appendix 9 - NCSCC Stroke Care Card

| Stroke Care NCSCC Stroke Care Card v12.8.6 Med. Record # | | | |
|---|---|---|---|
| ollaborative | Initial Prese | entation Data | Stroke ID |
| 1. Hospital Arrival: Date: | 6. Presumptive Hospital Diagnosis (at time of admission, related to stroke; check one): Collected concurrently ** □ Subarrachnoid Hemorrhage (ICH) Subarrachnoid Hemorrhage (ISAH No Stroke Related Diagnosis Stroke NOS TIA 7. Where was the patient when stroke was detected or when symptoms were discovered? (Check one) Not in a health care facility Another acute care facility Chronic health care facility While in-patient in this hospital Outpatient health care setting Cannot be determined 8. When was the patient: Last known to be well? Date:/ _ ND Time: | the patient first evaluated? (Check one) □ ED/Urgent care □ Direct admit, not via ED □ Imaging suite prior to ED | 13. Was brain imaging performed at this hospital as part of the initial evaluation for this episode of care or event? Yes, after ED admission No/ND NC (outside imaging prior to transfer or patient is DNR/CMO) Yes, prior to ED admission at this hospital IF YES: 13a. Date/Time of initial brain imaging: Date:/ ND ND ND ND ND 13b. Date/Time brain image results first read by a physician: Date:/ ND ND ND 13c. Brain Imaging Findings: No Hemorrhage New Hemorrhage Old Hemorrhage ND ND ND ND ND ND ND N |
| | | aphic Data | |
| 14. DOB:// | | 19. Documented past medical history o | F. (about all that apply) |
| ☐ Black/African American | 17. Gender: Male Female ND | Stroke □ DM □ TIA/VBI □ MI or CAD □ PAD □ Obesity □ HRT □ Migraines □ Heart Valve □ Carotid ste □ Hypertension □ Sickle cell □ Dyslipidemia □ Depression □ AF or Flutter □ CHF □ Drug/Alcohol abuse □ Sleep apn □ Smoking (≥1 cigarette in past yr.) □ Pregnancy w/in 6 weeks □ Chronic renal insufficiency □ Pregnancy w/in 6 weeks □ Family history of stroke 19b. Currently taking (prior to admission): (check all that apply) □ Cholesterol reducing medication □ Antiplatelet □ Antidepressant □ Antihypertensive □ Anticoagulant | |
| | t-PA | A Data | |
| 20. Was IV t-PA initiated for this pati | ent at this hospital? | f 21b is checked: | |
| Yes, Date:/_ ND Ti If q. 20 is YES: 20a. What were the first blood press SBP/DBP (mmHg) / Glucose (mg/dL) | me: ND No | 22b. Were there bleeding complications PA? ☐ Yes, detected prior to transfer ☐ Ye ☐ Unable to determine ☐ No | es, detected after transfer |
| 20b. If IV t-PA was initiated >60 minu eligibility or medical reasons do ☐ Yes ☐ No ☐ NA, IV t-PA ir | ocumented for cause of delay? | f q.20 is NO <u>and</u> 21b not checked:<br>24. Identify reason(s): (check all that app | ly) □ Collected Concurrently ** |
| 20c. Were there reasons for extending to 3.0-4.5 hours? ☐ Yes ☐ No | ng the initiation of IV thrombolytic | ☐ Contraindication (See NCSCC Data Manual for | |
| 21. Was other thrombolytic therapy a. No b. IV t-PA outside hos c. IA catheter based reperfusion at Date: ND ND If q. 20 is YES or 21b is checked: | this hospital - Give date & time: | IV or IA tPA given at outside hospital Advanced age Rapid improvement Severity too mild Patient/family refused Care team unable to determine eligibility | |
| 22a. Complications of thrombolytic t ☐ None ☐ Symptomatic ICH w | therapy: | ☐ CT findings of ICH, SAH, or major infar<br>☐ Life expectancy <1 year or severe | |

| | In-Hosp | ital Data | | |
|---|---|---|---|---|
| 27. Was patient NPO throughout the entire hospital st Yes | STOP, patient ineligible cation SKIP to Q49 SKIP to Q49 SKIP to Q49 SKIP to Q49 A steel No/ND Signature arrival? Signa | 34. Was the patient or caregiver provided smoking cessation counseling? Yes | | |
| ☐ Yes ☐ No/ND ☐ CI 33a. Did patient die on the 2nd day after arrival or later ☐ No ☐ Yes → Skip to Q49 | | □ Yes □ No/ND 45. Was patient treated for hospital-acquired pneumonia during this admission? □ Yes □ No/ ND □ CI | | |
| | Discha | rge Data | | |
| 46. Did the patient and/or caregiver receive stroke education and/or resource materials? (check all that apply) Personal modifiable risk factors | | ent's ambulatory le? (check one) independently swice) from person) ite Score ND (0-6) //Death: gnosis rhage (ICH) | □ ED only □ □ In-patient only □ □ S2. Discharge disposition: □ Home, self-care □ Home with home hea □ Hospice - Health care □ Acute care facility □ Other health care fac □ SNF □ Inpatient rehat □ Long-term care □ Intermediate ci □ Other □ Expired □ Left against medical is ND / unable to determ | Both ED and In-patient None : (check one) Ith care e facility illity (please specify) polititation e are facility advice/AMA |
| ☐ Patient/family refused rehab services | ☐ No stroke related dia☐ Stroke NOS☐ TIA | | 54. ICD-9 discharge dx | ICD-10 discharge dx |
| *ND = Not Documented; **Collected Concurrently = While | Patient Hospitalized: ** | *CI = Documented | Contraindication | 11/12/2014 |

## Appendix 10 - Screener and Consent (At 90 Days)

#### CONSENT LANGUAGE PULLED OUT OF THE SCREENER

#### **PURPOSE**:

We are calling to follow up on his/her/your recent hospital stay at [HOSPITAL]. This hospital is participating in the COMPASS study which is a research study looking at how patients are doing after their stroke.

#### **EXPLAIN [IF IRB MON=1]:**

[....] During this survey, you have the right to refuse to answer any questions you don't want to answer and you can stop participating at any time. [....]

#### **SECURITY:**

We wanted to also let you know that by participating you are giving us permission to keep a record of your responses to the survey. All of your responses and data will be strictly confidential and will be kept in a secure location.

#### **RISKBENEFIT:**

We do not anticipate that participation in this survey involves any risks. There is also no direct benefit to you for participating.

#### **PARTICIPATE/CONSENT:**

Do I have your permission to continue with the survey?

#### THANK YOU:

Thank you for agreeing to participate in the COMPASS Study.

#### IF IRB OFFER NUM:

If you have any additional questions about the study, I can provide the numbers of the Wake Forest and UNC Chapel Hill Institutional Review Boards. Their job is to protect your rights and welfare as a research participant. They have reviewed and approved this study. Would you like those numbers?

The survey also has a link to the COMPASS website.

#### IRB\_PI NUMBER [IF [IF IRB\_OFFER NUM=1]:

If you have any questions, comments or concerns about the study, please contact, anonymously if you wish, the Wake Forest IRB at 336-716-4542 or the UNC Chapel Hill Institution Review Board. You can reach them at 919-966-3113 or by email to <a href="mailto:IRB\_subjects@unc.edu">IRB\_subjects@unc.edu</a>. This information is also at the bottom of the survey that was mailed to you.

Information about how to reach the COMPASS project manager, the UNC Institutional Review Board, as well as the link to the COMPASS website, are at the bottom of the survey that was mailed to you.

## Screener

| LABEL | VALUE | TEXT | INSTRUCTIONS |
|---|---|---|---|
| DID ANSWER | 0-1 | INTERVIEWER: DIAL | |
| | 0=NO | ###-###- DID A | |
| | 1=YES | PERSON ANSWER? | |
| | | IF NO, HANG UP AFTER | |
| | | 12 RINGS. | |
| UNKNOWN HELLO | 1=PERSON NAMED ON | Hello, my name is [FULL | PRELOAD NAME |
| [IF DID ANSWER=1] | PHONE OR COMING | NAME] and I'm calling on | |
| | TO PHONE (GO TO | behalf of [HOSPITAL | |
| | SEL_HELLO) | NAME] and the | |
| | 2= PERSON NAMED | COMPASS STUDY. | |
| | NOT AVAILABLE (GO | | |
| | TO SCHEDULE_CB1) | May I places speek with | |
| | 3= PERSON NAMED ON PHONE IS IN THE | May I please speak with [FIRST NAME LAST] | |
| | HOSPITAL, INPATIENT | NAME]? | |
| | REHAB OR A NURSING | TVZ TIVILEJ: | |
| | HOME(GO TO | | |
| | IN FACILITY) | | |
| | 4= PATIENT UNABLE | | |
| | TO TALK ON PHONE | | |
| | DUE TO THEIR | | |
| | STROKE (GO TO | | |
| | MED_SPECIFY) | | |
| | 5= PERSON NAMED ON | | |
| | PHONE IS DECEASED | | |
| | (GO TO DECEASED) | | |
| | 6= PERSON NAMED NO | | |
| | LONGER AT THIS NUMBER, BUT NOT IN | | |
| | A FACILITY (GO TO | | |
| | ASK NEW#) | | |
| | 7=NO ONE BY THAT | | |
| | NAME KNOWN (GO TO | | |
| | MISMATCH) | | |
| | 99=HANG UP OR | | |
| | PERSON NAMED | | |
| | REFUSES TO COME TO | | |
| | PHONE | | |
| ASK_NEW# | 0=NO, GK WILL NOT | Does [Mr/Ms LAST | |
| | PROVIDE NUMBER | NAME] have a new | |
| | (GO TO END | personal or residential number where I could reach | |
| | INTERVIEW AND CODE REV1 | [him/her] regarding this | |
| | 1=YES, GK WILL | study? | |
| | PROVIDE NUMBER | Study: | |
| | (GO TO GET_NEW#) | IN: IF GK SAYS R IS | |
| | | DECEASED, IN A | |
| Application - IRB00035998 | | T | T |
|---|---|---|---|
| | | FACILITY OR | |
| | | MEDICALLY | |
| | | INCAPABLE, GO BACK | |
| | | TO UNKNOWN HELLO | |
| | | AND CHOOSE - | |
| | | APPROPRIATE | |
| | | RESPONSE. | |
| | | 1651 51 (55) | |
| | | IF NEEDED: For the | |
| | | purposes of this study, we | |
| | | are not able to speak with | |
| | | those in nursing homes or | |
| | | other facilities, but we | |
| | | might be able to speak with | |
| | | a family member or friend. | |
| GET NEW# | ENTER NUMBER | Thank you. What is that | |
| | | number? | |
| GET_ALT# | ENTER NUMBER (GO | Is there another number in | |
| _ | TO END INTERVIEW, | case we don't reach | |
| | THEN APPOINTMENT | [him/her] at that number? | |
| | TAB) | | |
| | , | IN: IF NO OTHER | |
| | | NUMBER, LEAVE | |
| | | EMPTY AND HIT ENTER | |
| | | TO CONTINUE | |
| SCHEDULE CB1 | 1=PREFERRED CB | I am calling in regard to a | |
| _ | TIME PROVIDED (GO | phone survey we would like | |
| | TO THANK CB) | you/[MR/MS LAST | |
| | 2= PERSON NAMED ON | NAME] to complete. | |
| | PHONE IS IN THE | You/she/he should have | |
| | HOSPITAL, INPATIENT | received some letters about | |
| | REHAB OR A NURSING | this survey. When would be | |
| | HOME (GO TO | a good time to call back? | |
| | IN FACILITY) | | |
| | 3= PATIENT UNABLE | IN: IF R IS NO LONGER | |
| | TO TALK ON PHONE | AT THIS NUMBER BUT | |
| | DUE TO THEIR | NOT IN A FACILITY, GO | |
| | STROKE (GO TO | BACK TO | |
| | MED_SPECIFY) | UNKNOWN_HELLO | |
| | 4= PERSON NAMED ON | AND CHOOSE #6 | |
| | PHONE IS DECEASED | | |
| | (GO TO DECEASED) | | |
| | A DEFENCE (CO TO | | |
| | 9=REFUSE (GO TO | | |
| IN EACH ITY | RESP_REF) | Do you think a/k a 11 1 | DDELOAD |
| IN_FACILITY | 0=NO (GO TO | Do you think s/he will be available and able to do a | PRELOAD |
| | FACILITY_SPECIFY) | | EXPIRATION |
| | 1=YES (GO TO | phone survey before | DATE |
| | SCHEDULE_CB2) | [EXPIRATION DATE MINUS 2DAYS?] | |
| | 8=DON'T KNOW (GO | | |
| | * | IF 'DON'T KNOW'. | |
| | TO SCHEDULE_CB2) | IF 'DON'T KNOW': | |

| Application - IRB00035998 | | | |
|---|---|---|---|
| | 9=REFUSE (GO TO | OK, I'll plan to try to call | |
| | FACILITY SPECIFY) | back before then to see if | |
| | | they are available. | |
| FACILITY_SPECIFY | 1=the hospital (GO TO | Could you please tell me, is | |
| | PROXY) | s/he currently in | |
| | 2=an in-patient | Sinc currently in | |
| | | IN: IF GK HAS | |
| | rehabilitation facility, or | | |
| | (GO TO PROXY) | ALREADY SPECIFIED | |
| | 3=a nursing home? (GO | FACILITY, CONFIRM | |
| | TO PROXY) | INFORMATION HERE | |
| | 4=OTHER (GO TO | | |
| | SPEC_OTHER) | | |
| SPEC_OTHER | OPEN TEXT | SPECIFY OTHER | |
| | (250 CHARACTERS) | | |
| MED SPECIFY | 1=DIFFICULTY | For our records, would you | ALL GO TO |
| _ | TALKING | mind telling me: Is | PROXY |
| | 2=DIFFICULTY | [Mr./Ms. LAST NAME] | |
| | UNDERSTANDING | unable to do the survey | |
| | 3=TOO SICK | because [he/she] has | |
| | 4=OTHER (GO TO | difficulty talking, difficulty | |
| | OTHER MED) | understanding, is too sick | |
| | OTHER_WED) | or is there some other | |
| | 9-DON'T L'NOW (CO | | |
| | 8=DON'T KNOW (GO | reason [he/she] is unable to | |
| | TO PROXY) | do the survey? | |
| | 9=REFUSE (GO TO | | |
| | PROXY) | IN: IF GK INFORMS YOU | |
| | | THAT R IS IN A | |
| | | FACILITY, GO BACK TO | |
| | | UNKNOWN_HELLO | |
| | | AND CODE | |
| | | APPROPRIATELY | |
| | | BEFORE CONTINUING | |
| OTHER_MED | OPEN TEXT | What other reason is that? | |
| 0 11121_1122 | 50 CHARACTERS | | |
| PROXY | 1= YES, WILLING | I'm sorry to hear that. I | IF |
| IKOXI | PROXY ON PHONE (GO | would like to complete the | UNK HELLO=3,4 |
| | TO RCV INFO, THEN | survey with someone else if | OR 5 OR |
| | PROXY NAME, THEN | possible. | SCHEDULE CB1=2 |
| | - | Does Mr/Ms [LAST | _ |
| | PROXY_REL, THEN | _ | ,3 OR 4AND |
| | EXPLAIN) | NAME] have an adult | IN_FACILITY=0 |
| | 2= YES, WILLING | relative or health care | AND PROXY=0, GO |
| | PROXY COMING TO | power of attorney who can | TO INEL AND |
| | PHONE (GO TO | be reached at this number | CODE PRE1 (IN |
| | SELECTED_HELLO, | and who has regular contact | FACILITY) |
| | RCV INFO, PROXY | with him/her and knows | |
| | NAME, PROXY REL) | about his/her health and | |
| | 3= YES, PROXY IS | could take the survey on | IF UNK_HELLO=6 |
| | UNAVAILABLE (GO TO | his/her behalf? | OR |
| | PROXY NAME, THEN | | SCHEDULE_CB1=5 |
| | SCHEDULE CB2) | | AND PROXY=0, GO |
| | 4= NO, THERE IS NO | | TO INEL AND |
| | PROXY (GO TO INEL) | | CODE MEDX |
| <u> </u> | (23 10 11,211) | L | |

| Application - IRB00035998 | 5= PROXY REFUSAL<br>(GO TO RESP_REF) | | |
|---|---|---|---|
| SEL_HELLO [IF UNKNOWN HELLO=1] | 0-3 0=NO 1=YES (GO TO RCV_INFO AND/OR PROXY_NAME, THEN EXPLAIN) 2=UNKNOWN UNAVAILABLE 3=UNKNOWN REFUSAL (GO TO RESP_REF) | IF PARTICIPANT OR PROXY IS ALREADY ON THE PHONE, ENTER "YES" IF PARTICIPANT JUST CAME TO THE PHONE, SAY: Hello, my name is [FULL NAME]. I'm calling on behalf of the COMPASS study. Am I speaking with [FILL IF PROXY=1 OR 2: an adult relative or health care power of attorney for ] [FIRST NAME LAST NAME]? | IF PROXY=3 OR 4, GO TO RCV_INFO THEN PROXY NAME |
| RCV_INFO [IF SELECTED HELLO = 1] | 1=CONTINUE (GO TO EXPLAIN) 2=R UNAVAILABLE (GO TO SCHEDULE_CB2) 3=R REFUSAL (GO TO RESP_REF) | We are calling to follow up on his/her/your recent hospital stay at [HOSPITAL]. This hospital is participating in the COMPASS study which is a research study looking at how patients are doing after their stroke. We recently sent him/her/you a description of the study and some reminder letters about this call Today I'm calling to ask you some questions about how you are feeling and about your health in general. IF PROXY=2: We were informed earlier that Mr./Ms. [LAST NAME] would be unable to participate in a phone survey due to his/her health | PRELOAD GENDER |

| Application - IRB00035998 | | T | I |
|---|---|---|---|
| | | but that you would be able | |
| | | to answer our questions on | |
| | | his/her behalf. | |
| | | INTERVIEWER: IF R CLAIMS HE IS | |
| | | UNAWARE OF THE | |
| | | STUDY, PROMPT BY | |
| | | DESCRIBING. IF | |
| | | STILL UNFAMILIAR, | |
| | | CODE FINAL | |
| | | REFUSAL. | |
| | | IN: THE LETTER IS | |
| | | NOT REQUIRED TO | |
| | | DO THE PHONE | |
| | | SURVEY | |
| PROXY_NAME | OPEN TEXT | Could you please tell me | PROGRAMMING: |
| | (10 CHARACTERS) | your first name so that I can | THIS IS A |
| | | refer to you personally? | REQUIRED |
| | GO TO PROXY | IN: THIS IS A REQUIRED | FIELD |
| | RELATION | FIELD. IF PROXY IS | |
| | | UNWILLING TO | |
| | | PROVIDE A NAME,<br>EXPLAIN THAT YOU | |
| | | NEED INITIALS OR A | |
| | | NICKNAME SO THAT IF | |
| | | YOU MUST CALL BACK | |
| | | YOU CAN BE SURE TO | |
| | | REACH THEM AND NOT | |
| | | SOME OTHER FRIEND | |
| | | OR FAMILY MEMBER. | |
| PROXY RELATION | 1=Legal guardian? | For our records, can you | |
| _ | 2=Health care agent named | tell us your relationship to | |
| | under a health care power | [R NAME]? | |
| | of attorney? | | |
| | 3=Spouse? | IN: IF NOT ONE OF | |
| | 4=Adult son and/or | THESE DELATIONSLIPS D | |
| | daughter?<br>5=Parent? | RELATIONSHIPS, R<br>MUST COMPLETE | |
| | 6=Adult brother and/or | ELIGIBILITY AND | |
| | sister? | CONSENT | |
| | 7=Uncle and/or aunt? | HIM/HERSELF BEFORE | |
| | 8=Other adult relative (GO | ALLOWING PROXY TO | |
| | TO OTHER_REL)? | COMPLETE; GO BACK | |
| | | TO UNK_HELLO AND | |
| | 88=DON'T KNOW (GO | CHOOSE APPROPRIATE | |
| | TO | RESPONSE TO SPEAK | |
| | 99=REFUSED (GO TO<br>RESP REF | TO R OR GO BACK TO PROXY AND CHOOSE | |
| | KLSI KLI | #4, NO PROXY | |
| OTHER REL | OPEN TEXT | SPECIFY OTHER | |
| | 50 CHARACTERS | RELATIONSHIP | |
| | | 1 | I |

#### March 19, 2021

Application - IRB00035998

| PROXY_AGE | 1=YES (GO TO | And I need to confirm, are | DON'T ALLOW |
|---|---|---|---|
| | HOSP_INFO) | you at least 18 years old? | REF OR DK |
| | | Di Hava da Di du | |
| | | IN: IF NO, GO BACK | |
| | | AND RE-ASK PROXY | |
| | | AND CODE | |
| MOMERCH | 0.0 | APPROPRIATELY. | |
| MISMATCH | 0-2 | Let me just confirm that I | |
| [IF UNKNOWN | 0=NO | dialed correctly. Did I | |
| HELLO=8] | 1=YES | reach you at ###-####? | |
| | 2=HANG UP BEFORE | | |
| | NUMBER | | |
| | VERIFICATION | | |
| MISDIAL | EMPTY | I'm sorry. I must have | REDIAL |
| [IF MISMATCH=0] | | misdialed. Thank you for | |
| | | your time. | |
| DECEASED | ENTER DATE (GO TO | I'm very sorry to hear that. | END CALL AND |
| | END INTERVIEW AND | Would you mind telling me | CODE DECX |
| | CODE DECX) | when s/he passed away so | |
| | DON'T KNOW(GO TO | that I can record that | |
| | END INTERVIEW AND | information and we do not | |
| | CODE DECX) | call again? | |
| | REFUSE(GO TO END | | |
| | INTERVIEW AND | | |
| | CODE DECX) | | |
| END INTERVIEW | EMPTY | Thank you for your time. | END CALL |
| [IF ASK_NEW#=0 OR 1 | | | |
| OR MISMATCH=1] | | | |
| T . | | | l . |

| HOSP INFO | 1=INFO ON RECORD IS | Our records show that | PRELOAD |
|---|---|---|---|
| <u> </u> | | | HOSPITAL AND |
| [IF IRB_CONF=1] | CORRECT (GO TO | he/she/you was/were | DISCHARGE DATE |
| | EXPLAIN) | hospitalized for a stroke or | DISCHARGE DATE |
| | 2=HOSPITAL IS | TIA at [HOSPITAL] and | |
| | WRONG (GO TO NEW | that he/she/you was/were | |
| | HOSP) | sent home on [DschrgD]. | |
| | 3=DISCHARGE DATE | T d i io | |
| | IS WRONG (GO TO | Is that correct? | |
| | NEW DISCHARGE) | | |
| | 4=R SAYS NOT | IF NEEDED: TIA stands | |
| | HOSPITALIZED FOR | for transient ischemic | |
| | STROKE (GO TO NEW | attack and is sometimes | |
| | ADMIT) | referred to as a mini-stroke | |
| | | or warning stroke. | |
| | 8=DON'T KNOW (GO | | |
| | TO EXPLAIN) | IN: R MAY HAVE BEEN | |
| | 9=REFUSE (GO TO | HOSPITALIZED ON | |
| | EXPLAIN) | OTHER DATES, BUT WE | |
| | | ARE NOT ASKING | |
| | | ABOUT THOSE. | |
| | | IT IS OKAY TO | |
| | | CONTINUE EVEN IF R | |
| | | DOES NOT REMEMBER | |
| | | HOSPITAL AND DATE | |
| | | INFORMATION. | |
| NEW_HOSP | OPEN TEXT | What was the name of the hospital where you were hospitalized for your | |
| | | stroke? | |
| NEW DISCHARGE | MM/DD/YYYY | What was the date of your discharge? | |
| NEW ADMIT | OPEN TEXT | What were you hospitalized | |
| TIEST TENTIFIE | VI ELI I ELIZI | for? | |
| EXPLAIN | 1-3 | Before I continue, I need to | |
| [IF IRB_MON=1] | 1=CONTINUE (GO TO | let you know that for quality | |
| [ | HOSP INFO) | control purposes, this call | |
| | 2=R UNAVAILABLE | may be monitored by my | |
| | 3=R REFUSAL (GO TO | supervisor. | |
| | RESP REF) | During this survey, you have | |
| | | the right to refuse to answer | |
| | | any questions you don't want | |
| | | to answer and you can stop | |
| 1 | İ | participating at any time. | |
| | | participating at any time. | |
| INELIGIBLE | | I'm sorry, but that means we | |
| INELIGIBLE | | | |
| INELIGIBLE | | I'm sorry, but that means we | |

| Application - IRB0003599 | 8 | |
|---|---|---|
| | | appreciate your talking with me. |
| ELIGIBLE | 1-3<br>1=CONTINUE (GO TO<br>PURPOSE) | INTERVIEWER: CASE IS<br>NOW ELIGIBLE, ENTER 1<br>TO CONTINUE |
| LENGTH | 1-3<br>1=CONTINUE (GO TO<br>SECURITY)<br>2=R UNAVAILABLE<br>3=R REFUSAL (GO TO<br>RESP_REF) | The survey should take about 20 minutes to complete. |
| SECURITY | 1-3<br>1=CONTINUE (GO TO<br>RISKBENEFIT)<br>2=R UNAVAILABLE<br>3=R REFUSAL (GO TO<br>RESP_REF) | We wanted to also let you know that by participating you are giving us permission to keep a record of your responses to the survey. All of your responses and data will be strictly confidential and will be kept in a secure location. |
| RISKBENEFIT | 1-3<br>1=CONTINUE (GO TO<br>INCENTIVE)<br>2=R UNAVAILABLE<br>3=R REFUSAL (GO TO<br>RESP_REF) | We do not anticipate that participation in this research survey involves any risks. There is also no direct benefit to you for participating. |
| IRB_OFFER NUM | 0-1<br>0=NO<br>1=YES (GO TO IRB_PI<br>NUMBER) | If you have any additional questions about the study, I can provide the numbers of the Wake Forest and UNC Chapel Hill Institutional Review Boards. Their job is to protect your rights and welfare as a research participant. They have reviewed and approved this study. Would you like those numbers? The survey also has a link to the COMPASS website. |
| IRB_PI NUMBER<br>[IF [IF IRB_OFFER<br>NUM=1] | EMPTY | If you have any questions, comments or concerns about the study, please contact, |

Application - IRB00035998

| Application - IRB00035998 | 3 | |
|---|---|---|
| | | anonymously if you |
| | | wish, the Wake Forest |
| | | IRB at 336-716-4542or |
| | | the UNC Chapel Hill |
| | | Institutional Review |
| | | Board. You can reach |
| | | them at 919-966-3113 or |
| | | by email to |
| | | IRB subjects@unc.edu. |
| | | IKB subjects(w)unc.edu. |
| | | Information about how to |
| | | reach the COMPASS project |
| | | manager, the UNC |
| | | Institutional Review Board, |
| | | as well as the link to the |
| | | COMPASS website, are at |
| | | the bottom of the survey that |
| | | was mailed to you. |
| BEGIN SURVEY | 1-3 | Do I have your permission |
| [IF IRB MON=1] | 1=YES, CONTINUE | to continue with the |
| | 2=YES, RESPONDENT | survey? |
| | UNAVAILABLE | |
| | 3=NO, RESPONDENT | INTERVIEWER: ANSWER |
| | REFUSAL | ANY RESPONDENT |
| | REI CS/IE | QUESTIONS, AND THEN |
| | | CONTINUE. |
| THANK_YOU | GO TO INTRO | Thank you for agreeing to |
| _ | | participate in the |
| | | COMPASS study. |
| WHO DO | 1=PATIENT | WHO IS COMPLETING |
| _ | 2=PROXY, WITH | THIS SURVEY? |
| | PATIENT CONSENT | |
| | (GO TO NON-LAR | IN: A NON-LAR PROXY |
| | NAME) | IS ALLOWED ONLY IF |
| | 3=PROXY AS LEGAL | THE PATIENT |
| | AUTHORIZED | CONSENTED |
| | REPRESENTATIVE | HIM/HERSELF. |
| | | DDOVIES MUST DE AT |
| | | PROXIES MUST BE AT |
| | | LEAST 18 YEARS OLD. |
| NON-LAR NAME | OPEN TEXT | ONCE NON-LAR PROXY |
| | ENTER NON-LAR NAME | IS ON THE PHONE: |
| | | Hello, my name is [FULL |
| | | NAME] and I'm calling |
| | | regarding the COMPASS |
| | | Study, which is a research |
| | | study looking at how |
| Ĭ | | |
| | | hattents are doing after their |
| | | patients are doing after their stroke. |

| Application - IRB00033998 | T | 1 | Т |
|---|---|---|---|
| | | Mr./Ms. [LAST NAME] has already given his/her consent to participate in the study but would like for you to answer the questions on his/her behalf. Could you please tell me your first name so that I can refer to you personally? | |
| NON-LAR AGE | 1=YES (GO TO SURVEY<br>INTRO) | Are you at least 18 years old? IN: IF NO, GO BACK TO BEGIN_SURVEY AND CODE APPROPRIATELY. | |
| SCHEDULE CB_2 | OPEN TEXT<br>[200 CHAR] | When would be a better time for me to speak with him/her/you? | SCHEDULE<br>CALLBACK THEN<br>END CALL |
| RESP REF | OPEN TEXT [200 CHAR] | To help us understand how to improve our study, may I ask why you don't want to participate? | END CALL |
| REF SPEC | OPEN TEXT<br>[200 CHAR] | ENTER SPECIFICALLY<br>WHAT WAS SAID<br>ABOUT REASON FOR<br>REFUSAL | ONLY COMES UP IF REFUSAL IS FINAL (2 <sup>ND</sup> SOFT REFUSAL OR 1 <sup>ST</sup> HARD REFUSAL) |
| THANK_CB | | Thank you. We will try back another time. | Ź |
| ANSWERING MACHINE MESSAGE [IF DID ANSWER=0 AND ANSWERING MACHINE PICKS UP] | EMPTY | Hello, my name is (FULL NAME) and I am calling from the University of North Carolina on behalf of [HOSPITAL NAME]. We are trying to get in touch with [PARTICIPANT FIRST AND LAST NAME]. We'll try you back again later or you may also call us, toll-free, at 1-866-862-4636 and leave a message letting us know the best time to call. | LEAVE A MESSAGE THE FIRST TIME AN ANSWERING MACHINE IS REACHED. WAIT UNTIL THE 4TH CALL ATTEMPT TO LEAVE A SECOND MESSAGE. |

## Appendix 11 – Sustain-Arm Patient Handout –COMPASS Study Brochure

## Your recent hospital visit means that you are eligible for the COMPASS Study. Will you help us?

Your hospital is participating in a statewide study called the Comprehensive Post-Acute Stroke Services (COMPASS) Study. This study includes people who have had a stroke or transient ischemic attack (TIA), sometimes referred to as a mini-stroke. The purpose of the COMPASS Study is to determine the best ways to care for patients after they go home – to help survivors find their way forward to recovery.

In the COMPASS Study, North Carolina hospitals have been randomly assigned into two groups (similar to flipping a coin). One group of hospitals is providing patients with their usual standard of care after the patient goes home. The other group of hospitals is providing their usual care with the addition of an evaluation by a nurse practitioner, physician assistant or doctor within two weeks of hospital discharge, during which patients will receive a plan of care that will be shared with their other doctors, therapists and nurses.

#### Our hospital is providing the COMPASS model of post-acute care, which includes:

- A follow-up phone call 2 days after discharge
- A visit with a nurse practitioner, physician assistant, or doctor 7-14 days after discharge
- A plan of care that will be shared with your other health care providers
- Additional follow-up phone calls 30 and 60 days after discharge

We are committed to finding the best way to improve health and recovery after experiencing this health episode. In addition to the COMPASS care, you will continue to receive high-quality care at our hospital and at your usual follow-up visits with your primary care doctors.

After you have left the hospital, the COMPASS team would like to learn about your overall experience. They will:

- Call you in 3 months to ask questions about your recovery and satisfaction with your care.
- Mail you 3 reminder letters before you are called. The last letter will include a small gift to thank you for your time, so be sure to open it.
- Mail a survey to the family member, friend, or neighbor whom you identify as helping you in your recovery (care helper).

Whether or not you choose to participate in the survey, our hospital is committed to providing you with high-quality care for you during your recovery. All information you and your *care helper* provide will be kept strictly confidential and secure.

**If you have any questions** about the COMPASS Study, or prefer not to participate, feel free to ask the stroke coordinator, or you can call the COMPASS Study team using the toll-free number below.

COMPASS toll-free number: 1-844-501-7668
COMPASS Study website: <a href="https://www.nccompass-study.org">www.nccompass-study.org</a>



### Appendix 13 - Intervention- Arm Patient Handout -COMPASS Roadmap



#### **Appendix 14 - COMPASS Blood Pressure Log**

## **Know Your Numbers**

Prevent stroke by monitoring your blood pressure

#### **COMPASS Blood Pressure Log**

My Home Blood Pressure Goal Is: \_\_\_\_/\_\_\_

Arm monitor

Wrist monitor

My blood pressure is taken by placing the cuff on my Left arm / Right arm (circle one)





#### Things to remember about your home blood pressure monitor:

- Take your blood pressure (BP) at least 3 times per week. COMPASS recommends taking BP once a day. Take some BP's first thing in the morning before you take any of your medicines & take some BP's later in the day or evening.
- It is VERY important to bring your home BP log book to every doctor's visit.
- It is VERY important to take your BP while seated, after 5 minutes of rest, with your back supported and your feel flat around the ground. The **position matters** as otherwise you can get falsely high or low numbers.

(see quick video to review the correct position at: http://tinyurl.com/BPinstructions)

Remind your provider that you are in the COMPASS Study.

#### Alert values when your numbers may be too high/low

Some healthcare providers tell patients to call them if their blood pressure gets too high or too low. Only you and your providers can come up with those exact "alert" values, but here is some general guidance.

While monitoring your blood pressure, if you get an upper number (systolic) reading of 180 mm Hg or higher <u>OR</u> a lower number (diastolic) reading of 110 mm HG or higher, wait a couple of minutes and take it again.

If the reading is still at or above that level, you should call your provider immediately and possibly seek immediate emergency medical treatment. If you cannot access the emergency medical services (EMS), have someone drive you to the hospital right away.\*

\*This text is modified from: http://www.heart.org/HEARTORG/Conditions/HighBloodPressure/AboutHighBloodPressure/Understanding-Blood-Pressure-Readings\_UCM\_301764\_Article.jsp

| Reading 1 | | Reading 2 | | Reading 3 | | Notes |
|---|---|---|---|---|---|---|
| Date & BP | Heart<br>Rate<br>(pulse) | Date & BP | Heart<br>Rate<br>(pulse) | Date & BP | Heart<br>Rate<br>(pulse) | (from you or your provider) |
| 3/1/2016 @ 2PM<br>132/85 | 81 | 3/3/2016 @ 8 AM<br>130/80 | 70 | 3/5/2016 @ 10 PM<br>126/80 | 72 | Medication changed to 100 mg, 2 times/day |

| Reading 1 | | Reading 2 | | Reading 3 | | Notes |
|---|---|---|---|---|---|---|
| Date & BP | Heart<br>Rate<br>(pulse) | Date & BP | Heart<br>Rate<br>(pulse) | Date & BP | Heart<br>Rate<br>(pulse) | (from you or your provider) |
| 3/1/2016 @ 2PM<br>132/85 | 81 | 3/3/2016 @ 8 AM<br>130/80 | 70 | 3/5/2016 @ 10 PM<br>126/80 | 72 | Medication changed to 100 mg, 2 times/day |

| Reading 1 | | Reading 2 | | Reading 3 | | Notes |
|---|---|---|---|---|---|---|
| Date & BP | Heart<br>Rate<br>(pulse) | Date & BP | Heart<br>Rate<br>(pulse) | Date & BP | Heart<br>Rate<br>(pulse) | (from you or your provider) |
| 3/1/2016 @ 2PM<br>132/85 | 81 | 3/3/2016 @ 8 AM<br>130/80 | 70 | 3/5/2016 @ 10 PM<br>126/80 | 72 | Medication changed to 100 mg, 2 times/day |

## **Know Your Numbers**

Prevent stroke by monitoring your blood pressure

#### What is blood pressure?

The heart pumps the blood through the body through channels called blood vessels. The pressure of the blood in these vessels is the "blood pressure".

If the blood pressure is too high, then the vessels can get damaged, clogged or even rupture that can cause strokes, heart attacks, damage to your kidney as other organs.

1. Keeping your blood pressure down can reduce the risk of having another stroke!



#### NOTES:

- High blood pressure is also called hypertension, but that does not mean you are "hyper," or nervous.
- A calm person can have high blood pressure and have no idea they have it unless it is checked using a blood pressure monitor. This is why high blood pressure is called the "silent killer".



- 2. The best way to make sure your blood pressure is not too high is to check your blood pressure often using a blood pressure monitor AND
  - Keep a log of these numbers (using your COMPASS BP log)
  - Discuss your numbers with your healthcare team!

| Date/Time | Reading | 1 | Reading | 2 | Reading | 3 | Notes |
|---|---|---|---|---|---|---|---|
| | BP | Heart<br>Rate<br>(pulse) | ВР | Heart<br>Rate<br>(pulse) | BP | Heart<br>Rate<br>(pulse) | (from you or your provider) |
| Example: 8/8/11,<br>8pm | 132/85 | 81 | 130/80 | 70 | 126/80 | 72 | Medication changed to 100<br>mg, 2 times/day |



#### **NOTES:**

Other things you can do to keep your blood pressure down:

- Take your medicines right (see chapter 2)
- Eat healthier (learn about the DASH or Mediterranean Diet)
- Be more active
- Don't add salt to your food at the table (find other ways to make food taste great.



#### 3. Other important things!

- Know your goal Blood Pressure numbers
- ASK YOUR DOCTOR to tell you what your goal Upper ("systolic") and Lower (diastolic") numbers should be and write them in the Target boxes below.
- Work with your Care Coordinator to understand your blood pressure numbers, how the numbers normally change from minute to minute and when to call your doctor.



#### **NOTES:**

- You may hear that "normal" blood pressure is when the upper number is under 120 and the lower number is under 80.
- You will also here that better blood pressure "control" is when the upper number is under 150 or 140 and lower number under 90.
- But since everyone is a little different, find out what your "target" numbers are and write them in the target box.

#### Questions or concerns

| If you have any questions or co | ncerns about any symptoms you have, | or |
|----------------------------------|-------------------------------------|----|
| your medicines, talk with your h | ealth care provider or contact your | |
| Post-Acute Care Coordinator | at | |



## More about High Blood Pressure and ways to keep your blood pressure numbers in your target range:

#### What causes high blood pressure?

The exact causes are unknown. Possible causes we cannot change are age, race, sex, and family history of high blood pressure. Lifestyle factors that can cause high blood pressure are:

- Smoking
- Using too much salt
- · Being overweight or obese
- Drinking too much alcohol (more than 2 drinks for men, 1 drink for women per day)
- Using birth control pills (women)
- · Being physically inactive



High blood pressure can be treated in one or more of these ways.

- Low Salt Diet Too much salt may be part of the cause of high blood pressure for many people. Prepared foods, such as TV dinners and packaged meals, have a lot of salt. Find out the amount of salt your doctor thinks you should have each day. Read food labels on processed foods to see how much salt (sodium) is in each serving. Don't add salt at the table to foods.
- Follow a "Mediterranean-like" diet. The Mediterranean-type diet emphasizes vegetables, fruits, and whole grains and includes low-fat dairy products, poultry, fish, legumes, olive oil, and nuts. It suggests limited intake of sweets and red meats. Learn more at http://www.mayoclinic.org/healthy-lifestyle/nutrition-and-healthy-eating/indepth/mediterranean-diet/art-20047801.
- Follow the DASH Diet. The DASH plan is a diet rich in fruits, vegetables, low fat or nonfat
  dairy. It includes grains, especially whole grains; lean meats, fish and poultry; nuts and
  beans. It is high fiber and low to moderate in fat and rich in potassium, magnesium, and
  calcium. It is a plan that follows US guidelines for sodium content. The DASH eating plan
  lowers cholesterol and makes it easy to lose weight. It is a healthy way of eating, designed
  to be flexible enough to meet the lifestyle and food preferences of most people.
- Other lifestyle changes Stopping smoking, losing weight, cutting down on or not drinking alcohol and exercising regularly may be things your doctor suggests to help lower your blood pressure. If your doctor has told you to make these changes, your COMPASS Program folder will have information about each of these. If your doctor did not mention these, but you are interested in having more information, let your COMPASS post-acute coordinator know when he/she calls you for your follow-up phone calls and he/she can send you more information.

#### High Blood Pressure Medicines

**Medicines** – Your doctor may want you to take medicine to help lower high blood pressure. These may be used alone or with other medicines.







There are several types of high blood pressure medicines. Each works in a different way to lower blood pressure or help your heart. Which medicines may be best for you and your high blood pressure?

This depends on:

- The causes of your high blood pressure
- How high your blood pressure is
- How your body responds to each medicine
- · Any other health problems you have

Your doctor will look at your risk factors that may be causing your high blood pressure to find out which medicine or medicines may work best for you.

The types of medicines most often used are:

- Angiotensin-converting enzyme (ACE) inhibitors These keep your body from making
  angiotensin II. It is a hormone that makes blood vessels tighten. ACE inhibitors lower the
  amount of this hormone so your blood vessels remain relaxed. Blood flows more easily,
  lowering your overall blood pressure.
- Angiotensin II receptor blockers (ARBs) ARBs block the action of angiotensin II. This
  also relaxes blood vessels so that blood can flow more easily.
- Diuretics Often called "water pills," these will make you urinate (pass water) and help your kidneys get rid of salt and water. Less water means you have less blood volume in your blood vessels. This leads to lower blood pressure. Taking a diuretic also means less fluid collects in your feet, ankles, legs and abdomen.
- Beta-blockers –Beta-blockers slow the heartbeat and keep the heart from pumping so hard. The blood then goes through your blood vessels with less force and the pressure inside the vessels goes down.
- Calcium channel blocker (CCB) Also called a calcium antagonist. Some CCBs keep
  blood vessels from tightening so much. They do this by preventing calcium from entering the
  muscle cells in your heart and blood vessels. Others slow your heart rate. As a result, blood
  can flow more easily through the vessels. This lowers your blood pressure.
- Alpha-blockers These reduce the nerve impulses that tell your blood vessels to tighten.
   Your blood vessels remain relaxed, lowering your blood pressure.
- Alpha-agonists These target receptors in your brain to help lower blood pressure.
- Renin inhibitors Renin inhibitors block the enzyme renin from triggering a process that
  helps regulate blood pressure. Blood vessels relax and widen, making it easier for blood to
  flow through the vessels. This lowers blood pressure.
- Combination medications –There are single tablets that have two heart-related or blood
  pressure medicines to make it easier to take the medicines.

If one drug does not work for your or you do not like the way it makes you feel, others are available. Work with your doctor to find which ones are best for you. Many people need more than one type of blood pressure medicine to get the best results.

Resources for this information include: National Heart, Lung and Blood Institute, NIH – nhlbi.nih.gov/health/health-topics/topics/hbp; Your Guide to Lowering High Blood Pressure – nhlbi.nih.gov/hbp/; mayoclinic.com/health/high-blood-pressure/DS00100; The DASH Diet - /





# March 19, 2021 Application - IRB00035998 Appendix 16 - Two-Day Post-Discharge Follow-up

| - | COMPREHENSIVE POST-ACUTE STROKE SERVICES Two-Day Post-Discharge Follow-Up |
|---|---|
| IL | D Number: Form Code: 2 D A Y Date: 7JUN2016 Version 1.0 |
| AD | MINISTRATIVE INFORMATION (0a-0b are auto-populated) |
| 0a. | Completion Date: / Ob. Staff ID: |
| A. | Hi. My name is, and I am calling on behalf of the stroke team of (name of hospital from which patient was discharged). May I speak to (patient name)? |
| | <ul> <li>☐ Yes, patient is available → Go to Question 1</li> <li>☐ No, patient is not currently available → Go to Section B</li> </ul> |
| | <ul> <li>No, patient is not currently available</li> <li>So to Section B</li> <li>No, patient is deceased</li> <li>→ End Two-Day Post-Discharge Follow-Up</li> <li>No, patient is hospitalized</li> <li>→ End Two-Day Post-Discharge Follow-Up</li> </ul> |
| | □ No, patient is in a skilled nursing facility → End Two-Day Post-Discharge Follow-Up |
| В. | May I please speak to (patient name)'s primary caregiver? |
| | ☐ Yes → Go to Section D ☐ No → Go to Section C |
| C. | May I please get the primary caregiver's name and number? |
| | Name of the primary caregiver: |
| | <ul> <li>☐ I don't know the primary caregiver's name or number</li> <li>☐ No, I refuse to provide caregiver's number</li> </ul> |
| | Number of primary caregiver: () |
| | <ul> <li>☐ I don't know the primary caregiver's name or number</li> <li>☐ No, I refuse to provide caregiver's number</li> </ul> |
| | → End Two-Day Post-Discharge Follow-Up |
| | (Patient name) was discharged from the hospital approximately two days ago, and I would like to follow up with you to see how he/she has been doing. |
| | To whom am I speaking with? Name: |
| | D (a). What is your relationship with (patient name)? □ Spouse |
| | ☐ Spodse ☐ Sibling ☐ Son/Daughter |
| | ☐ Neighbor/Friend |
| | <ul><li>□ Parent/Legal Guardian</li><li>□ Other → Go to Question E (c)</li></ul> |

| D (c). Does the (patient name) have communication challenges that prevent him/her from answering questions? No Yes, significant aphasia Yes, cognitive deficits Both, significant aphasia & cognitive deficits No response |
|---|
| → Go to Question 1 |
| The Post – Acute Care Coordinator will now ask the following open-ended questions of the patient: You were discharged from the hospital approximately two days ago, and I would like to follow up with you to see how you have been doing |
| <ol> <li>I would like to discuss your medications and any changes that have been made. (Obtain medication list. Complete medication reconciliation, and list any discrepancies). Was medication reconciliation completed? ☐ Yes → Go to Question 1a</li> </ol> |
| □ No → Go to Question 1c |
| <ul><li>1a. Were there any discrepancies during medication reconciliation?</li><li>☐ Yes</li><li>☐ No → Go to Question 2</li></ul> |
| 1b |
| 1c. Why was medication reconciliation not completed? |
| 2. Do you have any concerns about your medications? ☐ Yes ☐ No → Go to Question 3 |
| 2a. What are these concerns? |
| ☐ No Response |
| <ul><li>3. Are you on Coumadin (Warfarin)?</li><li>☐ Yes</li><li>☐ No → Go to Question 4</li></ul> |
| 3a. Have you had a test to see how long it takes for your blood to clot? This is known as an INR test. ☐ Yes ☐ No → Go to Question 4 |
| 3b. What is your INR (Typical normal range 2-3)? ☐ ☐ I don't know ☐ No response |
| 3c. When did you have your INR test? |
| Month Day Year |
| 2-Day Post-Discharge Follow-Up |

| Numbness or weakness of the face, arm, or leg, especially on one side of the body Confusion / trouble understanding | lo<br>onse |
|---|---|
| <ul> <li>No response</li> <li>4. Have you had any new stroke symptoms since being discharged from the hospital? Yes</li></ul> | |
| 4. Have you had any new stroke symptoms since being discharged from the hospital? ☐ Yes ☐ No → Go to Question 5 4a. What are these new symptoms? Yes No Respondent of the body ☐ | |
| Yes □ No → Go to Question 5 4a. What are these new symptoms? Yes No Responded for the face, arm, or leg, especially on one side of the body Confusion / trouble understanding | |
| 4a. What are these new symptoms? Yes No Respond to Question 5 Numbness or weakness of the face, arm, or leg, especially on one side of the body Confusion / trouble understanding | |
| ☐ Yes ☐ No → Go to Question 5 4a. What are these new symptoms? Yes No Responded in the body Confusion / trouble understanding ☐ ☐ ☐ ☐ ☐ ☐ ☐ ☐ ☐ ☐ ☐ ☐ ☐ ☐ ☐ | |
| Numbness or weakness of the face, arm, or leg, especially on one side of the body Confusion / trouble understanding | |
| Numbness or weakness of the face, arm, or leg, especially on one side of the body Confusion / trouble understanding | |
| Numbness or weakness of the face, arm, or leg, especially on one side of the body Confusion / trouble understanding | |
| Numbness or weakness of the face, arm, or leg, especially on one side of the body Confusion / trouble understanding | 000 |
| Side of the body Confusion / trouble understanding | |
| , , , | |
| 3 | |
| Severe headache | |
| No response | |
| 5. After being discharged from the hospital, some stroke survivors may need a primary careg | ver to |
| provide assistance with activities such as taking your medicines, bathing, dressing, perform | |
| housework, and/or going places around town. Is there a primary caregiver who is currently | |
| you with these tasks? | |
| ☐ Yes ☐ No → Go to Question 6 | |
| Fig. What activities is your primary caregiver assisting with? | |
| 5a. What activities is your primary caregiver assisting with? | |
| Yes No Response | |
| Medication management | |
| Assisting with ADLs (bathing, dressing, feeding, etc.) | |
| Assisting with IADLs (cooking, housework, shopping, etc.) | |
| None | - |
| No response | |
| | <del></del> |
| 5b. What is the name of the primary caregiver? | |
| 5b. What is the name of the primary caregiver? No response | |
| □ No response | |
| <ul> <li>□ No response</li> <li>5c. What is the primary caregiver's relationship to you?</li> <li>□ Spouse</li> <li>□ Sibling</li> </ul> | |
| <ul> <li>□ No response</li> <li>5c. What is the primary caregiver's relationship to you?</li> <li>□ Spouse</li> <li>□ Sibling</li> <li>□ Son/Daughter</li> </ul> | |
| <ul> <li>□ No response</li> <li>5c. What is the primary caregiver's relationship to you?</li> <li>□ Spouse</li> <li>□ Sibling</li> <li>□ Son/Daughter</li> <li>□ Neighbor/Friend</li> </ul> | |
| <ul> <li>□ No response</li> <li>5c. What is the primary caregiver's relationship to you?</li> <li>□ Spouse</li> <li>□ Sibling</li> <li>□ Son/Daughter</li> <li>□ Neighbor/Friend</li> <li>□ Parent/Legal Guardian</li> </ul> | |
| <ul> <li>□ No response</li> <li>5c. What is the primary caregiver's relationship to you?</li> <li>□ Spouse</li> <li>□ Sibling</li> <li>□ Son/Daughter</li> <li>□ Neighbor/Friend</li> </ul> | |
| <ul> <li>No response</li> <li>What is the primary caregiver's relationship to you?</li> <li>Spouse</li> <li>Sibling</li> <li>Son/Daughter</li> <li>Neighbor/Friend</li> <li>Parent/Legal Guardian</li> <li>Other → Go to Question 7d</li> <li>No response</li> </ul> | |
| <ul> <li>No response</li> <li>5c. What is the primary caregiver's relationship to you?</li> <li>Spouse</li> <li>Sibling</li> <li>Son/Daughter</li> <li>Neighbor/Friend</li> <li>Parent/Legal Guardian</li> <li>Other → Go to Question 7d</li> </ul> | |
| □ No response 5c. What is the primary caregiver's relationship to you? □ Spouse □ Sibling □ Son/Daughter □ Neighbor/Friend □ Parent/Legal Guardian □ Other → Go to Question 7d □ No response 5d. Specify "other": | |
| <ul> <li>No response</li> <li>What is the primary caregiver's relationship to you?</li> <li>Spouse</li> <li>Sibling</li> <li>Son/Daughter</li> <li>Neighbor/Friend</li> <li>Parent/Legal Guardian</li> <li>Other → Go to Question 7d</li> <li>No response</li> </ul> | |
| <ul> <li>No response</li> <li>5c. What is the primary caregiver's relationship to you?</li> <li>Spouse</li> <li>Sibling</li> <li>Son/Daughter</li> <li>Neighbor/Friend</li> <li>Parent/Legal Guardian</li> <li>Other → Go to Question 7d</li> <li>No response</li> <li>5d. Specify "other":</li> <li>Do you have a follow-up appointment scheduled with your primary care provider?</li> <li>Yes</li> <li>No → Go to Question 7</li> </ul> | |
| <ul> <li>No response</li> <li>5c. What is the primary caregiver's relationship to you?</li></ul> | |
| <ul> <li>No response</li> <li>5c. What is the primary caregiver's relationship to you?</li> <li>Spouse</li> <li>Sibling</li> <li>Son/Daughter</li> <li>Neighbor/Friend</li> <li>Parent/Legal Guardian</li> <li>Other → Go to Question 7d</li> <li>No response</li> <li>5d. Specify "other":</li> <li>Oo you have a follow-up appointment scheduled with your primary care provider?</li> <li>Yes</li> <li>No → Go to Question 7</li> <li>I don't know → Go to Question 7</li> </ul> | 2 - 6 2 |
| <ul> <li>No response</li> <li>5c. What is the primary caregiver's relationship to you?</li> <li>Spouse</li> <li>Sibling</li> <li>Son/Daughter</li> <li>Neighbor/Friend</li> <li>Parent/Legal Guardian</li> <li>Other → Go to Question 7d</li> <li>No response</li> <li>5d. Specify "other":</li> <li>Oo you have a follow-up appointment scheduled with your primary care provider?</li> <li>Yes</li> <li>No → Go to Question 7</li> <li>I don't know → Go to Question 7</li> </ul> | age 3 of 6 |

| 6a. What is the date and time of your follow-up visit at your primary care provider? |
|---|
| Month Day Year |
| ☐ I don't know ☐ No response |
| 6b. What is the first and last name of your primary care provider? □ □ I don't know □ No response |
| <ul> <li>7. Do you have a follow-up appointment scheduled with our comprehensive stroke clinic? (Post-Acute Care Coordinator will need to have appointment date readily available).</li> <li>☐ Yes, I do have an appointment → Go to Question 8</li> <li>☐ No, I don't have an appointment (Post-Acute Care Coordinator will confirm an appointment was not established) → Go to Question 9</li> </ul> |
| <ul> <li>☐ I don't know if I have an appointment (Post-Acute Care Coordinator will confirm appointment or establish an appointment)</li> <li>→ Go to Question 11</li> </ul> |
| <ul> <li>8. What is the date and time of your follow-up visit at our Comprehensive Stroke Clinic?</li> <li>□ Patient confirmed date and time correctly → Go to Question 11</li> <li>□ Patient didn't confirm date/time correctly or patient didn't know date/time → Go to Q 10</li> </ul> |
| 9. I will now establish an appointment for you to our Comprehensive Stroke Clinic. Your appointment is on (XX/XX/XXXX) at (XX:XX AM/PM). Did appointment get established? ☐ Yes → Go to Question 11 ☐ No |
| 9a. Why did appointment not get established? Patient prefers to follow-up with his/her own PCP or another doctor Patient reported that he/she is too sick or disabled to attend Patient cannot afford to attend the 7-14 day visit Patient does not have transportation Patient reported that he/she lives out of the area & doesn't want to travel No available appointment within 14 days Other: |
| 10. Your appointment at our Comprehensive Stroke Clinic is on (XX/XX/XXXX) at (XX:XX AM/PM) Did confirmation take place? ☐ Yes ☐ No |
| 11. Have you had any falls since your discharge? ☐ Yes ☐ No → Go to Question 11a |
| 11a. Did you sustain any injuries and have to go to the emergency room or see a doctor? ☐ Yes ☐ No ☐ No response |
| 12. Were you prescribed home health services after hospital discharge? ☐ Yes ☐ No → Go to Question 13 ☐ I don't know → Go to Question 13 |
| 2-Day Post-Discharge Follow-Up |

| 12a. What home health agency will provide | you with home | health care? | | |
|---|---|---|---|---|
| □ | | | | |
| 12b. What service(s) has been scheduled? | | | | |
| | Yes | No | N/A | |
| Home health PT | <u> </u> | | <u> </u> | |
| Home Health OT | | <del> </del> | | |
| Home Health SLP | | <del></del> | <del></del> | |
| Home Health Nursing No response | | | | |
| 140 response | _ ⊔ | 1 | | |
| 12c. Do you plan to receive and continue tl<br>☐ Yes ☐ No | ☐ No respon | se | | |
| 12d. [If a service(s) has not been scheduled ☐ I chose not to participate in home ☐ The home health agency has not ☐ Other | e health service | es | | |
| → Go to Question 14 | | | | |
| 13. Were you prescribed any outpatient therapy ☐ Yes ☐ No → Go to Qu | | discharge? | | |
| 13a. What service(s) has been scheduled? | | | | |
| | Yes | No | N/A | |
| Outpatient OT | | | | |
| Outpatient PT | | | | |
| Outpatient SLP | | | | |
| No response | | | | |
| 13b. Do you plan to attend and continue the scheduled? ☐ Yes ☐ No ☐ No | e therapy servio | ce(s) or appoint | ment(s) that ha | ve been |
| 13c. [If a service(s) has not been scheduled ☐ I chose not to participate in outpa ☐ There were not any available app ☐ Other | atient services | | | |
| You had a stroke, and it's important to rememb<br>to the emergency department. An easy way to r<br>Face. Look for an uneven smile.<br>Arm. Check if one arm is weak or numb.<br>Speech. Listen for slurred speech.<br>Time. Call 911 immediately. | | | | I when to go |
| 14. As a reminder, attending your appointment recovery, health, and independence. Do yo from attending your appointment? □ Yes → Go to Section F □ No | u have any iss | ues with transpo | | |
| 2-Day Post-Discharge Follow-Up | | | | |

| | ing the time to answer these follow- | | eduled you to |
|---|---|---|---|
| 15. Are there any o | | on reconciliation, or any conc | |
| 15a. What are | these challenges or concerns? | | |
| | END OF 2-DAY POST-DISCH | ARGE FOLLOW-UP | |

# March 19, 2021 Application - IRB00035998 Appendix 17 - Post-stroke Functional Assessment

| A LCOMPACC | |
|---|---|
| COMPASS Post-Stroke Functional Assessment | tor |
| COMPREHENSIVE POST-ACUTE STROKE SERVICES Personalized Care® | |
| For Each Patient, the "Right Care, Right Place, R | ight Time" |
| ID Number: Form Code: P S F A Date: 2JUN2016 | Version 1.0 |
| ADMINISTRATIVE INFORMATION (0a-0b are auto-populated) | |
| 0a. Completion Date: Day / Day / Year Ob. Staff ID: | |
| We are going to ask you a series of questions about your health and well-being, and your care of yourself and move around since your stroke. Some questions will also ask you about preferences for care. The goal is to share this information with your doctors, nurses, and that they can develop a care plan made especially for you. Please answer the following que the state of your health or function and the activities you would prefer to do to help you restay healthy. | out your<br>therapists so<br>lestions on<br>cover and |
| <ol> <li>Since you were hospitalized for your stroke, have you had enough to buy your medicines and<br/>your doctor prescribed?</li> <li>☐ Yes</li> <li>☐ No</li> <li>☐ No response</li> </ol> | take them as |
| 2. Do you know any of the risk factors that may lead to a stroke? $\Box$ Yes $\Box$ No $\rightarrow$ Go | to Question 3 |
| 2a. What are these risk factors? (check all that apply) ☐ High Blood Pressure ☐ Smoking ☐ Diabetes or High Blood Sugar | |
| <ul> <li>☐ Irregular Heart Beat (Atrial Fibrillation)</li> <li>☐ Heart Disease</li> <li>☐ High Cholesterol</li> <li>☐ Physical Inactivity</li> </ul> | |
| <ul> <li>☐ Sickle Cell Anemia</li> <li>☐ Family History of Stroke</li> </ul> | |
| <ul><li>☐ Prior Stroke</li><li>☐ Response not on this list</li></ul> | |
| 2b. Did the patient know <u>any</u> of the risk factors for stroke? ☐ Yes ☐ No | |
| Post Stroke Functional Assessment | Page 1 of 8 |

| 3. Compared to others your age, how would you rate your with 1 being "poor" and 5 being "excellent?" | health since your stroke using a scale of 1 to 5, |
|---|---|
| (1) Poor (2) Fair (3) Good (4) Very Good | (5) Excellent ☐ No response |
| 4. Can you go up and down 10 stair steps without help? | ☐ Yes ☐ No ☐ No response |
| 5. How difficult is it to use your hand most affected by your | r stroke? |
| (1) Cannot use at all (2) Very difficult (3) Somewhord ☐ No response | at difficult (4)A little difficult (5) Not difficult at all |
| 6. Have you fallen in the last 3 months? ☐ Yes | □ No → Go to Question 8 |
| 6a. In the last 3 months, did you get injured and nee<br>room due to a fall?<br>☐ Yes ☐ No ☐ No respons | end data → ecotorio ener subsensitori supre cerdane a Francia . |
| 6b. Have you fallen more than once in the last 3 more | onths? ☐ Yes ☐ No ☐ No response |
| 7. Have you fallen since your stroke? ☐ Yes ☐ No | → Go to Question 8 |
| 7a. How many times have you fallen since your strok | ke? □ don't know □ No response |
| 8. Please continue this sequence: 1, A, 2, B, 3, C, _, _, _, . | نات |
| Choose "yes" if the patient completed the entire sequen ☐ Yes ☐ No ☐ No respons | |
| 9. How many different medications do you take per day? | □ don't know □ No response |
| 10. Is there someone to help you move about, bathe, dress, ☐ Yes ☐ No → Go to Question | |
| 10a. What relationship is he/she to you? ☐ Spouse ☐ Sibling ☐ Son/Daughter ☐ Neighbor/Friend ☐ Parent/Legal Guardian ☐ Other (Specify) → Specify other in 10b ☐ No response | |
| 10b. Specify other: | |
| Post Stroke Functional Assessment | Page 2 of 8 |

| ☐ Yes ☐ No ☐ No respons | | | | |
|---|---|---|---|---|
| 12. Since your stroke, have you often been bothered by littl ☐ Yes ☐ No ☐ No respons | | r pleasure | in doing th | nings? |
| f the following criteria are met: Question 1: Yes Question 2: Yes or No Question 2b: Yes or No Question 3: (3) Good or (4) Very Good or (5) Excellent Question 4: Yes Question 5: (4) A little difficult or (5) Not difficult at all Question 6: No Question 8: Yes Question 9: 4 or less Question 10: Yes Question 11: No Question 12: No | Only the<br>Question<br>Question<br>Question<br>Question | 14<br>126-27<br>134-38<br>142-43 | question | s will be asked: |
| f the above criteria are met, BUT<br>Question 11: Yes<br>OR<br>Question 12: Yes | Only the Question Question Question Question Question Question Question | 14<br>126-27<br>134-38<br>140-41<br>142-43 | question | s will be asked: |
| 13. Over the next 3 months, do you think your health is goin Improve Stay the same Get worse No response 14. What are your primary reasons for staying as healthy a (Open-ended question) For example, | | | | |
| | | Yes | No | No Response |
| Work – return to work | | | | |
| Social – visit with friends, go out, and/or travel | | | | |
| Family – visit with family, play with my grandchildren | | | | |
| Independence – be independent, take care of myself | | | | |
| Better quality of life | | | | |
| Other → Specify other in 14b | | | | |
| No response | | | | l |

| 10. | Can you v | rest? | 15 minutes wi | vithout getting short of breath or needing to | |
|---|---|---|---|---|---|
| | | ☐ Yes | □ No | ☐ No response | |
| 16. | Can you | walk without fee<br>□ Yes | ling unsteady′<br>□ No | /?<br>□ No response | |
| 17. | Can you g | get up out of a c<br>□ Yes | thair <b>without</b> u<br>□ No | using your hands? □ No response | |
| 18. | Can you ı | use the phone to<br>□ Yes | o call your fam<br>□ No | mily or doctor if needed?<br>□ No response | |
| 19. | Can you լ | orepare your ow<br>□ Yes | n meals or do<br>□ No | o your own housework without any assistance?<br>□ No response | |
| 20. | Can you l | oathe/take a sho<br>□ Yes | ower and dres<br>□ No | ss yourself without any assistance?<br>□ No response | |
| 21. | Are you h | aving trouble co<br>□ Yes | ontrolling your<br>□ No | r bladder or bowels? □ No response | |
| que<br>que | stions ab | out this area o | f your life. Th | rtant for managing your health, I am going to ask a few<br>here really is no right or wrong answer. These are helpful<br>urses to help you have the assistance you need to manage | your |
| que<br>que<br>hea<br>22. | estions ab<br>estions to<br>alth.<br>Can you t | out this area o<br>assist your do | f your life. The ctors and number of the week, m | here really is no right or wrong answer. These are helpful urses to help you have the assistance you need to manage nonth, and year? (Choose "Yes" if the patient was able to corre | |
| que<br>que<br>hea<br>22. | estions ab<br>estions to<br>lith.<br>Can you t<br>identify da<br>n going to | out this area of assist your do assist your do sell me the day of the week, rule Yes | f your life. The ctors and number of the week, me month, and year one Nowords to you | here really is no right or wrong answer. These are helpful urses to help you have the assistance you need to manage month, and year? (Choose "Yes" if the patient was able to correctar.) | ctly<br>nen I |
| que<br>que<br>hea<br>22. | estions ab<br>estions to<br>lith.<br>Can you t<br>identify da<br>n going to | out this area of assist your do assist your do sell me the day of the week, rule Yes | f your life. The ctors and numer of the week, me month, and year of No words to you y words as you | here really is no right or wrong answer. These are helpful urses to help you have the assistance you need to manage month, and year? (Choose "Yes" if the patient was able to correct.) No response I that you will have to remember. Please listen carefully. Whou can remember. It doesn't matter in what order you say to | ctly<br>nen I |
| que<br>que<br>hea<br>22. | estions ab<br>estions to<br>alth.<br>Can you t<br>identify da<br>n going to<br>through, | out this area of assist your do assist your do dell me the day of the week, roughly of the week, roughly read a list of verepeat as many arrial 1: School | f your life. The ctors and number of the week, me month, and year of No words to you y words as you, blue, apple. | here really is no right or wrong answer. These are helpful urses to help you have the assistance you need to manage month, and year? (Choose "Yes" if the patient was able to correct.) No response I that you will have to remember. Please listen carefully. Whou can remember. It doesn't matter in what order you say to | ctly<br>nen I |
| que<br>que<br>hea<br>22. | estions ab<br>estions to<br>alth.<br>Can you t<br>identify da<br>n going to<br>through, | out this area of assist your do assist your do dell me the day of the week, roughly of the week, roughly read a list of verepeat as many arrial 1: School | f your life. The ctors and number of the week, me month, and year of No words to you y words as you, blue, apple. | here really is no right or wrong answer. These are helpful urses to help you have the assistance you need to manage month, and year? (Choose "Yes" if the patient was able to corregar.) No response I that you will have to remember. Please listen carefully. Whou can remember. It doesn't matter in what order you say to | ctly<br>nen I |
| que<br>que<br>hea<br>22. | estions ab<br>estions to<br>oth.<br>Can you to<br>identify da<br>n going to<br>through, | out this area of assist your do assist your do dell me the day of the week, red a list of vere at as many are at the list for the read the list for the area of the list for the area of the list for the area of the list for the list for the area of the area of | f your life. The ctors and number of the week, month, and year No No words to you y words as you, blue, apple. or a second ti , blue, apple. | here really is no right or wrong answer. These are helpful urses to help you have the assistance you need to manage month, and year? (Choose "Yes" if the patient was able to corregar.) No response I that you will have to remember. Please listen carefully. Whou can remember. It doesn't matter in what order you say to | ctly<br>nen I |
| que que hea 22. I an am I wi 23. | estions ab<br>estions to<br>lith. Can you to<br>identify da<br>n going to<br>through, If ask you Tell me w | out this area of assist your do assist your do dell me the day of the week, repeat a list of a repeat as many. Trial 1: School aread the list for the control of the second the second to recall these | f your life. The ctors and number of the week, month, and year No words to you y words as you, blue, apple. or a second tie, blue, apple. words again ag two of your | here really is no right or wrong answer. These are helpful urses to help you have the assistance you need to manage month, and year? (Choose "Yes" if the patient was able to correcar.) No response I that you will have to remember. Please listen carefully. Whou can remember. It doesn't matter in what order you say to time. Repeat as many words as you can. | ctly<br>nen I<br>hem. |
| que que hea 22. I an am I wi 23. | estions ab<br>estions to<br>lith. Can you to<br>identify da<br>n going to<br>through, If ask you Tell me w | out this area of assist your do assist your do dell me the day of the week, red a list of veread a list of veread as many. Trial 1: School read the list for the | f your life. The ctors and number of the week, month, and year No words to you y words as you, blue, apple. or a second tie, blue, apple. words again ag two of your | here really is no right or wrong answer. These are helpful urses to help you have the assistance you need to manage month, and year? (Choose "Yes" if the patient was able to corresear.) No response I that you will have to remember. Please listen carefully. Whou can remember. It doesn't matter in what order you say to time. Repeat as many words as you can. | ctly<br>nen I<br>hem. |

| | etc).<br>□ Yes | □ No | ☐ No response |
|---|---|---|---|
| 25. In the la | ast month, <b>were</b><br>□ Yes | you unable to<br>□ No | to buy your medicines because of not having enough money? ☐ No response |
| 26. Do you | stop taking you<br>□ Yes | r medicine if yo<br>□ No | rou feel better or worse? □ No response |
| 27. Do you | ever forget to tal Often Sometime Rarely Never No respon | es | sine? |
| | | | l you to remember. It doesn't matter in what order you list them.<br>ecall all 3 words : school, blue, apple).<br>☐ No response |
| 29. Since y | our stroke, do y<br>□ Yes | ou eat at least<br>□ No | t two meals a day?<br>□ No response |
| 30. Since y | our stroke, have<br>□ Yes | you had new<br>□ No | problems swallowing or chewing your food? ☐ No response |
| | rour stroke, have<br>s of daily living?<br>□ Yes | you had incre | eased stiffness in your hand, arm, or leg that interferes with your No response |
| 32. Since yo | our stroke, have<br>□ Yes | you been able<br>□ No | e to drive yourself to and from places?<br>☐ No response |
| 33. If unabl | e to drive, is the<br>□ Yes | re someone w<br>□ No | vho can take you to the doctor or pharmacy?<br>☐ No response |
| 34. Do you | have one docto<br>☐ Yes | | you and all of your medical conditions? Go to Question 39 |
| 35. What is | the doctor's firs | t and last Nan | me? □ don't know □ No response |
| 36. Have y | ou seen him/her<br>□ Yes | | months? Go to Question 38 |
| 37. Have yo | ou seen him <i>l</i> her<br>□ Yes | since your stro<br>□ No | oke? □ No response |
| | act 2 months di | d vou miss an | y scheduled appointments with this doctor? |

| | ork of family and friends who<br>am often lonely<br>can count on my family and<br>sponse | | | /n |
|---|---|---|---|---|
| | ation in which a person feels<br>or her mind is troubled all th | | | |
| □ Yes | □ No □ Nor | esponse | | |
| 41. Since your stroke h<br>□ Yes | as your relationship with you<br>□ No □ No r | r family become mo<br>esponse | ore difficult or s | tressed? |
| 42. In the last 3 months, department? | with the exception of your s | troke, how many tir | nes were you s | seen in the emergency |
| | □ don't know | ☐ No response | | |
| hospitalization due t | □ don't know<br>ervices are you currently rec | □ No response | | |
| | | Yes | No | No Boonones |
| None → C | So to Question 45 | res | INO | No Response |
| Nursing | o to Quodion 10 | | | |
| Physical Th | erapy | | | |
| Occupation | al Therapy | | | |
| Speech & L | anguage Therapy | | | |
| 1,000,000,000,000 | are Assistant | | | |
| No respons | e → Go to Question 45 | | | |
| 45. What type of outpati<br>( <b>Open-ended ques</b> | ent therapy are you currently | receiving? | No | No Poononos |
| None | | Tes | 140 | No Response |
| | Physical Therapy | | | |
| Outballeni | Occupational Therapy | | | |
| | anguage Therapy | | | |
| Outpatient ( | | | _ | |
| Outpatient ( | | * | · | [098] |

| (Open-ended question) | Yes | No | No<br>Response |
|---|---|---|---|
| None | | | • |
| Walker | | | |
| Cane | | | |
| Wheelchair | | | |
| Bath Safety Equipment (Toilet rails/frames, shower bench/seat) | | | |
| Bedside Commode | | | |
| No response | | | |
| <ul> <li>□ Telephone call → If checked, answer 4</li> <li>□ Text message → If checked, answer 4</li> <li>□ Email → If checked, answer 4</li> <li>□ I will visit My Health portal on the internet</li> <li>□ No response</li> </ul> | 7a<br>7b | | |
| a. What is the best number to reach you? | | don't know | ☐ No response |
| b. What is your email address? | 🗆 don't knov | v □ No res | sponse |
| our doctor and nurses want to take good care of you a<br>vants to make sure he/she understands your views on<br>lecause unexpected things can happen, you have the r<br>his includes the right to accept or refuse medical or su<br>lose the ability to participate in decision-making about<br>ight to plan and direct the types of healthcare and life | treatment so they o<br>ight to make decis<br>urgical treatment w<br>your own treatmen<br>sustaining treatme | can take god<br>ions about y<br>hen you are<br>t. Fortunate<br>nts you wish | od care of you. your healthcare. seriously ill or ly, you have the to receive in |
| rants to make sure he/she understands your views on<br>lecause unexpected things can happen, you have the i<br>his includes the right to accept or refuse medical or si<br>ose the ability to participate in decision-making about | treatment so they o<br>ight to make decis<br>urgical treatment w<br>your own treatmen<br>sustaining treatme | can take god<br>ions about y<br>hen you are<br>t. Fortunate<br>nts you wish | od care of you. your healthcare. seriously ill or ly, you have the to receive in |
| vants to make sure he/she understands your views on<br>because unexpected things can happen, you have the i<br>his includes the right to accept or refuse medical or si<br>ose the ability to participate in decision-making about<br>ight to plan and direct the types of healthcare and life<br>the future. You can do this by making an advance direc | treatment so they oright to make decisurgical treatment wyour own treatmen sustaining treatme tive (living will). Ar | can take god<br>ions about y<br>hen you are<br>t. Fortunate<br>nts you wish | od care of you. your healthcare. seriously ill or ly, you have the to receive in |
| vants to make sure he/she understands your views on lecause unexpected things can happen, you have the inhis includes the right to accept or refuse medical or subset he ability to participate in decision-making about hight to plan and direct the types of healthcare and lifes the future. You can do this by making an advance direct ou a voice in decisions about your medical care. | treatment so they oright to make decisurgical treatment wyour own treatment sustaining treatmetive (living will). Ar | can take god<br>ions about y<br>hen you are<br>t. Fortunate<br>nts you wish<br>advance di | od care of you. your healthcare. seriously ill or ly, you have the to receive in |
| vants to make sure he/she understands your views on because unexpected things can happen, you have the inhis includes the right to accept or refuse medical or subset he ability to participate in decision-making about 1 ght to plan and direct the types of healthcare and life inhe future. You can do this by making an advance direct ou a voice in decisions about your medical care. 8. Do you have a living will? Yes Go to Question 48a. Would you be interested in information to assis | treatment so they oright to make decisurgical treatment wyour own treatmen sustaining treatme tive (living will). Ar | can take god<br>ions about y<br>hen you are<br>t. Fortunate<br>nts you wish<br>a advance di | od care of you. your healthcare. seriously ill or ly, you have the to receive in |
| vants to make sure he/she understands your views on lecause unexpected things can happen, you have the inhis includes the right to accept or refuse medical or subset the ability to participate in decision-making about the ght to plan and direct the types of healthcare and lifes not future. You can do this by making an advance direct out a voice in decisions about your medical care. 8. Do you have a living will? □ Yes → Go to Question 48a. Would you be interested in information to assis □ Yes □ No □ No respons 9. Did someone other than the patient answer the majority | treatment so they oright to make decisurgical treatment wyour own treatmen sustaining treatme tive (living will). Ar | can take god<br>ions about y<br>hen you are<br>t. Fortunate<br>nts you wish<br>a advance di | od care of you. your healthcare. seriously ill or ly, you have the to receive in |
| vants to make sure he/she understands your views on the cause unexpected things can happen, you have the inhis includes the right to accept or refuse medical or stope the ability to participate in decision-making about the ght to plan and direct the types of healthcare and life she future. You can do this by making an advance direct ou a voice in decisions about your medical care. 8. Do you have a living will? □ Yes → Go to Question 48a. Would you be interested in information to assis □ Yes □ No □ No respons 9. Did someone other than the patient answer the majority □ Yes □ No 49a. What was their relationship to the patient? □ Spouse □ Sibling □ Son/Daughter □ Neighbor/Friend □ Parent/Legal Guardian □ Other (Specify) → Specify other in 49b | treatment so they oright to make decisurgical treatment wyour own treatmen sustaining treatme tive (living will). Ar | can take god<br>ions about y<br>hen you are<br>t. Fortunate<br>nts you wish<br>a advance di | od care of you. your healthcare. seriously ill or ly, you have the to receive in |

| What supp<br>you? | ort/services do you have to help you? And what resources would you like to receive i | n order to help |
|---|---|---|
| provider (<br>services t | ifor responding to our questions. I am going to discuss your questionnaire wi<br>nurse practitioner/physician assistant/physician) and use your responses to ar<br>hat will be useful to ensure the best possible<br>overy. Do you have any questions for me? | |
| [The ques<br>Site] | tion and checklist below will only be completed at Wake Forest Baptist Medical | Center – Vangua |
| | pleted by the interviewer. Which of the following factors do you think this patient will r with to speed their stroke recovery? | need help or |
| | Activities of Daily Living (Bathing, dressing, walking) | |
| | Exercise to improve strength, balance, and endurance | |
| | Falls prevention | |
| | Durable medical equipment or home modifications | |
| | Transportation to follow-up appointments | |
| | Manage medications (pill box, etc) | |
| | Monitor/control of stroke risk factors (blood pressure, hypertension) | |
| | Pharmacy referral | |
| | Financial assistance to purchase medications | |
| | Depression services, treatment, and support | |
| | Patient doesn't have a primary care physician & needs help getting one | |
| | Identify caregiver to assist & be available during instructions | |
| | Refer to Outpatient Therapy ( PT/OT) | |
| | Refer to Speech and Language | |
| | Refer to Home Health Services | |
| | Refer to Skilled Nursing Home Refer to Community Services | |
| | Assistance with Advance Directive | |
| | Nutritional support | |
| | None | |
| | Thank you! | |
| | Thanks for completing this questionnaire! | |
| | Go out and live the best day possible. | |
| | You deserve it. | |
| | END OF POST STROKE FUNCTIONAL ASSESSMENT | |

## Appendix 18 - Caregiver Assessment

| V | COMPASS COMPREHENSIVE POST-ACUTE STROKE SERVICES Stroke Caregiver Assessment® For Each Caregiver the "Right Care at the Right Time" |
|---|---|
| ID N | umber: Form Code: S C A Date: 27MAR2016 Version 1.0 |
| ADMIN | IISTRATIVE INFORMATION (0a-0c are auto-populated) |
| 0a. Cor | npletion Date: Day / Staff ID: Ob. Staff ID: |
| 0c. Car | egiver ID: |
| liv | tient name] has indicated that he/she has assistance with some, or all, routine activities of daily<br>ng and that he/she depend on the help of a caregiver. Are you [patient name]'s primary<br>egiver? |
| | ☐ Yes → Go to Section C ☐ No → Go to Section B |
| | o is the patient's primary caregiver, and what is the best number I can reach him/her? (Obtain and number so that Post-Acute Care Coordinator can call primary caregiver). |
| | Name of the authors are experienced |
| | Name of the primary caregiver: |
| | Name of the primary caregiver: |
| na | |
| na<br>qu | Number of primary caregiver: ()ce you are the primary caregiver, I would like to discuss the services and tasks that [patient me] needs assistance with during his/her stroke recovery. Do you have time to answer a few |
| na<br>qu<br>1. | Number of primary caregiver: ()ce you are the primary caregiver, I would like to discuss the services and tasks that [patient me] needs assistance with during his/her stroke recovery. Do you have time to answer a few estions? This will take about 5 minutes to complete. |
| na<br>qu<br>1. | Number of primary caregiver: () ce you are the primary caregiver, I would like to discuss the services and tasks that [patient me] needs assistance with during his/her stroke recovery. Do you have time to answer a few estions? This will take about 5 minutes to complete. What is your name? □ No response What is your relationship? □ Spouse |
| na<br>qu<br>1. | Number of primary caregiver: () ce you are the primary caregiver, I would like to discuss the services and tasks that [patient me] needs assistance with during his/her stroke recovery. Do you have time to answer a few estions? This will take about 5 minutes to complete. What is your name? |
| na<br>qu<br>1. | Number of primary caregiver: () ce you are the primary caregiver, I would like to discuss the services and tasks that [patient me] needs assistance with during his/her stroke recovery. Do you have time to answer a few estions? This will take about 5 minutes to complete. What is your name? □ No response What is your relationship? □ Spouse |
| na<br>qu<br>1. | Number of primary caregiver: () ce you are the primary caregiver, I would like to discuss the services and tasks that [patient me] needs assistance with during his/her stroke recovery. Do you have time to answer a few estions? This will take about 5 minutes to complete. What is your name? |
| na<br>qu<br>1. | Number of primary caregiver: () ce you are the primary caregiver, I would like to discuss the services and tasks that [patient me] needs assistance with during his/her stroke recovery. Do you have time to answer a few estions? This will take about 5 minutes to complete. What is your name? |
| na<br>qu<br>1. | Number of primary caregiver: () ce you are the primary caregiver, I would like to discuss the services and tasks that [patient me] needs assistance with during his/her stroke recovery. Do you have time to answer a few estions? This will take about 5 minutes to complete. What is your name? |
| na<br>qu<br>1.<br>2. | Number of primary caregiver: () |
| 5. | Do you | provide | assistance | for [ | patient | name] | with | any | of the | following | activities? |
|---|---|---|---|---|---|---|---|---|---|---|---|
|---|---|---|---|---|---|---|---|---|---|---|---|

| 6. | Which o | of those | activities | do yo | u need | additional | assistance | with? |
|---|---|---|---|---|---|---|---|---|
|---|---|---|---|---|---|---|---|---|

| | 5. Provide assistance?<br>If Yes, go to Q6 → | | 6. Caregiver | needs he | lp with task? |
|---|---|---|---|---|---|
| | Yes | No | Yes | No | No response |
| a. Bathing / showering | | | | | |
| b. Dressing | | | | | |
| c. Getting out of bed / chair | | | | | |
| d. Helping to / from bathroom | | | | | |
| e. Feeding | | | | | |
| f. Preparing Meals | | | | | |
| g. Shopping | | | | | |
| h. Laundry | | | | | |
| i. Handling finances | | | | | |
| j. Assistance with housework | | | | | |
| k. Transportation to medical appointments | | | | | |
| Transportation to grocery<br>store, places around town,<br>etc. | | | | | |
| None → Go to Section B | | | | | |
| No Response → Go to Section B | | | | | |

| _ | _ | _ | _ | | |
|----|---------------|----------|--------|-------|----------------|
| 7 | Do you assist | Inationt | namal | with | medications? |
| 1. | Do you assist | patient | Hallie | WILLI | illedications: |

| | □ Yes → G | o to Question | n 7a and b (skip 7c) | □ No → | Go to Question 7c | |
|---|---|---|---|---|---|---|
| 78 | a. Can you nam<br>medications? | | nedicines that [patient | t <b>name]</b> is ta | aking and why he/she | is taking these |
| | □ Yes<br>□ No<br>□ No Re | sponse | | | | |
| 71 | Do you need | assistance with | n managing the patient | 's medicatio | ns? | |
| | □ Yes | □ No | ☐ No response | | | |
| 70 | c. Does someon | e else assist w | ith managing the patie | nt's medica | tions? | |
| | □ Yes | □ No | ☐ No Response | | | |
| Stroke Caregi | ver Assessment | | | | | Page 2 of 3 |

### Appendix 19 - Post-stroke Advanced Practice Assessment

| ID Number: | <u> </u> | Form Code: PSAPADate: 31MAR2016 Version 1.0 |
|---|---|---|
| ADMINISTRATIV | E INFORMATION ( | 0a-0b are auto-populated) |
| 0a. Completion Dat | e: Month Da | Ob. Staff ID: |
| | e, on average, how | many minutes/ per day has the patient engaged in continuous physical |
| activity? □ Walking | g/moving about for | <10 min/day |
| | g/moving about for 1 | (F) |
| 10 - 10 Met 120 - 10 Met 20 Me | g/moving about for > | 40.00 (a) 1.00 (a) 1 |
| ☐ No resp | onse | |
| 2. Did you educat<br>□ Yes | e patient on importa<br>□ No | nce of physical activity? |
| ☐ Yes 3. How often does ☐ Not at a ☐ Some o ☐ Every o | □ No sthe patient smoke hall → Go to Quest days | cigarettes? |
| ☐ Yes 3. How often does ☐ Not at a | □ No sthe patient smoke hall → Go to Quest days | cigarettes? |
| ☐ Yes 3. How often does ☐ Not at a ☐ Some o ☐ Every o ☐ No resp | □ No sthe patient smoke tall → Go to Quest days lay ponse | cigarettes? tion 4 counseling to end addiction to cigarettes? |
| ☐ Yes 3. How often does ☐ Not at a ☐ Some o ☐ Every o ☐ No resp 3a. Has th | □ No sthe patient smoke tall → Go to Quest days lay ponse | cigarettes?<br>tion 4 |
| ☐ Yes 3. How often does ☐ Not at a ☐ Some o ☐ Every o ☐ No resp 3a. Has th | □ No sthe patient smoke tall → Go to Quest days lay conse e patient received conserves □ No ont exceed the recommendations. | cigarettes? tion 4 counseling to end addiction to cigarettes? |
| ☐ Yes 3. How often does ☐ Not at a ☐ Some o ☐ Every o ☐ No resp 3a. Has th ☐ | □ No sthe patient smoke tall → Go to Quest days lay conse e patient received conserves □ No ont exceed the recommendations. | cigarettes? tion 4 counseling to end addiction to cigarettes? ☐ No Response |
| ☐ Yes 3. How often does ☐ Not at a ☐ Some o ☐ Every o ☐ No resp 3a. Has th ☐ 4. Does the paties (Wine=5oz., bes ☐ Yes | □ No sthe patient smoke all → Go to Quest lays lay conse e patient received conserves □ No at exceed the recomer=12 oz.) □ No | cigarettes? tion 4 counseling to end addiction to cigarettes? □ No Response mended alcohol per day? ( 1-2 drinks/day for men, 1 drink for women) |
| ☐ Yes 3. How often does ☐ Not at a ☐ Some o ☐ Every o ☐ No resp 3a. Has th ☐ 4. Does the patier (Wine=5oz., bec ☐ Yes 5. Does the patier prescription op | □ No sthe patient smoke all → Go to Quest lays lay conse e patient received conserves □ No nt exceed the recommer=12 oz.) □ No nt engage in recreations) | cigarettes? tion 4 counseling to end addiction to cigarettes? □ No Response nmended alcohol per day? ( 1-2 drinks/day for men, 1 drink for women) □ No Response tional drug use? (marijuana, cocaine, heroin, street drugs/ non- |
| ☐ Yes 3. How often does ☐ Not at a ☐ Some of ☐ Every of ☐ No resp 3a. Has th ☐ 4. Does the paties (Wine=5oz., besome of ☐ Yes 5. Does the paties | □ No so the patient smoke all → Go to Quest alays alay conse e patient received conserves □ No at exceed the recommer=12 oz.) □ No at engage in recreations | cigarettes? tion 4 counseling to end addiction to cigarettes? □ No Response nmended alcohol per day? ( 1-2 drinks/day for men, 1 drink for women) □ No Response |
| ☐ Yes 3. How often does ☐ Not at a ☐ Some o ☐ Every o ☐ No resp 3a. Has th ☐ 4. Does the patier (Wine=5oz., ber ☐ Yes 5. Does the patier prescription op ☐ Yes | □ No sthe patient smoke all → Go to Quest lays lay conse e patient received construction of the exceed the recommer=12 oz.) □ No int engage in recreation of the exceed the recommer layer laye | cigarettes? tion 4 counseling to end addiction to cigarettes? No Response mended alcohol per day? ( 1-2 drinks/day for men, 1 drink for women) No Response ional drug use? (marijuana, cocaine, heroin, street drugs/ non- |
| ☐ Yes 3. How often does ☐ Not at a ☐ Some o ☐ Every o ☐ No resp 3a. Has th ☐ 4. Does the patier (Wine=5oz., ber ☐ Yes 5. Does the patier prescription op ☐ Yes | □ No sthe patient smoke all → Go to Quest lays lay conse e patient received construction of the exceed the recommer=12 oz.) □ No int engage in recreation of the exceed the recommer layer laye | cigarettes? tion 4 counseling to end addiction to cigarettes? □ No Response nmended alcohol per day? ( 1-2 drinks/day for men, 1 drink for women) □ No Response tional drug use? (marijuana, cocaine, heroin, street drugs/ non- |

| Systolic | |
|---|---|
| Diastolic | mm HG<br>mm HG |
| Diastolic | |
| 8. HgbA1c | Not Available |
| 9. INR | |
| 10. LDL | (mg/dL) |
| 11. Are there any sev<br>that require spee<br>□ Yes | vere communication deficits such as severe dysarthria, expressive or receptive aphasia ech therapy? |
| 12. If indicated, MOC<br>□ Not Indicat<br>□ Patient ref | |
| 13. If indicated, PHQ<br>□ Not Indicat<br>□ Patient ref | ted |
| 14. Modified Rankin | score |
| □ 1 No sig<br>□ 2 Slight | mptoms at all<br>gnificant disability despite symptoms; able to carry out all usual duties and activities<br>disability; unable to carry out all previous activities, but able to look after own affairs |
| ☐ 3 Moder<br>☐ 4 Moder | ut assistance rate disability; requiring some help, but able to walk without assistance rately severe disability; unable to walk without assistance and unable to attend to own reds without assistance |
| | re disability; bedridden, incontinent and requiring constant nursing care and attention |
| 15. If the nationt noo | eds a caregiver, does the patient have a willing and able caregiver? (provider opinion) |
| | □ No □ Patient does not need a caregiver |
| □ Yes | |
| ⊔ Yes | END OF POST STROKE AP ASSESSMENT |
| ⊔ Yes | END OF POST STROKE AP ASSESSMENT |
| ⊔ Yes | END OF POST STROKE AP ASSESSMENT |
| ⊔ Yes | END OF POST STROKE AP ASSESSMENT |
| ⊔ Yes | END OF POST STROKE AP ASSESSMENT |

### Appendix 20 - Individualized Patient Care Plan (eCare Plan)

### COMPASS: Finding My Way to Recovery, Independence, and Health My Goals for My Recovery, Independence, and Health are:

| COMPASS COMPREHENSIVE POST ACUTE STROKE SERVICES | What are my concerns? | Why is this important to me? | How do I find my way forward? |
|---|---|---|---|
| | My Blood Pressure<br>is VALUE | High blood pressure<br>damages the arteries<br>that bring blood to the<br>brain. This can cause<br>another stroke. A<br>blood pressure less<br>than 120/80 is<br>considered normal. | Healthy numbers lead to a healthy life.<br>Keeping track of my numbers will decrease my chances of having another stroke. |
| NUMBERS | My hemoglobin A1c<br>level is VALUE | Keeping track of my<br>blood sugar levels can<br>reduce my risk of<br>another stroke. My<br>ideal A1c level is 6-7. | |
| Numbers:<br>Know My Numbers. Know<br>my Risks. | My LDL(bad)<br>cholesterol level is<br>VALUE | A high LDL (bad)<br>cholesterol level puts<br>me at risk for another<br>stroke. My bad<br>cholesterol level<br>should be less than 70. | |
| | My INR is VALUE,<br>This means my<br>blood is (thinner or<br>thicker) than<br>desired. | If I am on warfarin<br>(Coumadin), frequent<br>monitoring is<br>important. The right<br>level is between 2.0 –<br>3.0, unless my health<br>care provider states it<br>should be higher. | |

| I do not know all of<br>the risk factors for<br>stroke. | There are risk factors I didn't realize could cause another stroke. It's important that I am aware of these risk factors, and my own specific risk factors, so I can make correct lifestyle choices to prevent or manage them. | There are many factors that can put me at a higher risk of having another stroke. These risk factors are: • High blood pressure • Smoking • Diabetes or high blood sugar • Irregular heartbeat or atrial fibrillation • Heart disease • High cholesterol • Physical Inactivity My specific risk factors are: |
|---|---|---|

| | Engage to M | | ess and Mood |
|---|---|---|---|
| | I have been<br>experiencing stress<br>that keeps my mind<br>troubled. | Stress can increase my<br>blood pressure. Stress<br>can lead to another<br>stroke. | I can reduce my stress by: Being physically active and having a daily exercise routine Getting individual or group counseling Attending a stroke support group. |
| | Since my stroke, my<br>relationship with<br>my family has<br>become more<br>difficult or stressed. | Strained relationships<br>with my family can<br>cause me to be more<br>stressed. More stress<br>can slow down my<br>recovery. | I can get help for my family and me to make our relationships better by: Going to a stroke or brain injury support group Using the services of Care Net |
| E ENGAGE | I feel hopeless and<br>sad, and have lost<br>interest in doing my<br>favorite things. | Sadness that does not<br>go away may be due to<br>depression.<br>Depression can slow<br>down my stroke<br>recovery. | Can feel better and less sad by: Being physically active and having a daily exercise routine Getting individual or group counseling Attending a stroke support group. Getting support from my church or other community groups Taking medicine for my mood |
| 4 | Engage to Promote Physical Activity & Safe Mobility | | |
| Engage:<br>Be engaged to manage<br>my recovery,<br>independence, and health | It is difficult to use<br>my hand affected by<br>my stroke | | I can improve the use of my hand and arm by: Working with a physical and/or occupational therapist in my home or an outpatient clinic. Exercising regularly on my own or in an exercise class. Being physically active in my daily life and trying to use my arm and hand as much as possible. |
| | My muscles feel stiff<br>and I am having<br>trouble moving,<br>walking, or using my<br>hand and arm. | Medicines, therapy, exercise, and physical activity can decrease the stiffness (also called spasticity) in my muscles. This will help me be more independent and safe in my daily activities. | Can decrease the stiffness in my muscles by: Working with a physical and/or occupational therapist in my home or an outpatient clinic. Doing stretching and strengthening exercises. Taking medicines to relax my muscles. Seeing a specialist in spasticity treatment. |
| | I have fallen or I am<br>at risk for falling | I am more likely to fall<br>since I had a stroke.<br>Improving my balance<br>and strength will help<br>decrease my chances<br>of falling and improve<br>my overall<br>independence. | I can decrease my chances of falling by: • Working with a physical therapist in my home or an outpatient clinic. • Attending a falls prevention class • Using appropriate walking aids for support • Having a home safety assessment. |

| active less than 10 minutes per day (or 10-20 minutes per day). | Movement matters for my stroke recovery. I my stroke recovery. I my stroke my risk for another stroke, ncrease my endurance, and feel petter if I am obysically active. | I can be more active by Working with a physical and/or occupational therapist in my home or an outpatient clinic. Exercising regularly on my own or in an exercise class. Walking every day for at least 20 minutes a day. I can break this up into smaller chunks 10 minutes at a time. Movement around the house can keep me physically active as well (e.g doing laundry, gardening, putting up groceries). |
|---|---|---|
| walking, being able to go up/down steps, or getting out of a chair. | Regaining safe mobility will prevent me from falling. If I have strength and halance, I will be safer and more ndependent. This will mprove my stroke ecovery. | Can work on my strength and balance With a home based program that encourages me to challenge my strength and balance during my usual daily activities. A physical therapist can help design the most appropriate exercises and activities for me to do. I can join a community exercise program or exercise is medicine program affiliated with my hospital |
| Engage for m | y Recovery t | o Independence |
| independent in some of my routine activities like dressing or bathing myself, or being able to control my | Being as independent is possible will increase my confidence in my recovery. This will make it easier for my oved ones to care for me. | can become more independent in my routine activities by: Working with a physical and/or occupational therapist in my home or an outpatient clinic. Working with a home health aide on bathing and dressing Getting adaptive equipment (e.g., tub chair) that can help with my activities |
| own meals, do housework, drive myself, or use the | Eating healthy meals<br>and taking care of my<br>nome is important for<br>ny recovery and<br>overall health. | I can get healthy meals from: Meals on Wheels Congregate meals I can get help with housework and meal preparation from: Senior Services aide services CAP worker referrals (as appropriate), Community resources for respite care Home health aide services I can improve my ability to prepare meals and do housework by: Working with an Occupational therapist in my home or an outpatient clinic. I can identify family members or community agencies that will help me with transportation. |
| Engage to Ma | nage my Coi | nmunication Recovery |
| I am having trouble speaking and communicating sclearly. | Therapy services can<br>help me with my<br>swallowing and<br>speaking and with my<br>thinking" tasks so I<br>can be more<br>ndependent. | I can improve my speaking, swallowing, and thinking by: Working with a speech therapist in my home or an outpatient clinic Working with an occupational therapist in my home or an outpatient clinic Attending a support group for stroke survivors who have trouble speaking or understanding language (sometimes called aphasia). |

| Engage wit | h my Health C | are Team |
|---|---|---|
| I need a regular<br>doctor (primary<br>care provider) who<br>knows my medical<br>history and<br>conditions | A primary doctor will<br>help me monitor my<br>cholesterol, blood<br>pressure, blood sugar<br>and blood thinning. | I can find a regular doctor by: Using the information given to me in the stroke clinic Using the information on free clinics if I do not have insurance. |
| I haven't seen my<br>regular doctor<br>(primary care<br>provider) in 3<br>months or since I<br>had my stroke, or I<br>have missed<br>scheduled<br>appointments. | Seeing my doctor<br>regularly will allow for<br>better management of<br>my blood pressure,<br>blood sugar,<br>cholesterol, and other<br>stroke risk factors. | Keep a calendar reminder for my appointments Ask for help with transportation to my doctor If you are not happy with your doctor there may be other doctors you connect with better |
| I am not receiving<br>home health or<br>outpatient therapy<br>services, but I may<br>benefit from this. | Skilled therapists can<br>help me improve my<br>strength, balance and<br>ability to safely care<br>for myself and be<br>more independent. | I can ask my doctor or health care provider to make the referrals for home health or outpatient therapy services. $ . $ |

| | Since my stroke, I do<br>not eat at least two<br>meals a day. | Eating enough healthy food is important for me to recover and can help reduce my chances of having another stroke. | I can get healthy meals from Meals on Wheels or at a congregate meal site. If I cannot afford food, a social worker can help. |
|---|---|---|---|
| | I am having trouble with transportation. | Being able to get to my<br>medical appointments<br>and social events is<br>important for my<br>recovery, health and<br>happiness. | I can get help with transportation by: Being referred to Transportation services Getting support from Faith Health for my medical and non-medical appointments. |
| | My caregiver needs additional assistance with helping me with my transportation needs. | Being able to get to my<br>medical appointments<br>and social events is<br>important for my<br>recovery, health and<br>happiness. | I can get help with transportation by: Being referred to Transportation services Getting support from Faith Health for my medical and non-medical appointments. |
| $\Leftrightarrow$ | My network of<br>family and friends<br>do not (or cannot)<br>visit me as often as I<br>would like. | Being around others<br>who understand what<br>I am going through can<br>help me stay positive<br>about my recovery. | I can get support from others who care about me at stroke support groups and/or day programs as well as from members of my faith community. |
| Support: Be Aware of my | I do not have<br>someone to help me<br>bathe/dress if I ever<br>get to the point<br>where I need<br>assistance | It is important that I have a someone to assist me to live at home. | I can get support and assistance from a personal care assistant |
| Community Support | My caregiver needs additional assistance with helping me bathe, go to the toilet, dress, etc. My caregiver also needs assistance with preparing my meals and handling my finances, etc. | My caregiver and I<br>need help with what I<br>have to do every day<br>to take care of myself<br>and get better. | My caregiver and I can get help with taking care of me by letting my health care provider know what we need and asking them to refer us to resources like: A rea Agency for Aging Caregiver specialist Home Health Occupational Therapy or Physical therapy Outpatient Occupational Therapy or Physical therapy PACE Personal Care Assistant Meals on Wheels Caregiver section of COMPASS website (American Heart Association resources and Care Living Guide) |
| | Since I had my<br>stroke, my caregiver<br>has been stressed. | If my caregiver is<br>under a lot of stress it<br>causes me stress,<br>which is not good for<br>my health and<br>recovery. | My caregiver and I can get help with dealing with our stress by telling our health care provider about it and asking them to refer us to resources for stress management like: • Area Agency for Aging Powerful Tools for Caregivers • Area Agency for Aging Caregiver Specialist • American Stroke Association - Stroke Warm 1-888-4-STROKE (1-888-478-7653) • Caregiver support groups • Faith-based organizations |

| | | Refer to caregiver section of COMPASS website (American Heart Association resources and CareLiving Guide) CareNet Respite Care Stroke support groups and/or day programs |
|---|---|---|
| My caregiver would like additional assistance with helping me take my medicines. | It is important for me to take my medicines as my health care provider directs me to so that I can recover from my stroke and not have another stroke. | My health care provider can get my caregiver and me help with my medicines by referring me to: Home Health Nursing for medication management Pharmacy referral for medication management assistance to help us understand my medicines and fill my pill box. |
| My caregiver needs<br>information about<br>stroke and<br>secondary<br>prevention. | It is important for my<br>caregiver to know the<br>signs and symptoms of<br>another stroke so that<br>they can get me help<br>fast if they see<br>something that<br>concerns them. | My health care provider can give my caregiver information about stroke signs and symptoms. We can also get information in: the Caregiver Section of the COMPASS Study website AHA/ASA website's CareLiving Guide http://www.heart.org/HEARTORG/Caregiver/Resources/OtherResources/OtherResources-for-Caregivers_UCM_301861_Article.jsp# |

| | I am taking a lot of<br>medicines<br>I am not sure I know<br>my medicines. | Taking multiple medicines after a stroke may be normal. Many of these medicines help to decrease your chance of having another stroke. You should review your medicines with your provider to make sure that all your medicines are still necessary to keep you healthy. | I can share my concerns about my medicines and can get help with how to take them by reviewing them with: • My doctor • My Home Health Nurse • My local Pharmacist I may need someone everyday to help manage my medicines, fill my pillbox, or remind me so I can take them right. |
|---|---|---|---|
| WILLINGNESS | Sometimes, I forget<br>to take my<br>medicines and/or I<br>quit taking my<br>medicines when I<br>begin to feel better<br>or worse | Most medicines prescribed after stroke must be taken for a long time to prevent another stroke. Stopping them or missing doses may increase my risk of another stroke. | |
| Willingness:<br>I am willing to Manage My<br>Medication and Lifestyle<br>Choices | I do not have<br>anyone to help me<br>manage my<br>medicines, and I<br>may be getting<br>confused about<br>when to take them. | Medicines help to<br>decrease the chance of<br>having another stroke.<br>They are also useful to<br>keeping you healthy.<br>Taking my medicines<br>as directed will give<br>me the best chance for<br>preventing stroke. | |
| | | Skipping doses or<br>stopping my<br>medicines may<br>increase my risk of<br>another stroke. | |
| | I have not been able<br>to purchase some of<br>my medicines for<br>financial reasons. | Most medicines following stroke need to be filled and started when I get home from the hospital. There may be other medicines for prevention that cost less. | My health care provider or my local pharmacist can help me find cheaper medicines. Other resources include: • Medication Management Assistance • Financial Resources |

| management: -Current use of cigarettes dischol (more than 2/day for men and more than 1/day for women), and the use of recreational drugs are habits that can increase my risk of another stroke. Should I get treatment for addiction? Should I get iffestyle. We overall well-being will be improved. | My concerns with lifestyle | Cigarette smoking,<br>drinking too much | I can get help with my habits through: • North Carolina Quit Line -1-800-QUIT-NOW (1-800-784-8669). |
|---|---|---|---|
| cigarettes -Current use of alcohol -Current use of recreational drugs are habits that can increase my risk of another stroke. Should I get treatment for addiction? addiction? Should I get treatment for treatment for paddiction will promote a happy and healthier lifestyle. My overall well-being will be | management:<br>-Current use of | alcohol (more than<br>2/day for men and | Behavioral Counseling |
| -Current use of recreational drugs are habits that can increase my risk of another stroke. Should I get treatment for addiction? addiction will promote a happy and healthier lifestyle. My overall well-being will be | -Current use of | women), and the use | |
| Should I get Getting counseling and treatment for radiction? addiction will promote a happy and healthier lifestyle. My overall well-being will be | -Current use of | are habits that can<br>increase my risk of | |
| addiction? addiction will promote a happy and healthier lifestyle. My overall well-being will be | Should I get | Getting counseling and | |
| lifestyle. My overall well-being will be improved. | addiction? | addiction will promote<br>a happy and healthier | |
| improved. | | lifestyle. My overall<br>well-being will be | |

#### My recovery and my health require that:

I manage my blood pressure Numbers: I am physically active Engage: Support: I ask for help when I need it I take my medicines correctly Willingness:

Living Will

Living wills (also called advance directives) can help make sure I get the kind of care I would want if I became too sick to make my own treatment choices Are you interested in making a living will?

treatment choices.

Begin a Conversation With Your Family and Doctor:

- Beginning the conversation with your family and health care providers.  $\underline{\text{http://www.begintheconversation.org/}}$
- Ask your primary care doctor to discuss your preferences for a living will.

  Contact agencies in your community

  to fully understand advanced directives and select your options (community agencies include the Community Care of North Carolina, palliative and hospice programs)

For additional information, and to investigate local resources, visit the COMPASS study website at: https://www.nccompass-study.org

#### Appendix 21 - Consent and HIPAA Authorization for Clinical Data



Do you have any questions?

### COMPASS STUDY Informed Consent and HIPAA Authorization

Your hospital is participating in a statewide study called the Comprehensive Post-Acute Stroke Services (COMPASS) Study. The purpose of the COMPASS Study is to determine the best ways to care for stroke survivors after they go home.

The PI for the COMPASS Study is Dr. Pamela Duncan at Wake Forest Baptist Medical Center (WFBMC). This study is funded by the Patient-Centered Outcome Research Institute (PCORI).

We would like to ask you for your consent and HIPAA authorization to keep a record of your personal health information and responses to the questions we asked you during the COMPASS telephone calls and this visit. This includes information from your recent hospitalization, visits to your doctor, and medications. We would like keep your responses to learn more about how we can improve the delivery of care to patients who have had a stroke. This information will be kept completely confidential and it will be kept in a secure place.

Your consent is completely voluntary. If you choose not to provide consent, you will still receive the same quality treatment and follow up. This medical facility may not condition (withhold or refuse) treating you on whether you sign this Authorization.

You may change your mind and withdraw your consent later. However, if you withdraw your consent, the organization may still use information that was previously collected about you. WFBMC and some study team members may financially benefit from the creation of an electronic tool that is being used in this study. The health information listed above may be used by and/or disclosed to the study investigators at this site and others, study management centers, the study sponsor, and other groups, including federal agencies, which have a responsibility to assist in the oversight and management of the research study. This Authorization does not have an expiration date.

If you have any questions or if you would like to withdraw your consent, you can call us toll-free at 1-844-501-7668 or if it easier, you can email us at: <a href="mailto:thecompassstudy@gmail.com">thecompassstudy@gmail.com</a>.

By signing below, you give permission to disclose your identifiable health information for the COMPASS research study. Would you like to give us permission to keep your data for research purposes?

Subject Name (Printed):

Subject Signature:

Date:

Time:

am pm

Person Obtaining Consent (Printed):

Date:

Time:

am pm

# Wake Forest\* School of Medicine

| capacity: | | | |
|---|---|---|---|
| Legally Authorized Representative Name (Print):_ | | | |
| The above named Legally Authorized Represent subject based upon (specify health care power of the control of th | ntative has legal author<br>of attorney, spouse, par | rity to act for the<br>rent, etc.) | e research |
| Relationship to the Subject: | | | |
| Legal Representative Signature: | Date: | Time: | am pm |

### Appendix 22 - 30 and 60 Day Call Forms (60 Day Call Form is Identical)

| D Number: Form Code: | D Y 3 0 Date: 06JUN2016 Version 1.0 |
|---|---|
| ADMINISTRATIVE INFORMATION (0a-0c are a a. Completion Date: | auto-populated) / Ob. Staff ID: |
| Instructions for the PAC: Please summarize during the 30-day follow-up call by answering | the outcome of your conversation with the patient<br>g the questions below. |
| 1. Does patient know what his/her target BP sh | ould be? □ Yes □ No |
| 2. Is patient monitoring their BP? ☐ Yes ☐ | No |
| a. If Yes, how many times per week on | average? |
| 3. Did the patient know their last blood pressure | |
| Has the patient received any <u>nome health</u> rel a. If Yes, indicate which types (check al | habilitation services since discharge? Yes No |
| □ Physical therapy | титат арргу) |
| ☐ Occupational therapy | |
| ☐ Speech therapy | |
| b. If No, what are the reason(s) for no h | ome health rehab services? (check all that apply) |
| ☐ Patient did not need therapy | ☐ No transportation |
| ☐ Financial / insurance | ☐ Patient did not think necessary / refused |
| ☐ No reason given | □ Other |
| Has the patient received any <u>outpatient</u> rehal | bilitation services since discharge? ☐ Yes ☐ No |
| a. If Yes, indicate which types (check al | I that apply) |
| ☐ Physical therapy | |
| ☐ Occupational therapy | |

| □ Patient did not need therapy | ☐ No transportation |
|---|---|
| ☐ Financial / insurance | ☐ Patient did not think necessary / refused |
| ☐ No reason given | □ Other |
| 6. Did the patient receive the support they need | ded from community services during this intervention? |
| □ No, none of the support needed | i e |
| ☐ Some of the support needed | |
| ☐ Most of the support needed | |
| ☐ All the support needed | |
| To be answered by PAC for administrative pu | ırposes: |
| 7. Did you complete the 30-day telephone call | including the telephone script? |
| ☐ Yes ☐ No → Go to Question | 1 7a |
| 7a. If no, why not | |
| ☐ Patient refused | |
| ☐ Unable to reach after 3 calls | |
| ☐ Partially complete / did not finis | h call |
| □ Other | |
| 8. Did you speak with the patient or a proxy? | □ Patient □ Proxy |
| END OF 30-DA | Y PAC CALL DATA FORM |

### **Appendix 23 - 90d Patient Survey (CATI/ Phone Format)**

### **COMPASS 90 Day Patient Survey**

| LABEL | VALUE | TEXT | INSTRUCTIONS |
|---|---|---|---|
| INTRO | 0=R DOES NOT HAVE Q'NAIRE FOR REFERENCE 1=R DOES HAVE Q'NAIRE FOR REFERENCE 8=DON'T KNOW | I'm going to be asking you a series of questions about [IF NO PROXY: your] [IF PROXY=1 OR 2: FILL R NAME]'s health and activities since NO PROXY: you were PROXY: he/she was hospitalized for stroke or TIA. Most of the questions are on the questionnaire we mailed [NO PROXY: to you] about a week ago. Do you have that in front of you or would you like to go get it? IN: GIVE THE R TIME TO GO GET IT, BUT IF THEY DON'T HAVE OR CAN'T FIND PAPER Q'NAIRE: That's OK, we can complete the call without it. IF NEEDED: TIA stands for transient ischemic attack and is sometimes referred to as a mini-stroke or warning stroke. | |
| SIS_INTRO | EMPTY | I'd like to start by asking you about the physical problems NO PROXY: you PROXY: he/she may have because of your/his/her stroke (or TIA). I want to know NO PROXY: [from YOUR POINT OF VIEW] how stroke has affected your/his/her physical | |

| , | |
|-------------|---------------|
| Application | - IRB00035998 |

| Application - IKB00033998 | | |
|---|---|---|
| | | function in the past two |
| | | weeks. |
| | | I'm going to read a list of tasks and for each one, I'd like you to tell me whether it is not difficult at all, a little difficult, somewhat difficult, very difficult or if the task can't be done at all. IF NEEDED: I'm required to ask all the questions, but |
| | | please just answer to the |
| | | best of your ability. |
| CICA | | |
| SIS1 | 1=Not difficult at all | In the past two weeks how |
| | 2=A little difficult | difficult was it PROXY: for |
| | 3=Somewhat difficult | him/her to dress the top |
| | 4=Very difficult | part of your/his/her body? |
| | 5=Or you could not do this | Would you say |
| | activity at all? | |
| | 8=DON'T KNOW | |
| SIS2 | 9=REFUSE<br>1 =Not difficult at all | In the past two weeks, how |
| 3132 | 2=A little difficult | difficult was it [for |
| | 3=Somewhat difficult | him/her]to bathe |
| | 4=Very difficult | yourself/himself/herself? |
| | 5=Or you could not do this | Would you say |
| | activity at all? | |
| | 8=DON'T KNOW | INTERVIEWER NOTE: |
| | 9=REFUSE | Bathing oneself does not |
| | | include getting into the tub. |
| SIS3 | 1 =Not difficult at all | In the past two weeks, how |
| | 2=A little difficult | difficult has it been [for |
| | 3=Somewhat difficult | him/her] to get to the toilet |
| | 4=Very difficult | on time? |
| | 5=Or you could not do this | |
| | activity at all? | (Would you say) |
| | 8=DON'T KNOW | |
| | 9=REFUSE | INTERVIEWER NOTE: For |
| | | this question we are |
| | | interested in how quickly |

| Application - IRB000359 | 798 | - the felt and the the |
|---|---|---|
| | | you/he/she can get to the |
| | | bathroom. |
| SIS4 | 1=NOT (DIFFICULT) AT ALL | In the past two weeks how |
| | 2=A LITTLE (DIFFICULT) | difficult has it been [for |
| | 3=SOMEWHAT (DIFFICULT) | him/her] to control |
| | 4=VERY (DIFFICULT) | your/his/her bladder, that |
| | 5=OR YOU COULD NOT DO | is, not have an accident? |
| | THIS ACTIVITY AT ALL? | |
| | 8=DON'T KNOW | (Would you say) |
| | 9=REFUSE | |
| | | IN: OKAY TO DROP |
| | | "DIFFICULT" WHEN |
| | | READING RESPONSE |
| | | OPTIONS |
| | | IN NOTE: LOSING A |
| | | LITTLE |
| | | URINE/DRIBBLING IS |
| | | CONSIDERED AN |
| | | ACCIDENT. IF PERSON |
| | | HAS INTERMITTENT |
| | | CATHETER AND IS |
| | | HAVING NO LEAKING |
| | | PROBLEMS CODE THEM |
| | | AS PER REPORT. IF |
| | | PERSON HAS AN IN- |
| | | DWELLING FOLEY |
| | | CATHETER, CODE AS |
| | | CANNOT DO AT ALL. |
| SIS5 | 1=NOT (DIFFICULT) AT ALL | In the past two weeks how |
| | 2=A LITTLE (DIFFICULT) | difficult has it been [for |
| | 3=SOMEWHAT (DIFFICULT) | him/her] to control |
| | 4=VERY (DIFFICULT) | your/his/her bowels, that |
| | 5=OR YOU COULD NOT DO | is, not have an accident? |
| | THIS ACTIVITY AT ALL? | |
| | 8=DON'T KNOW | (Would you say) |
| | 9=REFUSE | |
| | | IN NOTE: CONSTIPATION |
| | | IS NOT COUNTED HERE. |
| | | THE PERSON HAS TO |
| | | HAVE AN ACCIDENT. |
| SIS6 | 1=NOT (DIFFICULT) AT ALL | (In the past two weeks, how |
| | 2=A LITTLE (DIFFICULT) | difficult has it been [for |
| | 3=SOMEWHAT (DIFFICULT) | him/her] to) Stand without |
| | 4=VERY (DIFFICULT) | losing balance? |
| | , , , | |
| | | 1 |

| Application - IRB00035998 | | |
|---|---|---|
| | 5=OR YOU COULD NOT DO<br>THIS ACTIVITY AT ALL?<br>8=DON'T KNOW<br>9=REFUSE | (Would you say) |
| SIS7 | 1=NOT (DIFFICULT) AT ALL 2=A LITTLE (DIFFICULT) 3=SOMEWHAT (DIFFICULT) 4=VERY (DIFFICULT) | (In the past two weeks, how difficult has it been [for him/her] to) Go shopping? |
| | 5=OR YOU COULD NOT DO THIS ACTIVITY AT ALL? | (Would you say) |
| | 8=DON'T KNOW<br>9=REFUSE | IN NOTE: THIS CAN BE SHOPPING ALONE OR WITH SOMEONE. |
| SIS8 | 1=NOT (DIFFICULT) AT ALL 2=A LITTLE (DIFFICULT) 3=SOMEWHAT (DIFFICULT) 4=VERY (DIFFICULT) 5=OR YOU COULD NOT DO THIS ACTIVITY AT ALL? 8=DON'T KNOW | (In the past two weeks, how difficult has it been [for him/her] to) Do heavy household chores, for example, vacuum, laundry or yard work? |
| | 9=REFUSE | (Would you say) |
| SIS9 | 1=NOT (DIFFICULT) AT ALL 2=A LITTLE (DIFFICULT) 3=SOMEWHAT (DIFFICULT) 4=VERY (DIFFICULT) 5=OR YOU COULD NOT DO THIS ACTIVITY AT ALL? | (In the past two weeks, how difficult has it been[for him/her] to) Stay sitting without losing your/his/her balance? |
| | 8=DON'T KNOW<br>9=REFUSE | (Would you say) |
| SIS10 | 1=NOT (DIFFICULT) AT ALL 2=A LITTLE (DIFFICULT) 3=SOMEWHAT (DIFFICULT) 4=VERY (DIFFICULT) 5=OR YOU COULD NOT DO THIS ACTIVITY AT ALL? | (In the past two weeks, how difficult has it been [for him/her] to) Walk without losing your/his/her balance? |
| | 8=DON'T KNOW<br>9=REFUSE | (Would you say) |
| | | IN NOTE: THE DISTANCE IS NOT IMPORTANT |
| SIS11 | 1=NOT (DIFFICULT) AT ALL 2=A LITTLE (DIFFICULT) 3=SOMEWHAT (DIFFICULT) 4=VERY (DIFFICULT) 5=OR YOU COULD NOT DO | (In the past two weeks, how difficult has it been [for him/her] to) Move from a bed to a chair? |
| | THIS ACTIVITY AT ALL? | (Would you say) |

| Application - IRB00035998 | O DON'T WHO'' | T |
|---|---|---|
| | 8=DON'T KNOW | |
| 0.040 | 9=REFUSE | |
| SIS12 | 1=NOT (DIFFICULT) AT ALL | (In the past two weeks, how |
| | 2=A LITTLE (DIFFICULT) | difficult has it been [for |
| | 3=SOMEWHAT (DIFFICULT) | him/her] to) Walk fast? |
| | 4=VERY (DIFFICULT) | |
| | 5=OR YOU COULD NOT DO | (Would you say) |
| | THIS ACTIVITY AT ALL? | |
| | 8=DON'T KNOW | |
| | 9=REFUSE | |
| SIS13 | 1=NOT (DIFFICULT) AT ALL | (In the past two weeks, how |
| | 2=A LITTLE (DIFFICULT) | difficult has it been[for |
| | 3=SOMEWHAT (DIFFICULT) | him/her] to) Climb one |
| | 4=VERY (DIFFICULT) | flight of stairs? |
| | 5=OR YOU COULD NOT DO | |
| | THIS ACTIVITY AT ALL? | (Would you say) |
| | 8=DON'T KNOW | |
| | 9=REFUSE | |
| SIS14 | 1=NOT (DIFFICULT) AT ALL | (In the past two weeks, how |
| | 2=A LITTLE (DIFFICULT) | difficult has it been[for |
| | 3=SOMEWHAT (DIFFICULT) | him/her] to ) Walk one |
| | 4=VERY (DIFFICULT) | block? |
| | 5=OR YOU COULD NOT DO | |
| | THIS ACTIVITY AT ALL? | (Would you say) |
| | 8=DON'T KNOW | |
| | 9=REFUSE | IN NOTE: THIS COULD |
| | | INVOLVE WALKING WITH |
| | | SUPPORT, SUCH AS WITH A |
| | | CANE OR A WALKER. |
| SIS15 | 1=NOT (DIFFICULT) AT ALL | (In the past two weeks, how |
| | 2=A LITTLE (DIFFICULT) | difficult has it been[for |
| | 3=SOMEWHAT (DIFFICULT) | him/her] to) Get in and out |
| | 4=VERY (DIFFICULT) | of a car? |
| | 5=OR YOU COULD NOT DO | |
| | THIS ACTIVITY AT ALL? | (Would you say) |
| | 8=DON'T KNOW | |
| | 9=REFUSE | IN NOTE: IF THE |
| | | RESPONDENT WANTS |
| | | TO KNOW WHAT KIND |
| | | OF CAR SAY YOUR CAR |
| | | OR THE CAR YOU RIDE |
| | | IN THE MOST. |
| SIS16 | 1=NOT (DIFFICULT) AT ALL | (How about) Carry heavy |
| | 2=A LITTLE (DIFFICULT) | objects, for example, a bag |
| | 3=SOMEWHAT (DIFFICULT) | of groceries, with |

| Application - IRB00035998 | 1 | T | 1 |
|---|---|---|---|
| | 4=VERY (DIFFICULT) 5=OR YOU COULD NOT DO THIS ACTIVITY AT ALL? | your/his/her affected hand? | |
| | 8=DON'T KNOW | (Would you say) | |
| | 9=REFUSE | IF NEEDED: By 'affected' we mean the side of your body that was affected by your/his/her stroke. | |
| | | IN NOTE: THIS MEANS ANY PART OF THEIR BODY AFFECTED EVEN IF NOT THEIR HAND. E.G. FACE, LEG, ETC. | |
| HEALTH_INTRO | | The next two questions are about how you perceive or view your general health. | PROGRAMMING: SKIP<br>IF PROXY=1 OR 2 |
| RateHlt | 1=poor<br>2=fair<br>3=good<br>4=very good<br>5=excellent<br>8=DON'T KNOW<br>9=REFUSE | Compared to others your age, how would you rate your health since your stroke or TIA? Would you say | PROGRAMMING: SKIP IF PROXY=1 OR 2 |
| PredHlt | 1=Stay the same<br>2=Improve<br>3=Get worse<br>8=DON'T KNOW<br>9=REFUSE | Over the next 3 months, do you think your health is going to: | PROGRAMMING: SKIP<br>IF PROXY=1 OR 2 |
| MRS_INTRO | | This next set of questions is asking about the level of assistance you/he/she may or may not need with certain tasks and your/his/her ability to do things since your/his/her stroke or TIA." [IF INTRO=1, FILL]Depending on your responses I may skip some of the questions on the survey you have in front of you. | |

| Application - IKBOO | 033996 | 1 | T |
|---|---|---|---|
| | | IF NEEDED: TIA stands<br>for transient ischemic attack<br>and is sometimes referred to<br>as a "mini-stroke" or<br>"warning stroke." | |
| MRS1 | 0=NO (GO TO MRS4) 1=YES (GO TO MRS2) 8=DON'T KNOW (GO TO PA _INTRO) 9=REFUSE (GO TO PA_INTRO) | Could you/he/she live alone without any help from another person? This means being able to bathe, use the toilet, shop, prepare or get meals and manage finances. IN: AVOID DK OR REFUSE. ENCOURAGE THE R TO ANSWER YES OR NO. | |
| MRS2 | 0=NO (GO TO PA_INTRO) 1=YES (GO TO MRS3) 8=DON'T KNOW (GO TO PA_INTRO) 9=REFUSE (GO TO PA_INTRO) | Can you/he/she do everything that you/he/she were/was doing right before your/his/her stroke, even if slower and not as much? | |
| MRS3 | 0=NO (GO TO PA_INTRO) 1=YES (GO TO PA_INTRO) 8=DON'T KNOW (GO TO PA_INTRO) 9=REFUSE (GO TO PA_INTRO) | Are/Is you/he/she completely back to the way you/he/she were/was right before your/his/her stroke? | |
| MRS4 | 0=NO (GO TO MRS5) 1=YES (GO TO PA_INTRO) 8=DON'T KNOW (GO TO PA_INTRO) 9=REFUSE (GO TOPA_INTRO) | Can you/he/she walk from one room to another without help from another person? IN NOTE: WALKING FROM ONE ROOM TO ANOTHER WITHOUT THE HELP OF ANOTHER PERSON – INCLUDES WALKING WITH A CANE OR WALKER AS LONG AS THE PERSON DOES IT INDEPENDENTLY. | |

| Application - IRB00035998 | | <u>, </u> |
|---|---|---|
| MRS5 | 0=NO (GO TO PA_INTRO)<br>1=YES (GO TO PA_INTRO) | Can you/he/she sit up in bed without any help? |
| | | , |
| | 8=DON'T KNOW (GO TO | |
| | PA_INTRO) | |
| | 9=REFUSE (GO TO<br>PA INTRO) | |
| PA_INTRO | IA_INTROJ | The next few questions are |
| _ | | about the amount of time |
| | | you/he/she have/has spent |
| | | walking in the last 7 days. |
| PAday_YN | 0=NO (GO TO MOOD | In the past 7 days did |
| | INTRO)<br>1=YES (GO TO PADAY) | you/he/she walk continuously for at least 10 |
| | 1-123 (00 10 1 ADA1) | minutes on any day? |
| | 8=DON'T KNOW (GO TO | , |
| | MOOD INTRO) | |
| | 9=REFUSE (GO TO MOOD | |
| DAday | INTRO) | During the last 7 days are |
| PAday | ENTER A NUMBER FROM 0-7 | During the last 7 days <u>on</u><br>how many days did |
| | IF >0, THEN GO TO PAMIN | you/he/she walk |
| | IF 0 GO TO MOOD_INTRO | continuously, for at least 10 |
| | 8=DON'T KNOW (GO TO | minutes, for recreation, |
| | MOOD_INTRO) | exercise, or to get to or |
| | 9=REFUSE (GO TO MOOD | from places? |
| | INTRO) | IN: IF R RESPONDS 'DON'T KNOW', PROBE WHETHER |
| | | DON'T KNOW # OF DAYS (IF |
| | | THIS, ENCOURAGE BEST |
| | | GUESS) OR DON'T KNOW IF |
| | | 10 MINUTES |
| | | CONTINUOUSLY (IF THIS, |
| | | GO BACK TO PADAY_YN<br>AND CHOOSE DON'T |
| | | KNOW) |
| | | , |
| | | IF NEEDED: Think only |
| | | about the walking that |
| | | you/he/she do/does for at |
| | | least 10 minutes at a time. |
| PAmin | | On days when you/he/she |
| | | walked for at least 10 |
| | | minutes, how much total |

| Application - IRB00035998 | | T | |
|---|---|---|---|
| | Enter a numeric value between 10 and 840 (GO | time per day, did you/he/she spend walking? | |
| | TO MOOD INTRO) | | |
| | | IN: We're looking for an | |
| | 8=DON'T KNOW (GO TO | average time per day that | |
| | PAWALK) | you/he/she walked. | |
| | 9=REFUSE (GO TO PAWALK) | | |
| DA . II | | | |
| PAwalk | Enter a number of minutes | What is the total amount of time you/he/she spent | |
| | 8=DON'T KNOW | walking over the last 7 | |
| | 9=REFUSE | days? | |
| MOOD_INTRO | 9-KLI 03L | The next two questions are | PROGRAMMING: SKIP |
| WOOD_INTINO | | about your mood. I now | IF PROXY=1 OR 2 |
| | | want you to think about the | IF PROXI-1 OR 2 |
| | | 1 | |
| | | past <u>two weeks</u> , how often have you been bothered by | |
| | | · | |
| | | any of the following | |
| | | problems? | |
| | | IN: STRESS 2 WEEKS SINCE | |
| | | RESPONDENT JUST | |
| | | FOCUSED ON PAST WEEK. | |
| Mood1 | 1=Not at all | Little interest or pleasure in | PROGRAMMING: SKIP |
| | 2=Several days | doing things? | IF PROXY=1 OR 2 |
| | 3=More than half of the | Would you say you've been | |
| | days | bothered | |
| | 4=Nearly every day | | |
| | 8=DON'T KNOW | | |
| | 9=REFUSE | | |
| Mood2 | 1=Not at all | How about feeling down, | PROGRAMMING: SKIP |
| | 2=Several days | depressed, or hopeless? | IF PROXY=1 OR 2 |
| | 3=More than half of the | Would you say you've been | |
| | days | bothered | |
| | 4=Nearly every day | | |
| | 8=DON'T KNOW | | |
| | 9=REFUSE | | |
| | EMPTY | The next set of questions | PROGRAMMING: SKIP |
| | | are not on the paper | IF PROXY=1 OR 2 |
| | | survey. This is a memory | |
| | | assessment. I am going to | |
| | | read a list of words that you | |
| | | will have to remember now | |
| | | and later on. Please listen | |
| | ı | | 1 |

| Application - IRB00 |
|---------------------|
|---------------------|

| Application - IKB00033998 | | carefully but do not write them down. When I am through, tell me as many words as you can remember. It doesn't matter in what order you say them. Are you ready to hear the words? | |
|---|---|---|---|
| MOCA1_1 MOCA1_2 MOCA1_3 MOCA1_4 MOCA1_5 | 1=FACE<br>2=VELVET<br>3=CHURCH<br>4=DAISY<br>5=RED | IN: WHEN R IS READY, READ THE FOLLOWING OUT LOUD AT A RATE OF 1 WORD PER SECOND: Face, Velvet, Church, Daisy, Red Now, please tell me which words you remember. IN: IF R SAYS SIMILAR SOUNDING WORD, COUNT AS CORRECT AND SAY: Thank you. I will count that as the correct answer, but to clarify, the word was [REPEAT WORD], spelled [SPELL WORD]. WHEN THE SUBJECT INDICATES THAT (S)HE HAS FINISHED (HAS RECALLED ALL WORDS), OR CAN RECALL NO MORE WORDS, MOVE ON. | PROGRAMMING: SKIP IF PROXY=1 OR 2 |
| 125 | ЕМРТҮ | Thank you. I'm going to read the same list a second time. Try to remember and tell me as many words as you can, including words you said the first time. | PROGRAMMING: SKIP IF PROXY=1 OR 2 (do second trial even if 1st trial successful) |

| MOCA12_1 | 1=FACE | Aro you roady to boor the | PROGRAMMING: SKIP |
|---|---|---|---|
| MOCA12_1 | 2=VELVET | Are you ready to hear the | |
| | | words? | IF PROXY=1 OR 2 |
| | 3=CHURCH | | |
| | 4=DAISY | IN: WHEN R IS READY, READ | |
| | 5=RED | THE FOLLOWING: | |
| | 4 | Face, Velvet, Church, Daisy, | |
| MOCA12_2 | 1=FACE | Red | |
| | 2=VELVET | 1100 | |
| | 3=CHURCH | IE NEEDED: Now places tall | |
| | 4=DAISY | IF NEEDED: Now please tell | |
| | 5=RED | me which words you remember. | |
| MOCA12_3 | 1=FACE | | |
| | 2=VELVET | IN: IF R SAYS SIMILAR | |
| | 3=CHURCH | SOUNDING WORD, COUNT | |
| | 4=DAISY | AS CORRECT AND SAY: | |
| | 5=RED | Thank you. I will count that | |
| | | • | |
| MOCA12_4 | 1=FACE | as the correct answer, but | |
| _ | 2=VELVET | to clarify, the word was | |
| | 3=CHURCH | [REPEAT WORD], spelled | |
| | 4=DAISY | [SPELL WORD]. | |
| | 5=RED | | |
| MOCA12_5 | 1=FACE | CHECK EACH ONE THAT THE | |
| | 2=VELVET | R SAYS CORRECTLY THE 2 <sup>ND</sup> | |
| | 3=CHURCH | TIME. | |
| | 4=DAISY | 12 | |
| | 5=RED | WHEN THE SUBJECT | |
| | | INDICATES THAT (S)HE | |
| | | ` ' | |
| | | HAS FINISHED (HAS<br>RECALLED ALL | |
| | | WORDS), OR CAN | |
| | | RECALL NO MORE | |
| | | WORDS, MOVE ON. | |
| MOCA_THANKS | EMPTY | Thank you. I will ask you to | PROGRAMMING: SKIP |
| | | recall these words again at | IF PROXY=1 OR 2 |
| | | the end of the test. | |
| | | IN: DO NOT REPEAT THE | |
| | | WORDS OR TELL THE R | |
| | | WHICH ONES S/HE FORGOT | |
| MOCA2_01 | ANIMAL1=1 | I'd like you to name as | PROGRAMMING: SKIP |
| MOCA2_02 | ANIMAL2=2 | many animals as you can in | IF PROXY=1 OR 2 |
| MOCA2_03 | ANIMAL3=3 | , 2 | |
| MOCA2_04 | 7 | | |

| | T | 1 | |
|---|---|---|---|
| MOCA2_05 | ANIMAL4=4 | one minute. You can start | |
| MOCA2_06 | ANIMAL5=5 | now. | |
| MOCA2_07 | ANIMAL6=6 | IF NEEDED: Animal can | |
| MOCA2_08 | ANIMAL7=7 | include mammals, reptiles, | |
| MOCA2_09 | ANIMAL8=8 | fish, birds, insects, etc. | |
| MOCA2_10 | ANIMAL9=9 | Anything that moves on its | |
| MOCA2_11 | ANIMAL10=10 | own and eats. | |
| MOCA2_12 | ANIMAL11=11 | | |
| MOCA2_13 | ANIMAL12=12 | IN: DO NOT COUNT THE | |
| MOCA2_14 | ANIMAL12=12<br>ANIMAL13=13 | EXACT SAME ANIMAL | |
| MOCA2_15 | ANIMAL13=13 | TWICE; E.G. HORSE AND | |
| MOCA2_16<br>MOCA2_17 | ANIMAL14-14<br>ANIMAL15=15 | HORSE | |
| MOCA2_17 | | | |
| WOCAZ_18 | ANIMAL16=16 | <b>DO</b> COUNT VARIATIONS; | |
| | ANIMAL17=17 | E.G. BIRD AND EAGLE | |
| | ANIMAL18=18 | | |
| | | IN: CHECK THE BOX FOR | |
| | Value is missing (.) when no | EACH ANIMAL NAMED. | |
| | animal was named | STOP RESPONDENT AT ONE | |
| | | MINUTE OR WHEN 18 | |
| | | ANIMALS HAVE BEEN | |
| | | NAMED, WHICHEVER | |
| | | COMES FIRST. | |
| MOCA3_1 | 1=MONTH | COMES FIRST. Thank you. Can you tell me | PROGRAMMING: SKIP |
| MOCA3_1 | 1=MONTH<br>2=DATE | | PROGRAMMING: SKIP IF PROXY=1 OR 2 |
| MOCA3_1 | | Thank you. Can you tell me | |
| MOCA3_1 | 2=DATE | Thank you. Can you tell me | |
| | 2=DATE<br>3=YEAR<br>4=DAY OF THE WEEK | Thank you. Can you tell me today's date? IF RESPONDENT GIVES AN | |
| MOCA3_1 MOCA3_2 | 2=DATE 3=YEAR 4=DAY OF THE WEEK 1=MONTH | Thank you. Can you tell me today's date? IF RESPONDENT GIVES AN INCOMPLETE ANSWER, | |
| | 2=DATE 3=YEAR 4=DAY OF THE WEEK 1=MONTH 2=DATE | Thank you. Can you tell me today's date? IF RESPONDENT GIVES AN INCOMPLETE ANSWER, PROMPT ACCORDINGLY: | |
| | 2=DATE 3=YEAR 4=DAY OF THE WEEK 1=MONTH 2=DATE 3=YEAR | Thank you. Can you tell me today's date? IF RESPONDENT GIVES AN INCOMPLETE ANSWER, PROMPT ACCORDINGLY: Can you tell me the year, | |
| | 2=DATE 3=YEAR 4=DAY OF THE WEEK 1=MONTH 2=DATE | Thank you. Can you tell me today's date? IF RESPONDENT GIVES AN INCOMPLETE ANSWER, PROMPT ACCORDINGLY: Can you tell me the year, month, exact date, and day | |
| MOCA3_2 | 2=DATE 3=YEAR 4=DAY OF THE WEEK 1=MONTH 2=DATE 3=YEAR 4=DAY OF THE WEEK | Thank you. Can you tell me today's date? IF RESPONDENT GIVES AN INCOMPLETE ANSWER, PROMPT ACCORDINGLY: Can you tell me the year, | |
| | 2=DATE 3=YEAR 4=DAY OF THE WEEK 1=MONTH 2=DATE 3=YEAR 4=DAY OF THE WEEK 1=MONTH | Thank you. Can you tell me today's date? IF RESPONDENT GIVES AN INCOMPLETE ANSWER, PROMPT ACCORDINGLY: Can you tell me the year, month, exact date, and day of the week? | |
| MOCA3_2 | 2=DATE 3=YEAR 4=DAY OF THE WEEK 1=MONTH 2=DATE 3=YEAR 4=DAY OF THE WEEK 1=MONTH 2=DATE | Thank you. Can you tell me today's date? IF RESPONDENT GIVES AN INCOMPLETE ANSWER, PROMPT ACCORDINGLY: Can you tell me the year, month, exact date, and day of the week? IN: MARK EACH CORRECT | |
| MOCA3_2 | 2=DATE 3=YEAR 4=DAY OF THE WEEK 1=MONTH 2=DATE 3=YEAR 4=DAY OF THE WEEK 1=MONTH 2=DATE 3=YEAR | Thank you. Can you tell me today's date? IF RESPONDENT GIVES AN INCOMPLETE ANSWER, PROMPT ACCORDINGLY: Can you tell me the year, month, exact date, and day of the week? IN: MARK EACH CORRECT RESPONSE, THE DATE AND | |
| MOCA3_2 | 2=DATE 3=YEAR 4=DAY OF THE WEEK 1=MONTH 2=DATE 3=YEAR 4=DAY OF THE WEEK 1=MONTH 2=DATE | Thank you. Can you tell me today's date? IF RESPONDENT GIVES AN INCOMPLETE ANSWER, PROMPT ACCORDINGLY: Can you tell me the year, month, exact date, and day of the week? IN: MARK EACH CORRECT RESPONSE, THE DATE AND DAY OF THE WEEK CAN BE | |
| MOCA3_2 | 2=DATE 3=YEAR 4=DAY OF THE WEEK 1=MONTH 2=DATE 3=YEAR 4=DAY OF THE WEEK 1=MONTH 2=DATE 3=YEAR | Thank you. Can you tell me today's date? IF RESPONDENT GIVES AN INCOMPLETE ANSWER, PROMPT ACCORDINGLY: Can you tell me the year, month, exact date, and day of the week? IN: MARK EACH CORRECT RESPONSE, THE DATE AND DAY OF THE WEEK CAN BE OFF BY A DAY AND STILL BE | |
| MOCA3_2 MOCA3_3 | 2=DATE 3=YEAR 4=DAY OF THE WEEK 1=MONTH 2=DATE 3=YEAR 4=DAY OF THE WEEK 1=MONTH 2=DATE 3=YEAR 4=DAY OF THE WEEK | Thank you. Can you tell me today's date? IF RESPONDENT GIVES AN INCOMPLETE ANSWER, PROMPT ACCORDINGLY: Can you tell me the year, month, exact date, and day of the week? IN: MARK EACH CORRECT RESPONSE, THE DATE AND DAY OF THE WEEK CAN BE OFF BY A DAY AND STILL BE COUNTED. E.G. TODAY'S | |
| MOCA3_2 | 2=DATE 3=YEAR 4=DAY OF THE WEEK 1=MONTH 2=DATE 3=YEAR 4=DAY OF THE WEEK 1=MONTH 2=DATE 3=YEAR 4=DAY OF THE WEEK | Thank you. Can you tell me today's date? IF RESPONDENT GIVES AN INCOMPLETE ANSWER, PROMPT ACCORDINGLY: Can you tell me the year, month, exact date, and day of the week? IN: MARK EACH CORRECT RESPONSE, THE DATE AND DAY OF THE WEEK CAN BE OFF BY A DAY AND STILL BE COUNTED. E.G. TODAY'S DATE IS 5/10, SO 5/9, 5/10, | |
| MOCA3_2 MOCA3_3 | 2=DATE 3=YEAR 4=DAY OF THE WEEK 1=MONTH 2=DATE 3=YEAR 4=DAY OF THE WEEK 1=MONTH 2=DATE 3=YEAR 4=DAY OF THE WEEK 1=MONTH 2=DATE 3=YEAR 4=DAY OF THE WEEK | Thank you. Can you tell me today's date? IF RESPONDENT GIVES AN INCOMPLETE ANSWER, PROMPT ACCORDINGLY: Can you tell me the year, month, exact date, and day of the week? IN: MARK EACH CORRECT RESPONSE, THE DATE AND DAY OF THE WEEK CAN BE OFF BY A DAY AND STILL BE COUNTED. E.G. TODAY'S | |
| MOCA3_2 MOCA3_3 | 2=DATE 3=YEAR 4=DAY OF THE WEEK 1=MONTH 2=DATE 3=YEAR 4=DAY OF THE WEEK 1=MONTH 2=DATE 3=YEAR 4=DAY OF THE WEEK | Thank you. Can you tell me today's date? IF RESPONDENT GIVES AN INCOMPLETE ANSWER, PROMPT ACCORDINGLY: Can you tell me the year, month, exact date, and day of the week? IN: MARK EACH CORRECT RESPONSE, THE DATE AND DAY OF THE WEEK CAN BE OFF BY A DAY AND STILL BE COUNTED. E.G. TODAY'S DATE IS 5/10, SO 5/9, 5/10, | |
| MOCA3_2 MOCA3_3 | 2=DATE 3=YEAR 4=DAY OF THE WEEK 1=MONTH 2=DATE 3=YEAR 4=DAY OF THE WEEK 1=MONTH 2=DATE 3=YEAR 4=DAY OF THE WEEK 1=MONTH 2=DATE 3=YEAR 4=DAY OF THE WEEK | Thank you. Can you tell me today's date? IF RESPONDENT GIVES AN INCOMPLETE ANSWER, PROMPT ACCORDINGLY: Can you tell me the year, month, exact date, and day of the week? IN: MARK EACH CORRECT RESPONSE, THE DATE AND DAY OF THE WEEK CAN BE OFF BY A DAY AND STILL BE COUNTED. E.G. TODAY'S DATE IS 5/10, SO 5/9, 5/10, | |
| MOCA3_2 MOCA3_3 | 2=DATE 3=YEAR 4=DAY OF THE WEEK 1=MONTH 2=DATE 3=YEAR 4=DAY OF THE WEEK 1=MONTH 2=DATE 3=YEAR 4=DAY OF THE WEEK 1=MONTH 2=DATE 3=YEAR 4=DAY OF THE WEEK | Thank you. Can you tell me today's date? IF RESPONDENT GIVES AN INCOMPLETE ANSWER, PROMPT ACCORDINGLY: Can you tell me the year, month, exact date, and day of the week? IN: MARK EACH CORRECT RESPONSE, THE DATE AND DAY OF THE WEEK CAN BE OFF BY A DAY AND STILL BE COUNTED. E.G. TODAY'S DATE IS 5/10, SO 5/9, 5/10, | |
| MOCA3_2 MOCA3_3 | 2=DATE 3=YEAR 4=DAY OF THE WEEK 1=MONTH 2=DATE 3=YEAR 4=DAY OF THE WEEK 1=MONTH 2=DATE 3=YEAR 4=DAY OF THE WEEK 1=MONTH 2=DATE 3=YEAR 4=DAY OF THE WEEK | Thank you. Can you tell me today's date? IF RESPONDENT GIVES AN INCOMPLETE ANSWER, PROMPT ACCORDINGLY: Can you tell me the year, month, exact date, and day of the week? IN: MARK EACH CORRECT RESPONSE, THE DATE AND DAY OF THE WEEK CAN BE OFF BY A DAY AND STILL BE COUNTED. E.G. TODAY'S DATE IS 5/10, SO 5/9, 5/10, OR 5/11 ARE CORRECT | IF PROXY=1 OR 2 |

| Application - IRB00033 | 7770 | | |
|---|---|---|---|
| | | STREET ADDRESS ON | PROGRAMMING: |
| | | RECORD IS: [FILL] | THESE ARE |
| | | | PRELOADED |
| MOCA3f | ENTER CITY | Now, can you tell me the | PROGRAMMING: SKIP |
| | | city you live in? | IF PROXY=1 OR 2 |
| | | | PROGRAMMING: |
| | | CITY ON RECORD IS: [FILL] | THESE ARE |
| | | | PRELOADED |
| MOCA13_1 | 1=FACE | I read some words to you | PROGRAMMING: SKIP |
| | 2=VELVET | earlier, which I asked you to | IF PROXY=1 OR 2 |
| | 3=CHURCH | remember. Can you tell me | II TROXI-1 OR 2 |
| | 4=DAISY | those words? | |
| | 5=RED | | |
| | | CHECK EACH ONE THAT THE | |
| MOCA13_2 | 1=FACE | R SAYS CORRECTLY. | |
| _ | 2=VELVET | IN: IF R SAYS SIMILAR | |
| | 3=CHURCH | SOUNDING WORD, COUNT | |
| | 4=DAISY | AS CORRECT AND SAY: | |
| | 5=RED | Thank you. I will count that | |
| | | as the correct answer, but | |
| MOCA13_3 | 1=FACE | to clarify, the word was | |
| | 2=VELVET | [REPEAT WORD], spelled | |
| | 3=CHURCH | [SPELL WORD]. | |
| | 4=DAISY | [6. 22]. | |
| | 5=RED | | |
| MOCA13_4 | 1=FACE | | |
| | 2=VELVET | | |
| | 3=CHURCH | | |
| | 4=DAISY | | |
| | 5=RED | | |
| MOCA13_5 | 1=FACE | | |
| | 2=VELVET | | |
| | 3=CHURCH | | |
| | 4=DAISY | | |
| | 5=RED | | |
| MOCA_HELP | | Thank you. Let me help you | PROGRAMMING: SKIP |
| | | remember the ones you | IF PROXY=1 OR 2 |
| | | forgot. | |
| | | | PROGRAMMING: SKIP |
| | | | TO MED INTRO IF ALL |
| | | | FIVE (MOCA1a3- |
| | | | MOCA1e4) WERE |
| | | | CHECKED |
| MOCA4a_MISS | 1=FACE | IF MOCA1a3 MISSING: | PROGRAMMING: SKIP |
| | | | IF PROXY=1 OR 2 |
| | | | II TROXI-I OR 2 |

| Application - IRB00035998 | | | |
|---|---|---|---|
| | 8=DON'T KNOW (GO TO<br>MOCA4a_MISS2)<br>9=REFUSE (GO TO<br>MOCA4a_MISS2) | Do you remember the word that is a part of the body? | |
| MOCA4a_MISS2 | 1=FACE<br>2=OTHER RESPONSE<br>8=DON'T KNOW<br>9=REFUSE | Do you think the word was eyes, shoulder or face? | PROGRAMMING: SKIP IF PROXY=1 OR 2 PROGRAMMING: OTHER RESPONSE, DON'T KNOW AND REFUSE GO TO EITHER NEXT MISSED WORD OR MED INTRO IF NO MORE MISSED WORDS |
| MOCA4b_MISS | 1=VELVET<br>8=DON'T KNOW (GO TO<br>MOCA4b_MISS2)<br>9=REFUSE (GO TO<br>MOCA4b_MISS2) | IF MOCA1b3 MISSING:<br>Do you remember the word<br>that is a type of fabric? | PROGRAMMING: SKIP<br>IF PROXY=1 OR 2 |
| MOCA4b_MISS2 | 1=VELVET 2=OTHER RESPONSE 8=DON'T KNOW 9=REFUSE | Do you think the word was satin, velvet or cotton? | PROGRAMMING: SKIP IF PROXY=1 OR 2 PROGRAMMING: OTHER RESPONSE, DON'T KNOW AND REFUSE GO TO EITHER NEXT MISSED WORD OR MED INTRO IF NO MORE MISSED WORDS |
| MOCA4c_MISS | 1=CHURCH<br>8=DON'T KNOW (GO TO<br>MOCA4c_MISS2)<br>9=REFUSE (GO TO<br>MOCA4c_MISS2) | IF MOCA1c3 MISSING: Do you remember the word that is a place people go to worship? | PROGRAMMING: SKIP<br>IF PROXY=1 OR 2 |
| MOCA4c_MISS2 | 1=CHURCH<br>2=OTHER RESPONSE<br>8=DON'T KNOW<br>9=REFUSE | Do you think the word was library, church or store? | PROGRAMMING: SKIP IF PROXY=1 OR 2 PROGRAMMING: OTHER RESPONSE, DON'T KNOW AND REFUSE GO TO EITHER |

| Application - IRB000359 | 798 | | T |
|---|---|---|---|
| | | | NEXT MISSED WORD OR MED INTRO IF NO MORE MISSED WORDS |
| MOCA4d_MISS | 1=DAISY<br>8=DON'T KNOW (GO TO<br>MOCA4d_MISS2)<br>9=REFUSE (GO TO<br>MOCA4d_MISS2) | IF MOCA1d4 MISSING: Do you remember the word that is a type of flower? | PROGRAMMING: SKIP IF PROXY=1 OR 2 |
| MOCA4d_MISS2 | 1=DAISY<br>2=OTHER RESPONSE<br>8=DON'T KNOW<br>9=REFUSE | Do you think the word was rose, iris or daisy? | PROGRAMMING: SKIP IF PROXY=1 OR 2 PROGRAMMING: OTHER RESPONSE, DON'T KNOW AND REFUSE GO TO EITHER NEXT MISSED WORD OR MED INTRO IF NO MORE MISSED WORDS |
| MOCA4e_MISS | 1=RED<br>8=DON'T KNOW (GO TO<br>MOCA4e_MISS2)<br>9=REFUSE (GO TO<br>MOCA4e_MISS2) | IF MOCA1e4 MISSING: Do you remember the word that is a color? | PROGRAMMING: SKIP<br>IF PROXY=1 OR 2 |
| MOCA4e_MISS2 | 1=RED 2=OTHER RESPONSE 8=DON'T KNOW 9=REFUSE | Do you think the word was red, blue or green? | PROGRAMMING: SKIP IF PROXY=1 OR 2 PROGRAMMING: OTHER RESPONSE, DON'T KNOW AND REFUSE GO TO MED INTRO |
| MED_INTRO | | Thank you. The next 4 questions are about medications you take. Think about how you have taken your medications during the past four weeks when answering these questions. | PROGRAMMING: SKIP IF PROXY=1 OR 2 |
| MMAS1 | 0=NO (GO TO MMAS2<br>1=YES (GO TO MMAS2 | Do you ever forget to take your medicine? | PROGRAMMING: SKIP IF PROXY=1 OR 2 |

| Application - IRB0003: | 5998 | | |
|---|---|---|---|
| | 8=DON'T KNOW (GO TO | | |
| | MMAS2 | | |
| | 9=REFUSE (GO TO MMAS2 | | |
| MMAS2 | 0=NO (GO TO MMAS3 | Are you careless at times | PROGRAMMING: SKIP |
| | 1=YES (GO TO MMAS3 | about taking your | IF PROXY=1 OR 2 |
| | | medicine? | |
| | 8=DON'T KNOW (GO TO | | |
| | MMAS3 | | |
| | 9=REFUSE (GO TO MMAS3 | | |
| MMAS3 | 0=NO (GO TO MMAS4 | Sometimes if you feel | PROGRAMMING: SKIP |
| | 1=YES (GO TO MMAS4 | worse when you take the | IF PROXY=1 OR 2 |
| | | medicine, do you stop | |
| | 8=DON'T KNOW (GO TO | taking it? | |
| | MMAS4 | | |
| | 9=REFUSE (GO TO MMAS4 | | |
| MMAS4 | 0=NO (GO TO BPHome | When you feel better, do | PROGRAMMING: SKIP |
| | Intro) | you sometimes stop taking | IF PROXY=1 OR 2 |
| | 1=YES (GO TO BPHome | your medicine? | |
| | Intro) | | |
| | 8=DON'T KNOW (GO TO | | |
| | BPHome Intro) | | |
| | 9=REFUSE (GO TO BPHome | | |
| | Intro) | | |
| BPHome_Intro | | Now I'd like to ask some | |
| | | questions about checking | |
| | | your/his/her blood pressure | |
| | | and your/his/her usual or | |
| | | regular health care | |
| BBU | | provider. | |
| BPHome | 0=NO (GO TO BPVAL) | Do/Does you/he/she check | |
| | 1=YES (GO TO BPFREQ) | your/his/her blood pressure | |
| | | at home? | |
| | 8=DON'T KNOW(GO TO | IN. DD COLUD DE CLIECKED | |
| | PCP) | IN: BP COULD BE CHECKED | |
| | 0-DEFLICE/CO TO DCD) | BY A FAMILY MEMBER, | |
| | 9=REFUSE(GO TO PCP) | FRIEND. ANY CHECKING OF BP SINCE INITIAL | |
| | | HOSPITALIZATION WOULD | |
| | | QUALIFY AS A YES. | |
| BPFREQ | 1=daily (GO TO BPVALsys) | How frequently do/does | |
| BFFNEQ | 2=weekly or (GO TO | you/he/she check | |
| | BPVALsys) | your/his/her blood | |
| | 3=monthly? (GO TO | pressure? | |
| | BPVALsys) | Would you say | |
| | D: 17.123437 | Trodia you say | |

| Application - IKB00033998 | | |
|---|---|---|
| | 8=DON'T KNOW (GO TO<br>BPVALsys)<br>9=REFUSE (GO TO<br>BPVALsys) | |
| BPVALsys | Enter number between 50 and 250. (GO TO BPVALdia) 8=DON'T KNOW(GO TO PCP) 9=REFUSE(GO TO PCP) | What was the value of your/his/her last blood pressure? Please provide the systolic (top number) and diastolic (bottom number). IN: ENTER TOP NUMBER HERE AND BOTTOM NUMBER ON FOLLOWING SCREEN. IF NEEDED: We are interested in your most recent BP no matter who took the measurement. |
| BPVALdia | Enter number between 35 and 135. (GO TO BPWHO) | What was the value of your/his/her last blood pressure? Please provide the systolic (top number) and diastolic (bottom number). IN: ENTER BOTTOM NUMBER HERE |
| ВРЖНО | 1=you/the patient himself/the patient herself 2= a healthcare professional 3= a family member, or 4= someone else? (GO TO BPWHO_OTHER) | Was this blood pressure measurement taken by |
| BPWHO_OTHER | OPEN TEXT<br>(50 CHARACTERS) | Who took the blood pressure? |
| PCP | 0=NO (GO TO PTVIS) 1=YES (GO TO PCPVIS) 8=DON'T KNOW (GO TO PTVIS) 9=REFUSE (GO TO PTVIS) | Is there a particular doctor's office, health center, or other place that you/he/she usually go/goes if you/he/she are/is sick and |

| Application - IKB00035998 | T | |
|---|---|---|
| | | need/needs advice about your/his/her health? |
| | | IN: THIS COULD INCLUDE ANY TYPE OF DOCTOR IF THE RESPONDENT USES THEM REGULARLY. IT DOES NOT INCLUDE A HOSPITAL EMERGENCY DEPARTMENT. |
| PCPvis | 0=NO (GO TO PTVIS) 1=YES(GO TO PTVIS) 8=DON'T KNOW(GO TO PTVIS) 9=REFUSE(GO TO PTVIS) | Have/Has you/he/she visited a doctor or nurse from that office, health center or other place since you/he/she were/was discharged from the hospital after your/his/her stroke? |
| PTvis | 0=NO (GO TO OTvis) 1=YES (GO TO PTvisL) 8=DON'T KNOW (GO TO OTvis) 9=REFUSED (GO TO OTvis) | Since you/he/she were/was discharged home on [PRELOAD DISCHARGE OR NEW_DISCHARGE, IF FILLED] after your/his/her stroke or TIA, have/has you/he/she received any services from a physical therapist? IF NEEDED: Physical therapists help patients with their mobility, (for example, walking, moving from sitting to standing, going up stairs, getting in and out of bed) and physical activity. |
| PTvisL | 1=your/his/her home (GO TO OTvis) 2=an outpatient clinic, or (GO TO OTvis) 3=both? (GO TO OTvis) 8=DON'T KNOW (GO TO OTvis) 9=REFUSED (GO TO OTvis) | Did you/he/she receive the services in |

| Application - IKB000. | | |
|---|---|---|
| OTvis | 0=NO (GO TO STvis) 1=YES (GO TO OTvisL) 8=DON'T KNOW (GO TO STvis) 9=REFUSED (GO TO STvis) | Since you/he/she were/was discharged home on <autofill date=""> after your/his/her stroke or TIA, have/has you/he/she received any services from an occupational therapist? IF NEEDED: Occupational therapists help patients with their activities of daily</autofill> |
| | | living (for example, dressing, bathing, cooking, eating). |
| OTvisL | 1=your/his/her home (GO TO STvis) 2=an outpatient clinic, or (GO TO STvis) 3=both? (GO TO STvis) | Did you/he/she receive the services in |
| | 8=DON'T KNOW (GO TO<br>STvis)<br>9=REFUSED (GO TO STvis) | |
| STvis | 0=NO (GO TO FALL_INTRO) 1=YES (GO TO STvisL) 8=DON'T KNOW (GO TO FALL_INTRO) 9=REFUSED (GO TO FALL_INTRO) | Since you/he/she were/was discharged home on <autofill date=""> after your/his/her stroke or TIA, have/has you/he/she received any services from a speech therapist?</autofill> |
| | | IF NEEDED: Speech therapists help patients with their communication and swallowing. |
| STvisL | 1=your/his/her home<br>2=an outpatient clinic, or<br>3=both? | Did you/he/she receive the services in |
| | 8=DON'T KNOW (GO TO<br>FALL_INTRO)<br>9=REFUSED (GO TO<br>FALL_INTRO) | |
| Application - IRB0003 | 3778<br> | |
|---|---|---|
| FALL_INTRO | | The next few questions are about any falls or hospitalizations you've/he's/she's had since your/his/her stroke/TIA. |
| Fall1 | 0=NO (GO TO ReAdmit) 1=YES (GO TO Fall2) 8=DON'T KNOW (GO TO ReAdmit) 9=REFUSE (GO TO ReAdmit) | Since you/he/she were/was discharged from the hospital on [PRELOAD DISCHARGE DATE] after your/his/her stroke or TIA, have/has you/he/she fallen? |
| Fall2 | 0=NO (GO TO Fall3) 1=YES (GO TO Fall3) 8=DON'T KNOW (GO TO Fall3) 9=REFUSE (GO TO Fall3) | Did you/he/she get injured<br>and need to go to the<br>doctor or emergency room<br>due to a fall? |
| Fall3 | 0=NO (GO TO ReAdmit) 1=YES (GO TO FALL4) 8=DON'T KNOW (GO TO READMIT) 9=REFUSE (GO TO READMIT) | Have/Has you/he/she fallen<br>more than once since<br>your/his/her stroke? |
| FALL4 | Enter a number between 2<br>and 99. (GO TO ReAdmit)<br>8=DON'T KNOW (GO TO<br>ReAdmit)<br>9=REFUSE (GO TO ReAdmit) | How many times have/has you/he/she fallen? IF NEEDED: A best guess is fine. |
| ReAdmit | 0=NO (GO TO PROMIS_INTRO) 1=YES (GO TO READMITN) 8=DON'T KNOW (GO TO PROMIS_INTRO ) 9=REFUSE (GO TO PROMIS_INTRO ) | Since you/he/she were/was discharged from the hospital on <date>, have/has you/he/she been hospitalized overnight for any reason?</date> |
| ReAdmitN | Enter a number between 1 and 99. (GO TO PROMIS_INTRO) | How many times have/has you/he/she been in the |

| Application - IRB00035998 | | 1 | |
|---|---|---|---|
| | 8=DON'T KNOW (GO TO<br>PROMIS_INTRO)<br>9=REFUSE (GO TO<br>PROMIS_INTRO) | hospital overnight for any reason? IN NOTE: WE ARE | |
| | | INTERESTED IN NUMBER OF ADMISSIONS, NOT NIGHTS | |
| PROMIS_INTRO | | The next few questions are about feelings of tiredness or fatigue | PROGRAMMING: SKIP<br>IF PROXY=1 OR 2 |
| PROMIS1 | 1=Not at all 2=A little bit 3=Somewhat 4=Quite a bit 5=Very much 8=DON'T KNOW 9=REFUSE | During the past 7 days, how often have you felt tired or fatigued? Would you say | PROGRAMMING: SKIP IF PROXY=1 OR 2 |
| PROMIS2 | 1=Not at all 2=A little bit 3=Somewhat 4=Quite a bit 5=Very much 8=DON'T KNOW 9=REFUSE | During the past 7 days, how often have you had trouble starting things because you were tired? Would you say | PROGRAMMING: SKIP IF PROXY=1 OR 2 |
| PROMIS3 | 1=NOT AT ALL 2=A LITTLE BIT 3=SOMEWHAT 4=QUITE A BIT 5=VERY MUCH 8=DON'T KNOW 9=REFUSE | (In the past 7 days,) how run-down did you feel on average? (Would you say) | PROGRAMMING: SKIP IF PROXY=1 OR 2 |
| PROMIS4 | 1=NOT AT ALL 2=A LITTLE BIT 3=SOMEWHAT 4=QUITE A BIT 5=VERY MUCH 8=DON'T KNOW 9=REFUSE | (In the past 7 days,) how fatigued were you on average? (Would you say) | PROGRAMMING: SKIP IF PROXY=1 OR 2 |
| SATIS_INTRO | | The next several questions are about the care you've/he's/she's received from your/his/her physicians, nurses and other health care providers since you/he/she had your/his/her stroke or TIA. | |

| rippiication ittboo | | |
|---|---|---|
| Satis1 | 1=Never 2=Sometimes 3=Usually 4=Always 8=DON'T KNOW 9=REFUSE | Thinking about the care you/he/she have/has received for your/his/her stroke or TIA recovery since you/he/she were/was discharged from the hospital on [PRELOAD DISCHARGE DATE], how often did your/his/her physicians, nurses and other health care providers Explain things in a way that was easy [for him/her] to understand? Would you say INTERVIEWER NOTE: PATIENTS SHOULD THINK ABOUT THE CARE THEY'VE RECEIVED FROM ALL OF THEIR PHYSICIANS (E.G., SPECIALIST AND |
| Satis2 | 1=Never 2=Sometimes 3=Usually 4=Always 8=DON'T KNOW 9=REFUSE | PRIMARY CARE PROVIDERS) (Thinking about the health care providers you/he/she have/has seen since you/he/she were/was discharged from the hospital) How often did these providers listen carefully to you/him/her? Would you say |
| Satis3 | 1=NEVER 2=SOMETIMES 3=USUALLY 4=ALWAYS 8=DON'T KNOW 9=REFUSE | (Thinking about the health care providers you/he/she have/has seen since you/he/she were/was discharged from the hospital) How often did they seem to know the important |

| Application - IRB00035998 | | |
|---------------------------|--------------|-----------------------------|
| | | information about |
| | | your/his/her medical |
| | | history? |
| | | (Would you say) |
| Satis4 | 1=NEVER | (Thinking about the health |
| | 2=SOMETIMES | care providers you/he/she |
| | 3=USUALLY | have/has seen since |
| | 4=ALWAYS | you/he/she were/was |
| | 8=DON'T KNOW | discharged from the |
| | 9=REFUSE | hospital, |
| | J-KEI OSE | How often did they) Show |
| | | respect for what |
| | | you/he/she had to say? |
| Satis5 | 1_NEVED | (Would you say) |
| Jalisa | 1=NEVER | (Thinking about the health |
| | 2=SOMETIMES | care providers you/he/she |
| | 3=USUALLY | have/has seen since |
| | 4=ALWAYS | you/he/she were/was |
| | 8=DON'T KNOW | discharged from the |
| | 9=REFUSE | hospital, How often did |
| | | they) Spend enough time |
| | | with you/him/her? |
| | | (Would you say) |
| Satis6 | 1=NEVER | (Thinking about the health |
| | 2=SOMETIMES | care providers you/he/she |
| | 3=USUALLY | have/has seen since |
| | 4=ALWAYS | you/he/she were/was |
| | 8=DON'T KNOW | discharged from the |
| | 9=REFUSE | hospital, How often did |
| | | they)Talk about all the |
| | | prescription medicines |
| | | you/he/she were/was |
| | | taking? |
| | | (Would you say) |
| COMRES_INTRO | | Now I'd like to ask you |
| <del>-</del> | | about any community |
| | | services you/he/she |
| | | have/has used since |
| | | your/his/her stroke or TIA |
| ComRes1 | 0=NO | Thinking back since |
| | 1=YES | discharge from the hospital |
| | 1-123 | after your/his/her stroke, |
| | S-DON'T KNOW | |
| | 8=DON'T KNOW | have/has you/he/she used |
| | 9=REFUSE | any adult day care |
| | | programs or other adult |

| Αp | plication | _ | IRB00035998 | 8 |
|----|-----------|---|-------------|---|

| Application - IKB00033998 | | services for social support or recreation for stroke survivors? NOTE: These are programs that provide care and companionship for older adults who need assistance or supervision during the day. These programs offer some relief to family members and caregivers. |
|---|---|---|
| ComRes2 | 0=NO<br>1=YES<br>8=DON'T KNOW<br>9=REFUSE | Since discharge from the hospital after your/his/her stroke, have/has you/he/she used community services or classes to help with your ability to speak, read, or write? IN NOTE: An example would be an aphasia support group. |
| ComRes3 | 0=NO<br>1=YES<br>8=DON'T KNOW<br>9=REFUSE | Since discharge from the hospital after your/his/her stroke, have/has you/he/she used counseling services or therapy for stress or depression IN NOTE: (An example is CareNet counseling)? |
| ComRes4 | 0=NO<br>1=YES<br>8=DON'T KNOW<br>9=REFUSE | (Since discharge from the hospital after your/his/her stroke) How about any programs that promote healthy living like classes on diet or managing diabetes? IN NOTE: Other examples include classes on managing chronic pain, problems with |

Application - IRB00035998

| Application - IRB000 | 35998 | |
|---|---|---|
| | | breathing, high blood pressure. |
| ComRes5 | 0=NO<br>1=YES<br>8=DON'T KNOW<br>9=REFUSE | (Since discharge from the hospital after your/his/her stroke) How about exercise classes that are open to the general public, like ones offered at a church or fitness center? |
| ComRes6 | 0=NO<br>1=YES<br>2=DOES NOT SMOKE<br>8=DON'T KNOW<br>9=REFUSE | (Since discharge from the hospital after your/his/her stroke, how about) programs to help you quit smoking? |
| ComRes7 | 0=NO<br>1=YES<br>8=DON'T KNOW<br>9=REFUSE | (Since discharge from the hospital after your/his/her stroke, how about) a falls prevention program that teaches you how to improve your balance and strength so you don't fall? |
| ComRes8 | 0=NO<br>1=YES<br>8=DON'T KNOW<br>9=REFUSE | (Since discharge from the hospital after your/his/her stroke, how about) programs that provide meals – either delivered to your house or a central location like a church or community center? |
| ComRes9 | 0=NO<br>1=YES<br>8=DON'T KNOW<br>9=REFUSE | (Since discharge from the hospital after your/his/her stroke, how about) a support group for stroke survivors? IN NOTE: these are groups that provide social support, information, and resources for stroke survivors |
| ComRes10 | 0=NO<br>1=YES | (Since discharge from the hospital after your/his/her stroke, how about) |

| Application - IRB00035998 | | |
|---|---|---|
| | 8=DON'T KNOW 9=REFUSE | medication assistance or management services to help pay for the medications or to help understand and manage the medications? IN NOTE: management services are usually offered by pharmacists. |
| ComRes11 | 0=NO<br>1=YES<br>8=DON'T KNOW<br>9=REFUSE | (Since discharge from the hospital after your/his/her stroke, how about) transportation services to get you to your healthcare appointments or community activities? IN NOTE: THIS DOES NOT INCLUDE REGULAR PUBLIC |
| ComRes12 | 0=NO<br>1=YES<br>8=DON'T KNOW<br>9=REFUSE | TRANSPORTATION (Since discharge from the hospital after your/his/her stroke, how about) support services for your family or caregivers? IN NOTE: these are groups or services that provide social support, information, and resources for caregivers/family members of storke survivors? |
| ComRes13 | 0=NO (GO TO EDUC) 1=YES (GO TO COMRES14) 8=DON'T KNOW (GO TO EDUC) 9=REFUSE (GO TO EDUC) | Are there any other services you've/he's/she's used that I haven't mentioned? |
| ComRes14 | SPECIFY OTHER OPEN TEXT [250 CHAR] | What are those? |

| Educ | 1=8TH GRADE OR LESS 2=SOME HIGH SCHOOL, BUT DID NOT GRADUATE 3=HIGH SCHOOL GRADUATE OR GED 4=SOME COLLEGE OR 2- YEAR DEGREE 5=4-YEAR COLLEGE GRADUATE 6=MORE THAN 4-YEAR COLLEGE DEGREE 8=DON'T KNOW 9=REFUSE | What is the highest grade or level of school that you/he/she have/has completed? |
|---|---|---|
| PROMIS_INTRO | EMPTY | These last few questions are about your health and how you have been feeling. |
| Global01 | 1=Excellent<br>2=Very good<br>3=Good<br>4=Fair, or<br>5=Poor | In general, would you say your health is |
| Global02 | 1=Excellent<br>2=Very good<br>3=Good<br>4=Fair, or<br>5=Poor | In general, would you say your quality of life is |
| Global03 | 1=EXCELLENT<br>2=VERY GOOD<br>3=GOOD<br>4=FAIR, OR<br>5=POOR | In general, how would you rate your physical health? (Would you say) |
| Global04 | 1=EXCELLENT<br>2=VERY GOOD<br>3=GOOD<br>4=FAIR, OR<br>5=POOR | In general, how would you rate your mental health, including your mood and your ability to think? (Would you say) |
| Global05 | 1=EXCELLENT<br>2=VERY GOOD<br>3=GOOD<br>4=FAIR, OR<br>5=POOR | In general, how would you rate your satisfaction with your social activities and relationships? (Would you say) |

| Application - IRB0003. | | |
|---|---|---|
| Global09 | 1=EXCELLENT 2=VERY GOOD 3=GOOD 4=FAIR, OR 5=POOR | In general, please rate how well you carry out your usual social activities and roles. This includes activities at home, at work and in your community, and responsibilities as a parent, child, spouse, employee, friend, etc. (Would you say) |
| Global06 | 1=Completely 2=Mostly 3=Moderately 4=A little, or 5=Not at all | To what extent are you able to carry out your everyday physical activities such as walking, climbing stairs, carrying groceries, or moving a chair? Would you say |
| Global10 | 1=Never<br>2=Rarely<br>3=Sometimes<br>4=Often, or<br>5=Always | In the past 7 days, how often have you been bothered by emotional problems such as feeling anxious, depressed or irritable? Would you say |
| Global08 | 1=None 2=Mild 3=Moderate 4=Severe, or 5=Very severe | In the past 7 days, how would you rate your fatigue on average? Would you say |
| Global07 | ENTER NUMBER<br>(RANGE 0-10) | Picture a scale from 0 to 10, with zero being no pain and ten being the worst imaginable pain. In the past 7 days, how would you rate your pain on average? |
| THANK_YOU | | Thank you. That's the end of the survey. Goodbye. |

# Appendix 24 - 90d Patient Survey (Full Survey Mailed with the 80 day letter)



This is a copy of the questions you will be asked during the phone call. You do not have to fill this out, but can if you would like to prepare for the call. It will be helpful to have this copy with you during the call.

A. <u>PHYSICAL CHALLENGES SINCE YOUR HOSPITAL VISIT</u>: These questions are about the physical problems you may have experienced recently because of your stroke or TIA. ("TIA" stands for *transient ischemic attack* and is sometimes referred to as a *mini-stroke*, *warning stroke*, *brain episode*, or *brain bleed*.) We want to know <u>from your point of view</u> how your stroke or TIA has affected your physical function in the past 2 weeks?

| In the past 2 weeks, how difficult was it to | Not difficult at all | A little<br>difficult | Somewhat<br>difficult | Very<br>difficult | Could not do at all |
|---|---|---|---|---|---|
| Dress the top part of your body? | | | | | |
| Bathe yourself? | | | | | |
| Get to the toilet on time? | | | | | |
| Control your bladder (not have an accident)? | | | | | |
| Control your bowels (not have an accident)? | | | | | |
| Stand without losing balance? | | | | | |
| Go shopping? | | | | | |
| Do heavy household chores (e.g. vacuum, laundry or yard work)? | | | | | |
| Stay sitting without losing your balance? | | | | | |
| Walk without losing your balance? | | | | | |
| Move from a bed to a chair? | | | | | |
| Walk fast? | | | | | |
| Climb one flight of stairs? | | | | | |
| Walk one block? | | | | | |
| Get in and out of a car? | | | | | |
| Carry heavy objects (e.g. bag of groceries) with your affected hand? | | | | | |

| | ENERAL HEALTH Q<br>eneral health. | UESTIONS: These | questions are | about how you p | erceive or view | your |
|---|---|---|---|---|---|---|
| 1. | Compared to others scale between 1 and | | | | ur stroke or TIA | using a |
| | Poor | Fair | Good | Very Good | Excellent | |
| 2. | Over the next 3 mon Improve Stay the sa Get worse | - | 3<br>ur health is goi | ng to: | 5 | |
| as | EVEL OF ASSISTAN<br>ssistance you may or<br>roke (or TIA). | | | | | |
| 1. | Could you live alone use the toilet, prepa ☐ Yes ☐ No | | | | s being able to | bathe, |
| 2. | Can you do everythinot as much? ☐ Yes ☐ No | ng that you were do | ing right before | e your stroke (or | TIA), even if slo | wer and |
| 3. | Are you completely ☐ Yes ☐ No | back to the way you | were right befo | ore your stroke ( | or TIA)? | |
| 4. | Can you walk from o ☐ Yes ☐ No | one room to another | without help fr | om another pers | on? | |
| 5. | Can you sit up in be<br>☐ Yes<br>☐ No | d without any help? | | | | |
| | | | | | | 2 |

| haves | SICAL ACTIVITY QUESTIONS: The next few questions are about the amount of time you spent walking in the last 7 days. g the last seven days: |
|---|---|
| 1. | Did you walk continuously for at least 10 minutes on any day? ☐ Yes ☐ No |
| 2. | On how many days did you walk continuously, for at least 10 minutes, for recreation, exercise, or to get to or from places? |
| | Enter a number from 0 - 7: |
| 3. | On days that you walked for at least 10 minutes, how much total time <u>per day</u> did you spend walking? |
| | Enter a number minutes |
| 4. | What is the total amount of time you spent walking over the last seven days? Enter a number minutes |
| | D QUESTIONS: The next 2 questions are about your mood over the past 2 weeks. the <u>past two weeks</u> , how often have you been bothered by any of the following problems: |
| 1. Lit | tle interest or pleasure in doing things: |
| | <ul> <li>□ Not at all</li> <li>□ Several days</li> <li>□ More than half of the days</li> <li>□ Nearly every day</li> </ul> |
| 2. Fe | eling down, depressed, or hopeless: |
| | □ Not at all □ Several days □ More than half the days □ Nearly every day |
| | rviewer will now ask you some questions to assess your memory. |
| The inte | rviewer will now ask you some questions to assess your memory. |
| | re not printed on the survey because they need to be asked over the phone. |

| | EDICATION QUESTIONS: The next 4 questions are about medications you take. Think about w you have taken your medications during the past 4 weeks when answering these questions. |
|---|---|
| 1. | Do you ever forget to take your medicine? ☐ Yes ☐ No |
| 2. | Are you careless at times about taking your medicine? ☐ Yes ☐ No |
| 3. | Sometimes if you feel worse when you take the medicine, do you stop taking it? ☐ Yes ☐ No |
| 4. | When you feel better, do you sometimes stop taking your medicine? ☐ Yes ☐ No |
| i. <u>SE</u><br>yo | ELF-MANAGEMENT & USE OF CARE QUESTIONS: These next questions are about checking ur blood pressure and your usual health care provider. |
| 1. | Do you check your blood pressure <u>at home</u> ? ☐ Yes ☐ No |
| | 1a. If yes, how frequently do you check your blood pressure? ☐ Daily ☐ Weekly ☐ Monthly |
| | 1b. What was the value of your last blood pressure? Please provide the systolic (top number) and diastolic (bottom number). |
| | (systolic) /(diastolic) |
| | 1c. Who took this blood pressure measurement? ☐ You ☐ A healthcare professional ☐ A family member ☐ Someone else: (please specify) |
| 2. | Is there a particular doctor's office, health center, or other place that you usually go if you are sick and need advice about your health? ☐ Yes ☐ No |
| | 2a. If yes, have you visited a doctor or nurse from that office, health center, or other place since you were discharged from the hospital after your stroke (or TIA)? ☐ Yes ☐ No |

| 3.a. Since you were discharged home after your stroke (or TIA), have you received any services from: | | 3.b. If yes, did you receive services in: | | |
|---|---|---|---|---|
| | | Your home? | Outpatient clinic? | Both? |
| i. A physical therapist? | ☐ Yes<br>☐ No | | | |
| ii. An occupational therapist? | □ Yes<br>□ No | | | |
| iii. A speech therapist? | □ Yes<br>□ No | | | |
| fall?<br>□ Yes | from the l<br>tinjured a | hospital after you | ir stroke (or TIA), have the doctor or emerge | ncy room due to |
| | □ No | | | |
| 1c. If yes, how many | times hav | ve you fallen? | | |
| Enter a number | | | | |
| 2. Since you were discharged reason? | from the | hospital, have yo | u been hospitalized o | vernight for any |
| □ Yes □ No | | | | |
| 2a. If yes, how many | times hav | ve you been in the | e hospital overnight fo | or any reason? |

| | ng the past 7 days how often<br>you: | Not At all | A little b | t Sor | newhat | Quite | e a bit | Very<br>much |
|---|---|---|---|---|---|---|---|---|
| 1. | Felt tired or fatigued? | | | | | 1 | | |
| 2. | Had trouble <u>starting</u> things<br>because you were tired? | | | | | [ | 2 | - |
| n the | e past 7 days: | Not At all | A little b | t Soi | mewhat | Quite | e a bit | Very<br>much |
| 3. | How run-down did you feel<br>on average? | | 0 | | | | | |
| 4. | How fatigued were you on average? | | | | | | | |
| Γhink | oke (or TIA). king about the care you have re | eceived for yo | our stroke | (or TIA | ) recove | ry sind | ce you v | vere |
| str<br>Think | ************************************* | eceived for yo<br>often did you | r physicia | (or TIA<br>ns, nur<br>Never | ses, and | other | ce you v<br>healthc<br>Usually | are provide |
| str<br>Fhink<br>disch | king about the care you have re | often did you | r physicia | ns, nur | ses, and | other | healthc | are provide |
| str<br>Think<br>disch | king about the care you have re<br>narged from the hospital, how o | often did you | r physicia | Never | ses, and | other | Healthc<br>Usually | are provide Always |
| str<br>Think<br>disch | king about the care you have re<br>narged from the hospital, how o<br>l. Explain things in a way that<br>understand? | was easy to | r physicia | Never | Someti | other | Healthc Usually | are provide |
| str<br>Think<br>disch | ing about the care you have re<br>narged from the hospital, how on<br>the hospital, how on<br>the hospital, how on<br>the hospital, how on<br>the hospital has a way that<br>understand? | was easy to | r physicia | Never | Someti | other | Usually | Always |
| str<br>Fhink<br>Idisch | ing about the care you have reparted from the hospital, how consider the hospital from the hospital, how consider the hospital from the ho | was easy to | r physicia | Never | Ses, and | other | Usually | Always |

6

I. FATIGUE QUESTIONS: The next few questions are about feelings of tiredness or fatigue.

K. <u>COMMUNITY RESOURCES QUESTIONS</u>: These next questions are about any community services you have used since your stroke (or TIA).

Thinking back since you were discharged from the hospital after your stroke (or TIA), have you used any of the following services to assist you with your care?

| | d any of the following services to assist you with your care? | Yes | No |
|---|---|---|---|
| 1. | Adult day care programs or other services for social support or recreation for stroke (or TIA) survivors | 0 | |
| 2. | Community services or classes to help with your ability to speak, read, or write (e.g. Aphasia Support Group) | | 0 |
| 3. | Counseling services or therapy for stress or depression (e.g. CareNet counseling) | 0 | |
| 4. | Any programs that promote healthy living, like classes on diet or managing diabetes, chronic pain, problems with breathing, or high blood pressure | | |
| 5. | Exercise classes that are open to the general public, like ones offered at a church or fitness center (e.g. Silver Sneakers, Silver & Fit, Hospital wellness programs) | 0 | |
| 6. | Programs to help you quit smoking | | |
| 7. | Falls prevention program that teaches you how to improve your balance and strength so you don't fall | | |
| 8. | Programs that provide meals (delivered to your house or a central location like a church or community center) | П | |
| 9. | A support group for stroke (or TIA) survivors | | |
| 10 | . Medication assistance or management services to help pay for the medications or to help understand and manage the medications | | |
| 11 | . Transportation services to get you to your healthcare appointments or community activities | | |

| 12. Support services for your family/caregivers | | |
|---|---|---|
| 13. Other services? If yes, describe: | | |
| L EDUCATION QUESTION: | | |
| L. EDUCATION QUESTION: 1. What is the highest grade or level of school that you have completed? 8 <sup>th</sup> grade or less Some high school, but did not graduate High school graduate or GED Some college or 2-year degree 4-year college graduate More than 4-year college degree | | |
| M. <u>PRIMARY CAREGIVER</u> : Please verify who is the family member, friend, or nei have helped you with activities such as shopping and transportation since your receivable. | | |
| THIS IS THE END OF THE SURVEY - THANK YO | U! | |
| The website for this study can be accessed at: <a href="https://www.nccompass-study.org">https://www.nccompass-study.org</a> | rg/ | |
| If you have any questions about the study, please contact our project manager at 1 | -844-501- | 7668. |
| If you have any questions about your rights as a research study participant, you may anonymously if you wish, the Institutional Review Board. Their job is to protect your as a research participant. They have reviewed and approved this study. You can respect you go you will be you will be a subject of the study. You can respect you will be you will be you will be you will be you will be you will you will be you | rights and | d welfare |
| | | 8 |

# Appendix 25 – 90d Patient Non-Responder Survey and Letter (Mailed if unable to reach over phone)

Dear <NAME>, <DATE>

Greetings from the COMPASS Study team! We are working with your care team at <HOSPITAL NAME> to find the best ways to improve healthcare for people who had a transient ischemic attack (TIA), mini-stroke, stroke, or related episode. A few weeks ago we tried calling you and are sorry that we haven't been able to reach you!

We'd like to know how you've been doing since your hospital visit 3 months ago. Your participation is completely voluntary and confidential. Your response is very valuable and will help improve healthcare for others in North Carolina.

### How you can participate:

[-] Answer the questions on the next page and mail the completed survey back to us in the postage-paid envelope. Please return it within 5 days.

OR

[-] Contact us, toll-free, at 1-844-501-7668 if you would prefer to answer the questions by phone.

**This is your last chance to let us know how you are doing.** We need your help and thank you for your valuable contribution!

### Find out more about the COMPASS Study:

[-] To learn more about the COMPASS Study please visit our website:

### www.nccompass-study.org

[-] If you would like to speak with a team member about the study, call us at:

1-844-501-7668

Thanks for filling out the included survey and returning it to us!

Best regards,

The COMPASS Study Team



We are sorry to have missed you on the phone. We value your response and hope you will complete this brief questionnaire. Please return it within 5 days in the envelope provided.

A. <u>PHYSICIAL CHALLENGES SINCE YOUR HOSPITAL VISIT</u>: These questions are about the physical problems you may have experienced recently because of your stroke or TIA. ("TIA" stands for *transient ischemic attack* and is sometimes referred to as a *mini-stroke*, *warning stroke*, *brain episode*, or *brain bleed*.) We want to know <u>from your point of view</u> how has your stroke or TIA affected your physical function in the past 2 weeks?

| In the past 2 weeks, how difficult was it to | Not difficult at all | A little<br>difficult | Somewhat<br>difficult | Very<br>difficult | Could not do at all |
|---|---|---|---|---|---|
| Dress the top part of your body? | | | | | |
| Bathe yourself? | | | | | |
| Get to the toilet on time? | | | | | |
| Control your bladder (not have an accident)? | | | | | |
| Control your bowels (not have an accident)? | | | | | |
| Stand without losing balance? | | | | | |
| Go shopping? | | | | | |
| Do heavy household chores (e.g. vacuum, laundry or yard work)? | | | | | |
| Stay sitting without losing your balance? | | | | | |
| Walk without losing your balance? | | | | | |
| Move from a bed to a chair? | | | | | |
| Walk fast? | | | | | |
| Climb one flight of stairs? | | | | | |
| Walk one block? | | | | | |
| Get in and out of a car? | | | | | |
| Carry heavy objects (e.g. bag of groceries) with your affected hand? | | | | | |

1

| B. | <b>GENERAL HEALTH QUESTIONS:</b> | These questions are about how you perceive or view your |
|---|---|---|
| | general health. | |

1. Compared to others your age, how would you rate your health since your stroke or TIA using a scale between 1 and 5 with 1 being "poor" and 5 being "excellent?"

| Poor | Fair | Good | Very Good | Excellent |
|------|------|------|-----------|-----------|
| 1 | 2 | 3 | 4 | 5 |

| 2. | Over the next | 3 months, | do | you think | your | health | is | going 1 | to: |
|---|---|---|---|---|---|---|---|---|---|
|---|---|---|---|---|---|---|---|---|---|

☐ Improve

☐ Stay the same

☐ Get worse

| 3. | What was the value of your last blood pressure? | Please provide the systolic (top number) and |
|---|---|---|
| | diastolic (bottom number). | |

| (systolic) / | (diastolic) |
|--------------|-------------|
| (SVSIDIIC) / | totasioner |

### THIS IS THE END OF THE SURVEY - THANK YOU!

The website for this study can be accessed at: <a href="https://www.nccompass-study.org/">https://www.nccompass-study.org/</a>

If you have any questions about the study, please contact our project manager at 1-844-501-7668.

If you have any questions about your rights as a research study participant, you may contact, anonymously if you wish, the Institutional Review Board. Their job is to protect your rights and welfare as a research participant. They have reviewed and approved this study. You can reach them at 919-966-3113 or by email to <a href="mailto:IRB\_subjects@unc.edu">IRB\_subjects@unc.edu</a>.

### Appendix 26 - Caregiver Letter (First Attempt)



Dear < NAME CG>,

<DATE>

Greetings from the COMPASS Study team! We are writing to invite you to participate in our survey. With your help, we hope to understand more about the best way to care for stroke survivors and their families after they go home from the hospital - to help them find the way forward to recovery.

We know how important family, friends, and neighbors are during the recovery process. We also understand that it can be difficult to care for loved ones who have had a stroke. Through the COMPASS Study, we hope to learn more about the needs of those who provide care and assistance to stroke survivors.

<PATIENT NAME> has identified you as the person who has been helping <HIM/HER> recover following <HIS/HER> stroke. <HE/SHE> was discharged on <DSCHRGDATE> from <HOSPITAL NAME>, which is participating in the COMPASS study. We invite you to take part in the COMPASS Study by completing a survey about caring for <HIM/HER>. This survey should only take about 15 minutes and is completely voluntary and confidential.

Your input is important and will help us improve support systems for family members and friends who provide care to stroke survivors. Please complete the enclosed survey and send it back in the postage-free envelope we have provided by < Due Date>

### Find out more about the COMPASS Study



To learn more about the COMPASS Study and to find other useful information about care after stroke, please visit our website: www.nccompass-study.org



If you would like to speak with a team member about the study, call us at:

We thank you very much for your time and contribution to the COMPASS Study!

Best regards, The COMPASS Study Team

<CG\_ID>



# Appendix 27 - Caregiver Survey

| CAL | REG | HVER | <b>OUEST</b> | IONNA | IRE |
|-----|-----|------|--------------|-------|-----|

Please complete this questionnaire to the best of your abilities and return it in the enclosed postage-free envelope. If you have questions about the survey, you can contact a COMPASS Study Team Member at 1-844-501-7668.

- 1. During the past 3 months, did you help the stroke/TIA survivor with activities like preparing meals, shopping, getting and/or taking medications, scheduling and/or getting to doctor's appointments.
  - f O Yes, I helped with these activities ightarrow **PROCEED TO QUESTION 2**
  - O No, I did not help with these activities

| IF NO, did someone else help? O Yes | O No, the stroke survivor did not need help with these activities |
|---|---|
| You may stop the survey, please mail this survey back. Thank you for your time! | |

| 2. | How are you related to the stroke survivor? I am his/her | r | |
|---|---|---|---|
| 0 | Spouse O Neighbor or friend O Brother or sister | r O Parent or legal guardian | O Daughter or son |
| 0 | Other, please specify | | |
| | Since your loved one or friend was discharged from the bacare for him/her? (check only one) | nospital following his/her stroke, w | nat is the <u>total</u> length of time you provided |
| 0 | I have been providing care ever since he/she came home | O I provided care for 5-6 weeks | O I provided care for 11-12 weeks |
| 0 | I provided care for 1-2 weeks | O I provided care for 7-8 weeks | |
| 0 | I provided care for 3-4 weeks | O I provided care for 9-10 weeks | |
| 4. | At the time you were providing the <u>most</u> care, how many | y hours per week did you spend pro | oviding care? |

O Less than 10 hours per week O 10-19 hours per week O 20-29 hours per week O 30 or more hours per week

| 5. At any time over the past 3 months, have you provide the fo | | nce with ctivities? | | need help<br>nis assistance? | Did you also help wi<br>this before the strok | |
|---|---|---|---|---|---|---|
| | YES | NO | YES | NO | YES | NO |
| Bathing/showering | 0 | 0 | 0 | 0 | 0 | 0 |
| Dressing | 0 | 0 | 0 | 0 | 0 | 0 |
| Getting out of bed/chair | 0 | 0 | 0 | 0 | 0 | 0 |
| Helping to/from bathroom | 0 | 0 | 0 | 0 | 0 | 0 |
| Feeding | 0 | 0 | 0 | 0 | 0 | 0 |
| Preparing Meals | 0 | 0 | 0 | 0 | 0 | 0 |
| Shopping | 0 | 0 | 0 | 0 | 0 | 0 |
| Laundry | 0 | 0 | 0 | 0 | 0 | 0 |
| Handling Finances | 0 | 0 | 0 | 0 | 0 | 0 |
| Assistance with housework | 0 | 0 | 0 | 0 | 0 | 0 |
| Assisting with yardwork /house or car maintenance | 0 | 0 | 0 | 0 | 0 | 0 |
| Scheduling appointments (doctors, rehab, home health, etc.) | 0 | 0 | 0 | 0 | 0 | 0 |
| Transportation to pharmacy and medical appointments | 0 | 0 | 0 | 0 | 0 | 0 |
| Transportation to grocery store, places around town, etc. | 0 | 0 | 0 | 0 | 0 | 0 |
| Using Medication | 0 | 0 | 0 | 0 | 0 | 0 |

| If yes, please describe: | 100 1 0 0 0 0 0 0 0 0 0 0 0 0 0 0 0 0 0 | | | |
|---|---|---|---|---|
| 7. Does anyone else provid | de care for this stroke survivor? O Yes O No | | | _ |
| If YES, please indicate v | who these people are and how they are related to the stroke survivor. (Ch | eck all that apply) | | |
| O Spouse | O Neighbor or friend | | | |
| O Brother or sister | O Parent or legal guardian | | | |
| O Daughter or son | O Other, please specify | | | |
| | | Yes, on a | elp you think a | |
| | | regular basis | sometimes | No |
| My sleep is disturbed (light) | For example: the person I care for is in and out of bed or wanders around at | 0 | 0 | 0 |
| Caregiving is inconveniently help.) | ient (For example: helping takes so much time or it's a long drive over to | 0 | 0 | 0 |
| Caregiving is a physica required.) | d strain (For example: lifting in or out of a chair; effort or concentration is | 0 | 0 | 0 |
| Caregiving is confining | (For example: helping restricts free time or I cannot go visiting.) | 0 | 0 | 0 |
| There have been family privacy.) | v adjustments (For example: helping has disrupted my routine; there is no | 0 | ٥ | 0 |
| There have been chang<br>on vacation.) | es in personal plans (For example: I had to turn down a job; I could not go | 0 | 0 | 0 |
| 7. Does anyone else provide care for this stroke survivor? | | | | |
| | onal adjustments (For example: severe arguments about caregiving.) | 0 | 0 | 0 |
| There have been emotion | | 0 | 0 | 0 |
| Some behavior is upset | the person reale for accuses people of taking timigs.) | | 0 | 0 |
| Some behavior is upset<br>remembering things; or t | he person I care for has changed so much from his/her former self (For | 0 | 100000 | |
| Some behavior is upset remembering things; or to the sample: he/she is a different to the sample: he/she is a different to the sample: he/she is a different to the sample: he/she is a different to the sample to the sample. | the person I care for has changed so much from his/her former self (For ferent person than he/she used to be) | 20-50 | 0 | 0 |
| Some behavior is upset remembering things; or to the example: he/she is a difference have been work. | he person I care for has changed so much from his/her former self (For ferent person than he/she used to be) adjustments (For example: I have to take time off for caregiving duties.) | 0 | 86 | |

# Appendix 28 - Proxy SIS-16

Removed – COMPASS is no longer asking caregiver's questions about the patient. The Proxy SIS-16 has been removed.

## Appendix 29 - Caregiver Letter (Second Attempt)



Dear < NAME CG>,

Greetings from the COMPASS Study team! We are writing to invite you to participate in our survey. With your help, we hope to understand more about the best way to care for stroke survivors and their families after they go home from the hospital - to help them find the way forward to recovery.

We know how important family, friends, and neighbors are during the recovery process. We also understand that it can be difficult to care for loved ones who have had a stroke. Through the COMPASS Study, we hope to learn more about the needs of those who provide care and assistance to stroke survivors.

<PATIENT NAME> has identified you as the person who has been helping <HIM/HER> recover following <HIS/HER> stroke. <HE/SHE> was discharged on <DSCHRGDATE> from <HOSPITAL NAME>, which is participating in the COMPASS study. We invite you to take part in the COMPASS Study by completing a survey about caring for <HIM/HER>. This survey should only take about 15 minutes and is completely voluntary and confidential.

Your input is important and will help us improve support systems for family members and friends who provide care to stroke survivors. Please complete the enclosed survey and send it back in the postage-free envelope we have provided by <Due Date>

### Find out more about the COMPASS Study



To learn more about the COMPASS Study and to find other useful information about care after stroke, please visit our website: www.nccompass-study.org



We thank you very much for your time and contribution to the COMPASS Study!

Best regards,

The COMPASS Study Team

<CG\_ID>



# Appendix 30 - Caregiver Thank You Note

Removed – COMPASS will no longer be sending a 10 dollar gift card to caregivers.

## Appendix 31 - IRB Approval Letter for PCORI Stakeholder Interviews



Office of Research
INSTITUTIONAL REVIEW BOARD

#### MEMORANDUM

To: Sabina Gesell Ph D

PHS-Social Sciences

From: Protocol Analyst, Institutional Review Board

Date: 8/4/2015

Subject: Human Protocol: IRB00028495

Stakeholder interviews to shape PCORI Pragmatic Clinical Trial application

Amendment 2 for IRB Study #IRB00028495

#### Study Documents:

Protocol Version: PCORI Focus Group\_Protocol.docx, Protocol\_Stakeholder Interviews\_v2.doc; Other Documents: PCORI Focus Group\_Consent Form\_compensated\_CLEAN.docx, PCORI Focus Group\_Consent Form\_not compensated\_CLEAN.docx, PCORI Interviewing Script.docx, PCORI Interviewing\_Consent Form\_v3\_CLEAN.docx

The amendments listed below have been approved in accordance with HHS regulations for the protection of human research subjects that provides for the expedited review and approval of minor changes in previously approved research [45 CFR 46.110(b)(2)]. This action of the Board does not extend the term of approval for this protocol.

The amendment includes the following:

garrel Sexics

- A new protocol for focus groups has been added that will ask more specific questions about the recent developments of the COMPASS Intervention.
- 2. Two new consent forms that align with the new focus group protocol have been added. One consent form will be for participants that will not be compensated for their time in the study. The other consent form will be for participants that will be compensated for their time in the study.

This IRB is in compliance with the requirements of Part 56, 21 Code of Federal Regulations published as of April 1994 and Part 46, Subpart A of 45 CFR published January 26, 1981.

Jeannie Sekits

Medical Center Boulevard, Winston-Salem, NC 27157-1023 (336) 716-4542 / fax (336) 716-4480

### **Appendix 32 - DSMB Template Sections**

### List of Report Sections

- 1. Executive Summary
- 2. Protocol Synopsis
  - a. Project Organizational Chart
  - b. Study Purpose
  - c. Projected Timetable And Schedule
  - d. List Of Participating Hospitals
- 3. Narrative & Trial Summary
  - a. Study Status
- 4. Recruitment And Randomization
- 5. Training
- 6. Implementation Of The Compass Study And Assessment Of Fidelity
- 7. Vanguard Hospital
- 8. Safety And Privacy Of Participants
- 9. Outcomes
- 10. Publications
- 11. Contract Modifications
  - a. Recommendations From The DSMB
  - b. Summary Of Protocol Changes
- 12. Recruitment And Participant Status: Figures & Tables
  - a. Hospital Recruitment And Randomization
  - b. Participant Enrollment And Outcome Ascertainment
- 13. Data Quality Tables
  - a. Study Activity Completion
  - b. Quality Analysis Of Implementation
  - c. Summary Of Data Form Completion
- 14. Appendices
  - a. Bimonthly Survey For Implementation Site Webinars With Post-Acute Coordinators (Pac) And Advanced Practice Providers (App)
  - b. Monthly Performance Report Templates
  - c. Bimonthly Survey For Implementation Site Webinars With Home Health And Outpatient Rehabilitation Teams
  - d. List Of Publications And Presentations For Compass

# Appendix 33 - CTSI Supplemental Proposal (Implementation of COMPASS)

Implementation of an evidence-based chronic disease care model: Identifying individual, organizational, and community facilitators (Gesell / Lutz)

### **RESEARCH PLAN**

### Specific Aims:

**Aim 1.** Evaluate the Reach, Adoption, Implementation, and Maintenance (RE-AIM) of the COMPASS intervention, an evidence-based chronic disease care management model.

**Aim 2.** Identify individual, organizational, and community factors that facilitate or are challenges to implementation of COMPASS.

**Aim 3.** Identify strategies to build, maximize, and sustain community resource networks working together with the local hospital-based post-acute care coordination teams to support local implementation of COMPASS.

### **Design & Methods**

**Study Design:** We will capture quantitative data via (1) bi-weekly questionnaires to the hospital-based post-acute care (PAC) teams and Home Health Outpatient Therapy (HHOP) Teams to capture perceived barriers to uptake, and (2) real-time data on enrollment and performance measures at each site. We also will capture qualitative data via (1) transcription and coding of bi-weekly phone calls with PAC teams, and HOPP team and (2) semi-structured interviews with the Director of Implementation for the COMPASS study and members of the Implementation Committee. These calls will be facilitated by the Director of Implementation for the COMPASS study (S. Coleman) and will allow post-acute care coordinators to problem-solve together. These 4 data sources, collected from 20 health systems over one year, will identify which patient, staffing, and community-level factors drive intervention uptake, challenges to uptake, and how health systems can improve performance on pre-defined performance measures.

**Sample:** In the COMPASS study, 41 hospitals have been randomized (stratified by stroke volume and primary stroke center status) to receive COMPASS or usual care (control group). The proposed pilot will include the 20 hospitals randomized to receive COMPASS. Roll-out of these 20 intervention sites has occurred in 3 waves (n=5, n=5, n=10), starting in August 2016. Within each wave, hospitals trained together and started implementation at the same time; they also participate in bi-monthly problem-solving calls together. We are adapting strategies after each wave to meet health systems' unique environments and optimize approaches accordingly.

**Measurement Framework:** The RE-AIM Framework, developed by Glasgow et al (1999), will guide the process evaluation of the implementation of COMPASS. RE-AIM guides the assessment of the **Reach**, **Effectiveness**, **Adoption**, **Implementation**, and **Maintenance** of public health interventions (e.g., policy or programmatic). **Table 1** defines the RE-AIM components for COMPASS. **Table 2 (Appendix)** shows how the RE-AIM framework will guide the proposed process evaluation. Re-Aim has been used to evaluate the implementation of other large trials (e.g., ATTEND https://clinicaltrials.gov/ct2/show/NCT02123875).

**Table 1. RE-AIM Components Defined for COMPASS** 

| Reach | Effectiveness | Adoption | Implementation | Maintenance |
|---|---|---|---|---|
| of intended | | by target staff, | consistency, and | of intervention effects |
| population | | settings, or | adaptations made | in individuals and |
| | | institutions | during delivery | settings over time |

Application - IRB00035998

| The absolute number, | The impact of | The absolute number, | The intervention | The extent to which |
|---|---|---|---|---|
| proportion, and | COMPASS on | proportion, and | agents' fidelity to the | COMPASS becomes |
| representativeness of | important outcomes, | representativeness of | various elements of | institutionalized or |
| patients who are | including potential | hospitals and | an intervention's | part of the routine |
| enrolled in | negative effects, | clinicians who are | protocol, including | organizational |
| COMPASS at | quality of life, and | willing to initiate | consistency of | practices and policies |
| hospital discharge | economic outcomes | COMPASS | delivery as intended | |
| | | | and the time and cost | |
| | | | of the intervention | |

**Data Collection:** In this mixed methods design, we will collect quantitative data via (1) bi-weekly questionnaires to the hospital-based post-acute care (PAC) teams and HHOP teams to capture perceived barriers to uptake (see **Appendix** for survey), and (2) how well the clinic is actually implementing the new care model (i.e., real-time data on enrollment and performance measures). We also will capture qualitative data via (1) transcription and coding of bi-weekly phone calls with PAC teams and HHOP Calls (2) semi structured interviews with the Director of Implementation for the COMPASS study and members of the Implementation Committee (see **Table 3**). The bi-weekly calls are facilitated by the Director of Implementation for the COMPASS study (Coleman) and allow PAC teams across the state to problem-solve together. These 4 data sources, collected from 20 health systems over one year, will allow us to triangulate which patient, staffing, and community-level factors drive intervention uptake, which pose challenges to uptake, and which drive health systems' ability to improve performance.

**Table 3. Data Sources** 

| Quantitative Data Source | Qualitative Data Source |
|---|---|
| Bi-weekly questionnaires to the hospital-based post-acute care (PAC) and HHOP teams to capture perceived barriers to uptake | Transcription of bi-weekly phone calls with PAC and HHOP teams to problem solve barriers to uptake |
| Real-time data on patient enrollment | Semi-structure interviews with the Director of Implementation for the COMPASS study (Coleman, RN) |
| Real-time data on 6 performance measures | Semi-structured interviews with members of the COMPASS Implementation Committee |

**Quantitative Data Analysis:** Descriptive statistics (e.g., frequencies) will be used to aggregate questionnaire responses.

Qualitative Data Collection and Analysis: PAC team phone calls and interviews with the Director of Implementation and members of the Implementation Committee will be audio recorded and transcribed verbatim by Accukey Transcription (vendor #25466). Transcripts will be de-identified and verified by study investigators. Transcripts will be imported into NVivo for data management and analysis. The transcripts will be coded independently by members of the research team including the PI and Co-PI, and a graduate student research assistant (RA) trained in qualitative research methods. Initially, phone calls and interviews will be coded using open coding procedures as described by Charmaz (2006) and Ryan and Bernard (2003). The research team will meet to discuss the codes identified in the data. Codes will be sorted and categorized into themes that represent the factors that affect implementation (e.g. challenges, facilitators, and strategies). A coding schema will be developed collaboratively by the PI, Co-PI (Gesell / Lutz), and student RA. This schema will be used to code subsequent team meeting transcripts. The coders will meet regularly (monthly) to discuss the ongoing coding and resolve discrepancies. Major themes will be reported with supporting quotations. Credibility of analysis will be enhanced by (1) independent coding; (2) examination of negative cases and situations of considerable agreement or disagreement; (3) qualitative assessment of agreement between coders over time; and (4) discussing the major themes with the PACs in the 3 Waves to get input and feedback (member checking). Our analysis will also include cross-comparisons of subgroups (urban/rural sites, large/small volume sites) to determine differences within a heterogeneous population of health systems.

Table 4. Mapping the RE-AIM framework (Glasgow et al 1999) to the proposed process evaluation

| Table 4. Mapping the RE-AIM framework (Glasgow et al 1999) to the proposed proces | 5 ev | aiuai | 1011 | | |
|---|---|---|---|---|---|
| | Reach | Effectiveness* | Adoption | Implementation | Maintenance |
| Characteristics of enrolled patients (age, language, sex, race, Hispanic, insurance, diagnosis, aphasia, ambulatory status at discharge, NIH stroke score) | Х | | | | |
| PM1. Receipt of follow-up telephone call within 2 business days of hospital discharge | | | | Χ | |
| PM2. Receipt of follow-up visit within 7 to 14 days of hospital discharge | | | | Χ | |
| PM3. Receipt of e-Care plan during follow-up clinic visit | | | | Χ | |
| PM4. Receipt of all home health and outpatient rehabilitation services (including physical therapy, occupational therapy, and speech and language therapy) prescribed at hospital discharge, 2-day follow-up call, or 7-14-day follow-up clinic visit by 30-days after hospital discharge | | | | Х | |
| PM5. Receipt of all home health rehabilitation services (including physical therapy, occupational therapy, and speech and language therapy) prescribed at hospital discharge, 2-day follow-up call, or 7-14-day follow-up clinic visit by 30-days after hospital discharge | | | | Х | |
| PM 6. Receipt of all <u>outpatient</u> rehabilitation services (including physical therapy, occupational therapy, and speech and language therapy) prescribed at hospital discharge, 2-day follow-up call, or 7-14-day follow-up clinic visit by 30-days after hospital discharge | | | | х | |
| Characteristics of enrolled health systems (size, location, Comprehensive Stroke Center certification) | | | Х | | |
| Characteristics of PAC teams (number of FTE, license, etc) | | | Х | | |
| Characteristics of Community Resource Networks | | | Χ | | |
| Characteristics of clinical staff participating in bi-weekly problem solving calls | | | Χ | | |
| Challenges with enrollment, 2 day call, 14 day visit, e care plan, receipt of therapy, community resource network, administrative tasks | | | | Х | |
| Requests for additional training | | | | Х | |
| Time it takes to integrate COMPASS components into system (ramp up) | | | | | Х |
| What are sites doing to maintain COMPASS? What are they changing? Are they returning to their original model of care? | | | | | Х |
| *90-day outcomes and claims data are part of the COMPASS trial, not this pilot | | *X | | | |
| PM = Performance Measure | 1 | | 1 | 1 | |
# March 19, 2021 Application - IRB00035998 Appendix 34 – 2Day Disposition Form

| ID Number: | Form Code: C D S P Date: 07JUN2016 Version 1.0 |
|---|---|
| ADMINISTRA | Date: Day |
| Did you c hospital? | complete a follow-up call with the patient or caregiver after the patient was discharged from the |
| | s → Go to Q1a |
| □ No | → Go to Q1b |
| | Month Day Year |
| 2b. Reas | son for no follow-up call: |
| | □ Did not attempt call |
| | ☐ Could not reach patient/caregiver after 2 attempts |
| | □ Patient/caregiver refused |
| | <ul> <li>□ Patient/caregiver could not complete (e.g. confused, unable to communicate, too sick, etc.)</li> <li>□ Patient/caregiver did not have workable number</li> </ul> |
| | ☐ Patient hospitalized |
| | ☐ Patient transferred to a skilled nursing facility |
| | □ Patient deceased |
| | □ Other (specify) |
| | END OF 2-DAY CALL DISPOSITION FORM |

# March 19, 2021 Application - IRB00035998 Appendix 35 – Clinic Disposition Form

| | Clinic Visit Disposition Form Form Code: V D S P Date: 10Feb2017 Version 2.0 |
|---|---|
| ADMINISTE<br>0a. Completio | RATIVE INFORMATION (0a-0c are auto-populated) n Date: Day |
| 1. Was the | e follow-up clinic visit conducted? |
| □ Y | es → Go to Q1a |
| □N | o → Go to Q1b, then END OF FORM |
| 1a. Dat | e of clinic visit: |
| 1b. If n | o visit was completed, select reason: |
| | <ul> <li>□ Visit NOT scheduled: Patient prefers to follow-up with his/her own PCP or another doctor</li> <li>□ Visit NOT scheduled: Patient reported that he/she is too sick or disabled to attend</li> <li>□ Visit NOT scheduled: Patient cannot afford to attend the scheduled visit</li> <li>□ Visit NOT scheduled: Patient does not have transportation</li> <li>□ Visit NOT scheduled: Patient reported that he/she lives out of the area and doesn't want to travel</li> </ul> |
| | <ul> <li>□ Visit was scheduled, but patient did not attend Transportation Issues No insurance coverage for visit Conflicting medical appointment </li> </ul> |
| | Patient/caregiver preferred not to drive a long distance for the follow-up visit Patient cancelled No show / reason unknown Other: |
| | □ Patient transferred to nursing home □ Patient hospitalized □ Patient deceased □ Other |
| | e Stroke Caregiver Assessment triggered by the Post-Stroke Functional Assessment? es → Go to Q2a |
| _ 11 | * |

| 2a. Was it performed? | |
|---|---|
| □ Yes | |
| $\square$ No $\rightarrow$ Go to Q2b | |
| 2b. Why not? | |
| <ul><li>□ Primary caregiver not present</li><li>□ Primary caregiver refused</li></ul> | |
| 3. Was the eCare Plan generated? | |
| <ul> <li>□ Yes, electronically on the iPad → Go to Q3a</li> <li>□ No → Go to Q3b</li> </ul> | |
| 3a. Was the eCare Plan printed and shared with the patient? | |
| □ Yes | |
| □ No | |
| 3b. Reason for no eCare Plan: | |
| ☐ Acute change of patient's status requiring emergent care | |
| ☐ Technical error / server problem | |
| ☐ Clinic workflow wouldn't allow generation of eCare Plan | |
| □ Other | |
| 4. Is the patient in need of any rehabilitation services that they are not currently receiving? | |
| ☐ Yes → Go to Q4a | |
| □ No | |
| 4a. What referrals were made after the clinic visit (check all that apply)? | |
| ☐ Home health PT ☐ Outpatient PT | |
| ☐ Home health OT ☐ Outpatient OT☐ Home health SLP☐ Outpatient SLP☐ | |
| <ul><li>5. Were referrals made to any pharmacy-based services?</li><li>☐ Yes → Go to Q5a</li></ul> | |
| □ No | |
| <ul> <li>5a. Which services (check all that apply)?</li> <li>☐ Community Care of North Carolina (CCNC) pharmacy network</li> <li>☐ Local pharmacy outside of the CCNC pharmacy network</li> <li>☐ Free clinic with on-site pharmacist</li> <li>☐ Hospital-based pharmacist follow-up</li> </ul> | |
| Clinic Visit Disposition Form | Page 2 of 3 |

| 6 Were referral | s made to community resources such as Area Agency on Aging, support groups, etc. | |
|---|---|---|
| (check all that | t apply?) | |
| □ Yes → | Go to Q6a | |
| □ No | | |
| | community services (check all that apply)? | |
| | Adult Services/Social Support Services<br>Stroke Support Group | |
| | Counseling Services for stress, depression (e.g. CareNet) | |
| | Chronic Disease Management Programs | |
| | Community Exercise Programs<br>Falls Prevention Programs | |
| | Nutrition Assistance Programs | |
| | Aphasia Support Group | |
| | Smoking Cessation Program<br>Transportation Services | |
| | Caregiver Support Services | |
| | Other Services: | |
| o <del></del> | END OF CLINIC VISIT DISPOSITION FORM | |
| | END OF CLINIC VISIT DISPOSITION FORM | |
| | END OF CLINIC VISIT DISPOSITION FORM | _ |
| | END OF CLINIC VISIT DISPOSITION FORM | _ |
| | END OF CLINIC VISIT DISPOSITION FORM | _ |
| | END OF CLINIC VISIT DISPOSITION FORM | |
| | END OF CLINIC VISIT DISPOSITION FORM | _ |
| | END OF CLINIC VISIT DISPOSITION FORM | _ |
| | END OF CLINIC VISIT DISPOSITION FORM | _ |
| | END OF CLINIC VISIT DISPOSITION FORM | _ |
| | END OF CLINIC VISIT DISPOSITION FORM | _ |
| | END OF CLINIC VISIT DISPOSITION FORM | _ |
| | END OF CLINIC VISIT DISPOSITION FORM | _ |
| | END OF CLINIC VISIT DISPOSITION FORM | |
| | END OF CLINIC VISIT DISPOSITION FORM | |
| | END OF CLINIC VISIT DISPOSITION FORM | |
| | END OF CLINIC VISIT DISPOSITION FORM | |

## **Appendix 36 - Phase 2 Patient Brochure for Sustaining COMPASS Hospitals**

#### Your recent hospital visit means that you are eligible for the COMPASS Study.

Your hospital is participating in a statewide study called the Comprehensive Post-Acute Stroke Services (COMPASS) Study. This study includes people who have had a stroke or transient ischemic attack (TIA), sometimes referred to as a mini-stroke. The purpose of the COMPASS Study is to determine the best ways to care for patients after they go home – to help survivors find their way forward to recovery.

#### Our hospital is providing the COMPASS model of post-acute care, which includes:

- A follow-up phone call 2 days after discharge
- A visit with a nurse practitioner, physician assistant, or doctor 7-14 days after discharge
- A plan of care that will be shared with your other health care providers
- Additional follow-up phone calls 30 and 60 days after discharge

We are committed to finding the best way to improve health and recovery after experiencing this health episode. In addition to the COMPASS care, you will continue to receive high-quality care at our hospital and at your usual follow-up visits with your primary care doctors.

**After you have left the hospital,** the COMPASS team would like to learn about your overall experience. They will:

- Call you in 3 months to ask questions about your recovery and satisfaction with your care
- Mail you 3 reminder letters before you are called. The last letter will include a small gift to thank you for your time, so be sure to open it.

Whether or not you choose to participate in the survey, our hospital is committed to providing you with high-quality care for you during your recovery. All information provide will be kept strictly confidential and secure.

**If you have any questions** about the COMPASS Study, or prefer not to participate, feel free to ask the stroke coordinator, or you may call the COMPASS Study team using the toll-free number below.

COMPASS Study toll-free number: 1-844-501-7668 COMPASS Study website: <a href="https://www.nccompass-study.org">www.nccompass-study.org</a>



## Appendix 37 - Phase 2 Patient Brochure for Intervention Sites (formerly Usual Care)

#### Your recent hospital visit means that you are eligible for the COMPASS Study.

Your hospital is participating in a statewide study called the Comprehensive Post-Acute Stroke Services (COMPASS) Study. This study includes people who have had a stroke or transient ischemic attack (TIA), sometimes referred to as a mini-stroke. The purpose of the COMPASS Study is to determine the best ways to care for patients after they go home – to help survivors find their way forward to recovery.

#### Our hospital is providing the COMPASS model of post-acute care, which includes:

- A follow-up phone call 2 days after discharge
- A visit with a nurse practitioner, physician assistant, or doctor 7-14 days after discharge
- A plan of care that will be shared with your other health care providers
- Additional follow-up phone calls 30 and 60 days after discharge

We are committed to finding the best way to improve health and recovery after experiencing this health episode. In addition to the COMPASS care, you will continue to receive high-quality care at our hospital and at your usual follow-up visits with your primary care doctors.

**After you have left the hospital,** the COMPASS team would like to learn about your overall experience. They will:

- Call you in 3 months to ask questions about your recovery and satisfaction with your care.
- Mail you 3 reminder letters before you are called. The last letter will include a small gift to thank you for your time, so be sure to open it.

Whether or not you choose to participate in the survey, our hospital is committed to providing you with high-quality care for you during your recovery. All information provide will be kept strictly confidential and secure.

**If you have any questions** about the COMPASS Study, or prefer not to participate, feel free to ask the stroke coordinator, or you may call the COMPASS Study team using the toll-free number below.

COMPASS Study toll-free number: 1-844-501-7668 COMPASS Study website: <a href="https://www.nccompass-study.org">www.nccompass-study.org</a>



# March 19, 2021 Application - IRB00035998 Appendix 38 – Phase 2Enrollent Form

| COMPAS COMPREHENSIVE POST-ACI | Dautiain and Envallment Fauna | |
|---|---|---|
| ID Number: | | Version 2.0<br>(Phase 2) |
| ADMINISTRATIVE INFORM | MATION (auto-populated) | |
| 0a. Completion Date: | / Day / Pear Ob. Staff ID: | |
| 0c. NCSCC ID: | Od. Hospital ID: Of. | Form Status: |
| A. PATIENT CONTACT IN | FORMATION | |
| Patient full name | First Middle | Last |
| 2. Telephone number(s) | | |
| a. Primary number: ( | | |
| | lome □ Mobile □ Work □ Other<br>Veekday daytime □ Weekday evening □ Weekend □ Anytime | |
| b. Alternate 1: ( | ) | |
| | lome ☐ Mobile ☐ Work ☐ Other | |
| Best time to call: □ V | Veekday daytime ☐ Weekday evening ☐ Weekend ☐ Anytime | |
| c. Alternate 2: | ) | |
| 505 | lome Mobile Work Other | |
| Best time to call: $\square V$ | Veekday daytime ☐ Weekday evening ☐ Weekend ☐ Anytime | <u> </u> |
| 4. Home address | Address line 1 | |
| 7 | Address line 2 | |
| ( | Dity State Zip | County |
| Participant Enrollment Form v2.0 for Ph | uase 2 | Page 1 of 5 |

| ,, | .g 0aop0 | ng to doctor |
|---|---|---|
| ontact / not documented | → Go to Qu | estion 16 |
| S- | _, | |
| Middle | | Last |
| Other | | |
| ☐ Other | | |
| | - | |
| State | Zip | |
| | medications, scheduling medica | Other Other State Zip |

| ☐ Asian☐ American☐ Native HI | ):<br>rican American<br>Indian / Alaska Native<br>/ Other Pacific Islander | |
|---|---|---|
| 18. Hispanic ethnicity: ☐ Yes | □ No | |
| ☐ Medicare | Supplemental Insurance / Med<br>surance<br>npus / other | ligap |
| 20. Does the patient have documented | ed past medical history of the f | ollowing (check all that apply): |
| <ul><li>☐ Stroke</li><li>☐ Transient ischemic attack</li></ul> | ☐ Hypertension☐ Dyslipidemia | <ul><li>☐ Chronic renal insufficiency</li><li>☐ Heart Valve</li><li>☐ Current pregnancy or within 6</li></ul> |
| <ul> <li>□ Atrial Fibrillation or Flutter</li> <li>□ Myocardial infarction or CAD</li> <li>□ Congestive heart failure</li> <li>□ Carotid stenosis</li> <li>□ Peripheral arterial disease</li> </ul> | <ul> <li>☐ Smoking</li> <li>☐ Depression</li> <li>☐ Drug/alcohol abuse</li> <li>☐ Family history of stroke</li> <li>☐ Migraines</li> </ul> | weeks post-partum Hormone replacement therapy Sickle cell Sleep apnea Diabetes mellitus |
| 21. Please enter the body mass inde | x (BMI) kg/m² | □ Not documented |
| 22. What was the patient's ambulator | ry status <u>prior to admission</u> ? | |
| | | vithout a device) |
| 23. Initial NIH Stroke Scale Score (00 | )-42) | Not documented |
| 25. Did the initial exam show aphasia | a? ☐ Yes ☐ No / not do | ocumented |
| 26. Hospital admission date for this e | event: / / | / |
| ☐ No admission date; patient was | not admitted as an inpatient (s | select reason below) |
| | lirectly from ED to home rom observation status without | inpatient admission |

| 2/a. If YES | S, check all that apply: | |
|---|---|---|
| ☐ Hom | e health Physical Therapy e health Occupational Therapy e health Speech Therapy Outpatient Physical Therapy Outpatient Occupational Therapy Outpatient Speech Therapy | |
| 27b. If NO | indicate why not | |
| ☐ Patie | nt not evaluated for need of rehab services<br>nt not in need of rehab services<br>nt / family refused<br>r reason | |
| 28. What w | as the patient's ambulatory status at discharge? | |
| | <ul> <li>□ Able to ambulate independently (with or without a device)</li> <li>□ With assistance (from person)</li> <li>□ Unable to ambulate</li> <li>□ Not documented</li> </ul> | |
| 30. Hospita | I discharge date: | |
| | ollow-up clinic visit with a nurse, nurse practitioner, or physician assistant (i.e. p<br>nal care clinic, neurologist, or other doctor visit) scheduled prior to discharge? | rimary care, |
| | ☐ Yes → Fill in type and date below | |
| 31a | ☐ No If YES, check all visit types that apply and enter the date (if known) | |
| 0.4 | □ Primary care | |
| | COMPASS clinic visit | |
| | Other transitional care visit with nurse and APP | |
| | ☐ Other transitional care visit with primary care | I · |
| | □ Rehab | |
| | □ Neurologist | |
| | □ Cardiologist | |
| | □ Other | |
| 32. Name o | f patient's primary care provider: | _ □ Not known |

| ppnemier resources | |
|---|---|
| 34. Did the PAC notify the patient of the COMPASS study by distributing the brochure? | |
| <ul> <li>☐ Yes, distributed the brochure in person</li> <li>☐ Yes, mailed brochure to patient</li> <li>☐ No</li> </ul> Fill in date below Fill in date below | |
| If YES, enter date of notification or mailing: | |
| Month Day Year | |
| END OF PARTICIPANT ENROLLMENT FORM | |
| Participant Enrollment Form v2.0 for Phase 2 | Page 5 of 5 |

### **Appendix 39 - Consent Matrix**



#### **MEMORANDUM**

To: Wake Forest Health Sciences IRB

From: Mysha Sissine, MSPH

Date: May 12, 2016

Subject: Outlines how data from COMPASS will be used for research purposes

The COMPASS Study is enrolling all eligible patients from participating hospitals. All patients are informed about the study and they are enrolled. This is done prior to gaining explicit consent from the patient. This is permissible because of the low-risk nature of the study and meeting the criteria for HIPAA Waivers.

Recognizing that this process is novel and different from other traditional approaches to consent, the study team worked through a number of scenarios to better define who is included in research analysis and who is excluded. That is detailed in the consent matrix on the next page.

Like all other studies, COMPASS patients can opt out (or withdraw) from the study at any time. At four time points COMPASS letters are provided to each enrolled patient and each letter includes information on how they can opt-out from the study (a brochure, 30d letter, 60d letter, & 80d letter).

In determining what data were acceptable to use for analysis, our team considered both the regulatory requirements and additional protections to conservatively maintain the rights and welfare of study participants. In particular, we determined that we would not use any data past the eligibility screening form from patients who withdrew from the study regardless of the time point of withdrawl. This is more stringent from the regulation, which says that studies can use data up until the point that a patient withdraws. However, since COMPASS is not explicitly gaining consent prior to enrollment (instead we are relying on the patient to out-out) we will make the assumption that if someone was to opt-out (i.e. withdraw) that same patient would not have initially provided consent to be enrolled.

In addition, if a patient withdrawals from the study (again at any time point) that withdrawal will also remove that patient's <u>clinical data from research analysis</u>, even if that patient had provided signed clinical consent (at the 7-14 day visit). This was put in place because the study team made the conservative estimate that a study patient would not be able to adequately distinguish between the two consent processes and articulate their wish to withdraw from some but all parts of the study.



### **Data Usage for Research Purposes**

| Data Form | Covered by | Rules for Use | Exclusions from<br>Analysis |
|---|---|---|---|
| ELG | Limited HIPAA waiver | All patients ( <u>includes patients who withdrew</u> ). | |
| ENR | Full HIPAA waiver | All patients, <u>except</u> any patients who withdrew from the study (at any time point). | Withdraw=1 |
| NCSCC | Full HIPAA waiver | All patients, <u>except</u> any patients who withdrew from the study (at any time point). | Withdraw=1 |
| 2-d call | eCare consent | Include all patients who provided signed "clinic consent" and who have not withdrawn. | Research_consent ^=1<br> withdraw =1 |
| Clinic forms | eCare consent | Include all patients who provided signed "clinic consent" and who have not withdrawn. | Research_consent ^=1<br> withdraw =1 |
| eCare Plan | eCare consent | Include all patients who provided signed "clinic consent" and who have not withdrawn. | Research_consent ^=1<br> withdraw =1 |
| 30-d Call | eCare consent | Include all patients who provided signed "clinic consent" and who have not withdrawn. | Research_consent ^=1<br> withdraw =1 |
| 60-d Call | eCare consent | Include all patients who provided signed "clinic consent" and who have not withdrawn. | Research_consent ^=1<br> withdraw =1 |
| 90-d Data | 90-d verbal consent | All patients, <u>except</u> any patients who withdrew from the study (at any time point). | Withdraw=1 |
| Claims data | Full HIPAA waiver | We have a HIPAA Waiver to collect claims data on all patients. The data that we are using to link is from the COMPASS Dataset. Here is our linkage plan: • ELG form: We will use patient data from all records even if they withdrew from the study. • ENR form: We will use patient data to link them as long as they have not withdrawn from the study (at any time point). | |
| 2-d Dispo | Full HIPAA waiver | All patients, <u>except</u> any patients who withdrew from the study (at any time point). | Withdraw=1 |
| Clinic Dispo | Full HIPAA waiver | All patients, <u>except</u> any patients who withdrew from the study (at any time point). | Withdraw=1 |

March 19, 2021 Application - IRB00035998